# 1. TITLE PAGE



PROTOCOL NUMBER: 217-MDD-201 / NCT03000530
A PHASE 2, TWO-PART (OPEN-LABEL FOLLOWED BY DOUBLE-BLIND) STUDY EVALUATING THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND EFFICACY OF SAGE-217 IN THE TREATMENT OF ADULT SUBJECTS WITH MODERATE TO SEVERE MAJOR DEPRESSIVE DISORDER

**IND NUMBER: 132,131** 

Investigational Product SAGE-217

Clinical Phase 2a

Sponsor Sage Therapeutics, Inc.

Sponsor Contact , M.D., Ph.D.

Sage Therapeutics 215 First Street

Cambridge, MA 02142

Phone:

Sponsor Medical Monitor , M.D., M.P.H.

Study Physician Sage Therapeutics 215 First Street

Cambridge, MA 02142

Phone:

Date of Original Protocol Version 1.0, 24 October 2016

Date of Amendment One Version 2.0, 13 January 2017

Confidentiality Statement

The confidential information in this document is provided to you as an Investigator or consultant for review by you, your staff, and the applicable Institutional Review Board/Independent Ethics Committee. Your acceptance of this document constitutes agreement that you will not disclose the information contained herein to others without written authorization from the Sponsor.

# PROTOCOL SIGNATURE PAGE

**Protocol Number:** 

217-MDD-201

**Product:** 

SAGE-217 Oral Solution

IND No.:

132,131

Study Phase:

2a

Sponsor:

Sage Therapeutics

Date of Amendment One: Version 2.0 13 January 2017



# **INVESTIGATOR'S AGREEMENT**

I have received and read the Investigator's Brochure for SAGE-217. I have read the Clinical Protocol 217-MDD-201 and agree to conduct the study as outlined. I agree to maintain the confidentiality of all information received or developed in connection with this protocol.

| Printed Name of Investigator |
|------------------------------|
| Signature of Investigator |
| Date |

# CONTACTS IN CASE OF EMERGENCY

**Table 1:** Emergency Contact Information

| Name | Address and Telephone Number | |
|------|------------------------------|----------------------------------------|
| | LICA | |
| | USA | |
| | Name | Name Address and Telephone Number USA |

# 2. SYNOPSIS

## Name of Sponsor/Company:

Sage Therapeutics 215 First Street

Cambridge, MA 02142

# Name of Investigational Product:

SAGE-217 Oral Solution

#### Name of Active Ingredient:

SAGE-217

**Title of Study:** A Phase 2, Two-Part (Open-Label Followed by Double-Blind) Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of SAGE-217 in the Treatment of Adult Subjects With Moderate to Severe Major Depressive Disorder

**Study centers:** Approximately 3 sites in Part A and approximately 15 sites in Part B

Phase of development: 2a

#### Methodology:

This study will assess the safety, tolerability, pharmacokinetics (PK), and efficacy of SAGE-217 Oral Solution in adult subjects diagnosed with moderate to severe major depressive disorder (MDD).

There are two parts to the study:

**Part A**: Open-label dosing with SAGE-217 Oral Solution (14 days)

All subjects will receive a 30 mg SAGE-217 Oral Solution dose administered at 8:00 PM ( $\pm 15$  minutes) with food on Day 1 to Day 14 as tolerated.

**Part B**: Randomized, double-blind, parallel-group, placebo-controlled (14 days)

Based on the results of Part A, eligible subjects will be stratified based on use of antidepressant treatment (current/stable or not treated/withdrawn ≥30 days) and randomized within each stratum in a 1:1 fashion to receive SAGE-217 Oral Solution 30 mg or matching placebo for 14 days beginning on Day 1 as tolerated. All doses of study drug will be administered at 8:00 PM (±15 minutes) with food. Dose adjustments based on tolerability are detailed in Section 9.3.

Separate cohorts of subjects will be enrolled in Part A and Part B; subjects participating in Part A cannot enroll in Part B. Part B may be initiated and enrollment into Part A stopped if there is a clear signal of activity based on the 17-item Hamilton Rating Scale for Depression (HAM-D) scores and/or other scales being assessed.

Both parts of the study will consist of an up to 7-day Screening Period (Days -7 to -1), a 14-day Treatment Period, and a 2-week Follow-up Period. During the study Treatment Period, subjects must remain inpatient for the first 7 days at minimum and per Investigator's judgement thereafter.

Screening Period: The Screening Period begins with the signing of the informed consent form (ICF) at the Screening Visit, which can occur on any two consecutive calendar days of the 7-day window (from Day -7 through Day -1). The diagnosis of MDD must be made according to Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Axis I Disorders (SCID-I) performed by a qualified healthcare professional. Subjects will undergo preliminary screening procedures at the Screening Visit to determine eligibility, including completion of the HAM-D, Hamilton Anxiety Rating Scale (HAM-A), Clinical Global Impression - Severity (CGI-S), and Montgomery-Åsberg Depression Rating Scale (MADRS). The Screening Period assessments will be conducted on an outpatient basis. Most eligibility criteria are the same for both parts of the study.

## **Treatment Period:**

Part A – Once subjects are confirmed as eligible, they will receive a 30 mg dose of study drug at 8:00 PM ( $\pm15$  minutes) with food for 14 days (Day 1 to Day 14) as tolerated. Subjects who cannot tolerate 30 mg will receive 20 mg for the rest of the Treatment Period. Subjects who cannot tolerate 20 mg will be terminated from the study. The following assessments will be performed: HAM-D, HAM-A, and MADRS total scores and Clinical Global Impression – Improvement (CGI-I).

Enrollment into Part A may be stopped and Part B initiated if there is a clear signal of activity based on the HAM-D scores and/or other scales being assessed. Alternatively, upon completion of Part A, Part B may begin. The study may be terminated if there is clear lack of activity based on HAM-D scores during Part A. Separate cohorts of subjects will be enrolled in Part A and Part B; subjects participating in Part A cannot enroll in Part B.

Part B - Based on the results of Part A, eligible subjects will be stratified based on use of antidepressant treatment (current/stable or not treated/withdrawn  $\geq 30$  days) and randomized within each stratum to one of two treatment groups (SAGE-217 Oral Solution 30 mg or matching placebo) in a 1:1 ratio. Subjects will be administered study drug at 8:00 PM ( $\pm 15$  minutes) with food for 14 days. Subjects who cannot tolerate 30 mg will receive 20 mg for the rest of the Treatment Period. Subjects who cannot tolerate 20 mg will be terminated from the study.

In both parts of the study, subjects may be discharged after a minimum 7-day inpatient stay, following completion of the Day 7 assessments. If their clinical condition does not allow discharge, the Investigator may keep the subjects as inpatients for a longer period of time.

In both parts of the study, subjects discharged from the inpatient unit may receive treatment with study drug for the remainder of the 14-day Treatment Periods as outpatients. The outpatient phase treatment may be provided at the clinical site or, if suitable arrangements can be made, via home administration. Home administration of study drug will be performed according to a site-specific plan by a healthcare professional trained on the protocol and delivery of the study drug.

With the exception of subjects permitted to use current stable antidepressant treatment, initiation of psychotropic medications and other medications that may potentially have an impact on efficacy or safety endpoints will not be allowed between screening and completion of the Day 15 assessments (Parts A and B). Psychotropic medications, which must have been initiated at least 14 days prior to screening, must remain at a stable dose until completion of the Day 15 assessments (Parts A and B).

Efficacy and safety assessments will be performed periodically during the study, and blood samples will be collected for analysis of SAGE-217 as outlined in the Schedule of Events (Table 2 and Table 3).

**Follow-up Period:** Follow-up visits will be conducted on an outpatient basis. Follow-up visits for Parts A and B will be conducted at 1 week (21±1 day) and 2 weeks (28±3 days) after the last dose of study drug.

#### **Objectives:**

#### Part A:

#### **Primary:**

The primary objective of the study is to evaluate the safety and tolerability of SAGE-217 Oral Solution 30 mg.

#### **Secondary:**

The secondary objective of Part A is to determine if treatment with SAGE-217 Oral Solution 30 mg for 14 days reduces depressive symptoms.

#### Part B:

#### **Primary:**

The primary objective of the study is to evaluate the safety and tolerability of SAGE-217 Oral Solution 30 mg.

#### Secondary:

The secondary efficacy objective for Part B of the study is to determine if treatment with SAGE-217 Oral Solution 30 mg reduces depressive symptoms in subjects with moderate to severe MDD compared to matching placebo.

## **Endpoints:**

#### Part A:

#### **Primary:**

The primary endpoint is the safety and tolerability of SAGE-217 as assessed by the frequency and severity of adverse events; changes from baseline in clinical laboratory measures, vital signs, and electrocardiograms (ECGs); Stanford Sleepiness Scale (SSS) score; physical examination; and suicidal ideation using the Columbia-Suicide Severity Rating Scale (C-SSRS).

# **Secondary:**

Reduction in depressive symptoms as assessed by the following:

- Change from baseline in HAM-D total score at all time points;
- HAM-D response;
- HAM-D remission;
- Change from baseline in the MADRS total score at all time points;
- Change from baseline in HAM-D subscale and individual item scores at all time points; and
- CGI-I response.

#### Part B:

#### **Primary:**

The primary endpoint is the safety and tolerability of SAGE-217 as assessed by the frequency and severity of adverse events; changes from baseline in clinical laboratory measures, vital signs, and ECGs; SSS score; physical examination; and suicidal ideation using the C-SSRS.

#### **Secondary:**

Reduction in depressive symptoms, compared to placebo, as assessed by the following:

- Change from baseline in the 17-item HAM-D total score at all time points;
- HAM-D response;
- HAM-D remission;
- Change from baseline in the MADRS total score at all time points;
- Change from baseline in HAM-D subscale and individual item scores at all time points;
- CGI-I response; and
- 36-item short form survey (SF-36) and fatigue associated with depression (FAs-D) patient-reported outcome.

#### Pharmacokinetic:

The PK objective of Part A and Part B is:

• To assess the PK profile of SAGE-217 Oral Solution in plasma samples.

## Number of subjects (planned):

Approximately ten subjects will be enrolled in Part A. Up to 52 subjects may be randomized in Part B.

# Diagnosis and main criteria for inclusion:

#### **Inclusion criteria:**

- 1. Subject has signed an ICF prior to any study-specific procedures being performed.
- 2. Subject is an ambulatory male or female between 18 and 65 years of age, inclusive.
- 3. Subject is in good physical health and has no clinically significant findings, as determined by the Investigator, on physical examination, 12-lead ECG, or clinical laboratory tests.
- 4. Subject agrees to adhere to the study requirements.
- 5. Subject has a diagnosis of MDD that has been present for at least a 4-week period as diagnosed by SCID-I.
- 6. Subject has a HAM-D total score of  $\geq$ 22 at screening and Day 1 (prior to dosing).
- 7. Subject has a HAM-A total score of ≥20 at screening and Day 1 (prior to dosing) (Part B only).
- 8. Subject is willing to delay start of other antidepressant or antianxiety medications and any new pharmacotherapy regimens, including as-needed benzodiazepine anxiolytics, during the screening and treatment periods.
- 9. Subject agrees to practice an acceptable method of highly effective birth control at screening and throughout study participation. Highly effective methods of birth control include sexual abstinence (for males and females); vasectomy; or a condom with spermicide in combination with a highly effective female partner's method (for males); and hormonal methods of contraception (ie, established use of oral, implantable, injectable, or transdermal hormones); placement of an intrauterine device; placement of an intrauterine system; and mechanical/barrier method of contraception (ie, condom or occlusive cap [diaphragm or cervical/vault cap] in conjunction with spermicide [foam, gel, film, cream, or suppository]) (for females).

#### **Exclusion criteria:**

- 1. Subject has a history of suicide attempt.
- 2. Subject has a recent history or active clinically significant manifestations of metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, musculoskeletal, dermatological, urogenital, neurological, or eyes, ears, nose, and throat disorders, or any other acute or chronic condition that, in the Investigator's opinion, would limit the subject's ability to complete or participate in this clinical study.
- 3. Subject has a history of treatment-resistant depression, defined as persistent depressive symptoms despite treatment with adequate doses of antidepressants from two different classes for an adequate amount of time (ie, at least 4 weeks of treatment).
- 4. Subject has a known allergy to SAGE-217, allopregnanolone, or related compounds.
- 5. Subject has a positive pregnancy test at screening or on Day 1 prior to the start of study drug administration.
- 6. Subject has detectable hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV), or human immunodeficiency virus (HIV) antibody at screening.
- 7. Subject has active psychosis per Investigator assessment.
- 8. Subject has a medical history of seizures.
- 9. Subject has a medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder.

- 10. Subject has a history of alcohol or drug dependence (including benzodiazepines) in the 12 months prior to screening.
- 11. Subject has had exposure to another investigational medication or device within 30 days prior to screening.
- 12. Subject has been treated or randomized in this study (eg, Part A) or any other study employing SAGE-217 previously (ie, subject may not have received study drug and then re-enroll).
- 13. Subject has had administration of psychotropics that have been initiated within 14 days prior to screening and/or are not being taken at a stable dose.
- 14. Use of any known strong inhibitors and/or inducers of cytochrome P450 (CYP)3A4 within the 14 days or five half-lives (whichever is longer) or consumed grapefruit juice, grapefruit, Seville oranges, or St. John's Wort or products containing these within 30 days prior to receiving the first dose of study drug.
- 15. Subject has a positive drug and/or alcohol screen at screening or on Day 1 prior to dosing.

#### Investigational product, dosage and mode of administration:

SAGE-217 Oral Solution is available as a 6 mg/mL stock aqueous solution of SAGE-217 Drug Substance containing 40% hydroxypropyl- $\beta$ -cyclodextrin (HP $\beta$ CD) and 0.0025% sucralose, which is further diluted with Sterile Water for Injection to achieve the selected dose.

#### **Duration of participation:**

**Part A:** Up to 38 days (14 days of treatment) **Part B:** Up to 38 days (14 days of treatment)

#### Reference therapy, dosage and mode of administration:

Reference therapy is taste-matched placebo.

#### **Randomization:**

Subjects participating in Part A of the study will be administered study drug (SAGE-217 Oral Solution) in an open-label manner. Subjects in Part B will be randomized within each antidepressant treatment stratum to receive SAGE-217 Oral Solution or matching placebo oral solution in a 1:1 ratio. Subjects, clinicians, and the study team will be blinded to treatment allocation. The pharmacist and/or designated pharmacy staff, who will prepare the oral solutions according to the randomization schedule, will be unblinded.

#### Dose Adjustment for Safety/Tolerability Reasons:

During the Treatment Period, subjects will be able to receive study drug as long as there are no dose-limiting safety/tolerability concerns. Subjects who experience moderate or severe adverse events that according to the clinical judgement of the Investigator are related to study drug while receiving the 30 mg dose of study drug will receive 20 mg for the remaining of the Treatment Period. Subjects who experience moderate or severe related adverse events while receiving the 20 mg dose of study drug may not be able to continue receiving study drug based on the evaluation and clinical judgment of the Investigator, and may be terminated from the study. Dosing may also be modified based on tolerability as assessed with SSS scores.

Enrollment into Part A may be stopped and Part B initiated if there is a clear signal of activity based on the HAM-D scores and/or other scales being assessed. The study may be terminated if there is clear lack of activity based on HAM-D scores during Part A. A Data Review Team will assess the HAM-D and other data on an ongoing basis during Part A.

# **Inpatient Length of Stay and Discharge Instructions**

The minimum length of inpatient stay in both parts of this study is 7 days. It is the Investigator's responsibility to assess whether the subject can safely be discharged home and continue taking study drug administered by a healthcare professional trained on the protocol and delivery of the study drug for the rest of the treatment days (Days 8 to 14 for Parts A and B) or by returning to the clinic daily. The Investigator may decide to extend the subject's inpatient stay to maximize safety oversight. In making this assessment, the Investigator may consider not only the drug tolerability but also clinical factors including, but not limited to, availability of social support, transportation, severity of symptoms, and suicidality.

Discharge instructions must include warnings about avoiding activities for which sedative effects of the study drug may impair performance, such as driving a motor vehicle and operating machinery.

## Criteria for evaluation:

#### **Efficacy:**

Reduction of depressive symptoms will be assessed by the change from baseline at various time points in HAM-D total score; HAM-D response; HAM-D remission; change from baseline in the MADRS total score; CGI-I response; change from baseline in HAM-D subscale and individual item scores; change from baseline in HAM-A total score; change from baseline in SF-36; and change from baseline in FAs-D.

#### **Pharmacokinetics:**

Plasma samples will be collected to assay for concentrations of SAGE-217. The following PK parameters will be derived from the plasma concentrations (where evaluable): area under the concentration-time curve (AUC), AUC from time zero to infinity (AUC $_{\infty}$ ), maximum (peak) plasma concentration ( $C_{max}$ ), time at maximum (peak) plasma concentration ( $t_{max}$ ), steady-state drug concentration in the plasma during oral intake ( $C_{ss}$ ), and in the plasma at steady state during a dosing interval.

### Safety:

The safety and tolerability of SAGE-217 Oral Solution will be evaluated by frequency, type, and severity of adverse events; mean changes from baseline in clinical laboratory measures, vital signs, and ECGs; SSS score; physical examination; and suicidal ideation using the C-SSRS during both Part A and Part B.

## **Statistical methods:**

#### General

For the purpose of all safety and efficacy analyses where applicable, baseline is defined as the last measurement prior to the start of study drug administration.

Continuous endpoints will be summarized with n, mean, standard deviation, median, minimum, and maximum. In addition, change from baseline values will be calculated at each time point and summarized descriptively. For categorical endpoints, descriptive summaries will include counts and percentages.

## **Analysis Populations and Methods:**

The Safety Population (for both Part A and Part B), defined as all subjects administered study drug, will be used to provide descriptive summaries of safety data. Adverse events will be classified by type, incidence, severity, and causality. The overall incidence of adverse events will be summarized by Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Data for vital signs, clinical laboratory measurements, ECG, physical examinations, and concomitant medication usage will also be summarized. Safety data will be summarized and examined for possible relationships between subject characteristics and plasma SAGE-217 concentrations, as appropriate. Suicidality data collected using the C-SSRS at baseline and at each visit during the active Treatment Period will be listed for all subjects. The C-SSRS listings will include behavior type and/or category for suicidal ideation and suicidal behavior of the C-SSRS. Out-of-range safety endpoints may be categorized as low or high, where applicable. Subjects will be summarized according to treatment received.

The Efficacy Population (for both Part A and Part B), defined as all subjects in the Safety Population who complete at least 1 day of dosing of study drug and have at least one post-baseline efficacy evaluation, will be used to analyze efficacy data. Efficacy data will be analyzed using appropriate descriptive statistics and pre-specified statistical methods, as well as other data presentation methods where applicable; subject listings will be provided for all efficacy data. For (the open-label) Part A, efficacy data will be summarized descriptively. For Part B, subjects will be analyzed according to randomized treatment.

For Part B, the change from baseline in HAM-D total score will be analyzed using a mixed effects model for repeated measures (MMRM); the model will include treatment, baseline HAM-D total score, antidepressant use strata, assessment time point, and time point-by-treatment as explanatory variables. All post-baseline time points will be included in the model. The primary comparison will be between SAGE-217 Oral Solution and matching placebo at the 15-day time point. Model-based point estimates (ie, least squares [LS] means), 95% confidence intervals, and p-values will be reported. An unstructured covariance structure will be used to model the within-subject errors. Continuous variables will be analyzed using similar methods.

Binary efficacy endpoints, including responder and remission endpoints, will be analyzed using logistic regression model.

The PK Population will consist of all subjects in the Safety Population with sufficient plasma concentrations for PK evaluations, and will be used to summarize PK data. PK parameters will be summarized using appropriate descriptive statistics and listed by subject. The PK parameters to be summarized where possible will include  $AUC_{\infty}$ ,  $C_{max}$ ,  $t_{max}$ ,  $t_{1/2}$ , and  $C_{ss}$ .

#### Sample Size Calculation

The sample size of ten subjects for Part A was selected based on clinical and not statistical considerations.

For Part B, assuming a two-sided t-test at an alpha level of 0.10, a sample size of 23 subjects per group would provide 80% power to detect an effect size of 0.75 between the SAGE-217 Oral Solution and matching placebo groups with regard to the secondary efficacy outcome variable of change from baseline in HAM-D total score. An effect size of 0.75 corresponds to a matching placebo-adjusted difference of 7.5 points in the change from baseline in HAM-D total score at 15 days with an assumed SD of 10 points. By including two treatment groups and using a 1:1 randomization, a total of 46 subjects are required. Assuming a non-evaluability rate of 10%, up to 52 subjects will be randomized.

**Table 2:** Schedule of Events (Part A)

| | <b>Screening Period</b> | | | | | ( | Open-L | abel Tr | eatmen | t Perio | d | | | | | Follo | ow-up Po | eriod |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visits | OUTPATIENT | | | IN | PATIE | NT | | | | INPA | TIENT | or OU | TPATI | ENT | | OUTPATIENT | | |
| Visit Days | D-7 to D-1 | D1* | D2 | D3 | D4 | D5 | D6 | D7 | D8 | D9 | D10 | D11 | D12 | D13 | D14 | D15/<br>ET | D21<br>(+1d) | D28<br>(±3d) |
| Study Procedure | | | | | | | | | | | | | | | | | | |
| Informed Consent | X | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion | X | X | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | |
| Medical/Family History | X | | | | | | | | | | | | | | | | | |
| SCID-I | X | | | | | | | | | | | | | | | | | |
| Confinement | | | | | X | | | | | | | (X) | | | | | | |
| Physical Examination | X | | | | | | | | X | | | | | | | X | X | X |
| Body Weight/Height | X | | | | | | | | | | | | | | | X (wt<br>only) | X (wt only) | X (wt only) |
| Clinical Laboratory<br>Assessments | X | | | | | | | | X | | | | | | | X | X | X |
| Drug & Alcohol Screen | X | X | | | | | | | | | | | | | | | | |
| Pregnancy Test | X | X | | | | | | | | | | | | | | X | | X |
| Hepatitis & HIV Screen | X | | | | | | | | | | | | | | | | | |
| Blood Sample f | О | | | | | | | | О | | | | | | | О | | |
| Genetic Sample | 0 | | | | | | | | | | | | | | | | | |
| Vital Signs | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pulse Oximetry | | X | X | X | X | X | X | X | X | | | | | | | | | |
| 12-Lead ECG | X | X | X | | | | | X | | | | | | | X | | X | |
| C-SSRS <sup>j</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| CGI-S | X | X | X | X | | | | | X | | | | | | | X | X | X |

| | <b>Screening Period</b> | | | | | ( | Open-L | abel Tr | eatmen | nt Perio | d | | | | | Foll | ow-up P | eriod |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visits | OUTPATIENT | INPATIENT | | | | | | | | INPA | TIENT | | OUTPATIENT | | | | | |
| Visit Days | D-7 to D-1 | D1* | D2 | D3 | D4 | D5 | D6 | <b>D</b> 7 | D8 | D9 | D10 | D11 | D12 | D13 | D14 | D15/<br>ET | D21<br>(+1d) | D28<br>(±3d) |
| Study Procedure | | | | | | | | | | | | | | | | | | |
| CGI-I <sup>k</sup> | | | X | X | | | | | X | | | | | | | X | X | X |
| HAM-A <sup>k</sup> | X | X | X | X | | | | | X | | | | | | | X | X | X |
| HAM-D <sup>k</sup> | X | X | X | X | X | X | X | X | X | | | | | | | X | X | X |
| MADRS <sup>k</sup> | X | X | X | X | X | X | X | X | X | | | | | | | X | X | X |
| SSS | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Plasma PK | | | X | X | X | X | X | X | X | | | | | | X | X | | |
| Study Drug<br>Administration | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | |
| Adverse Events | | | | • | | • | • | • | X | | | • | | • | | | | |
| Prior/Concomitant<br>Medications | | | | | | | | | X | | | | | | | | | |

CGI-I = Clinical Global Impression - Improvement; CGI-S - Clinical Global Impression - Severity; C-SSRS = Columbia Suicide Severity Rating Scale; D = day; ET = early termination; ECG = electrocardiogram; HAM-A = Hamilton Anxiety Rating Scale; HAM-D = Hamilton Rating Scale for Depression, 17-item; HIV = human immunodeficiency virus; MADRS = Montgomery-Åsberg Depression Rating Scale; PK = pharmacokinetic; SCID-I = Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Axis I Disorders; SSS = Stanford Sleepiness Scale

- \*D1 procedures are to be completed prior to dosing
- <sup>a</sup> Outpatient visits may take place at the subject's residence or in the clinic.
- <sup>b</sup> Safety laboratory tests will include hematology, serum chemistry, coagulation, and urinalysis. Laboratory assessments are to be completed in the morning on Days 8 and 15 and during the follow-up visits on Day 21 and Day 28.
- <sup>c</sup> Urine toxicology for selected drugs of abuse and serum or breath test for alcohol.
- <sup>d</sup> Serum pregnancy test at screening and urine pregnancy test at Day 1 and Day 28.
- <sup>e</sup> Female subjects who prematurely discontinue will have a pregnancy test performed at the ET visit.
- f An optional blood sample for hormone and exploratory biochemistry testing, where consent is given.
- <sup>g</sup> An optional genetic sample for biomarker testing, where consent is given.
- h Vital signs include oral temperature (°C), respiratory rate, heart rate, and blood pressure (supine and standing). Vital signs will be obtained within ±5 minutes of the scheduled time point through 0.5 hours after dosing and ±30 minutes of the scheduled time point from 1 hour after dosing and greater, unless the subject is asleep between the hours of 23:00 h and 06:00 h. From Day 1 through Day 7, vital signs will be completed at the following time points: predose, 0.25, 0.5, 1, 2, and 12 hours after dosing. During the outpatient treatment period, vital signs will be completed prior to dosing and 1 hour after dosing. Vital signs may be repeated at the discretion of the Investigator or Visiting Home Healthcare Provider as clinically indicated.
- Will be performed 1 hour ±15 minutes after dosing on Days 1, 2, 7, and 14, and during the follow-up visit on Day 21.

- <sup>j</sup> The "Baseline/Screening" C-SSRS form will be completed at screening. The "Since Last Visit" C-SSRS form will be completed at any time of day at all subsequent time points.
- k To be completed to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28. The assessment timeframe for HAM-D and HAM-A scales will refer to the past 7 days (1 week) on Screening, Day 1, Day 15/ET, Day 21, and Day 28 visits, and the past 24 hours on visits occurring on Days 2 through 8.
- <sup>1</sup> To be completed within ±5 minutes of the scheduled time point through 0.5 hours after dosing and ±15 minutes of the scheduled time point from 1 hour after dosing and greater, unless the subject is asleep between 23:00 h and 06:00 h during the inpatient treatment period. From Day 1 through Day 7, SSS will be completed at the following time points: predose, 0.25, 0.5, 1, and 2 hours after dosing. During the outpatient treatment period, SSS will be completed prior to dosing and 1 hour after dosing.
- m Plasma samples for PK analysis in Part A and Part B will be collected predose on Days 2, 3, 4, 5, and 6, predose and 0.25, 0.5, 1, 2, 10, and 12 hours postdose on Day 7 (within ±5 minutes of the scheduled time point through 0.5 hours after dosing and ±15 minutes of the scheduled time point from 1 hour after dosing and greater), prior to discharge on Day 8 for subjects being discharged or 16 hours postdose for subjects remaining as inpatients, predose on Day 14, and in the morning on Day 15. The time of study drug administration is time zero and all post-dosing sampling times are relative to this time. In the event of a dose adjustment, an unscheduled PK sample should be collected just prior to the dose change. Plasma samples for PK analysis will be collected per protocol and subjects may need to be awoken for sample collection.
- <sup>n</sup> To include those taken within 30 days prior to informed consent and throughout the study.

 Table 3:
 Schedule of Events (Part B)

| | <b>Screening Period</b> | | Double-Blind, Placebo-Controlled Treatment Period | | | | | | | | | | Follow-up Period | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visits | OUTPATIENT | | | IN | PATIE | NT | | | INPATIENT or OUTPATIENT <sup>a</sup> | | | | | | | | OUTPATIENT | |
| Visit Days | D-7 to D-1 | D1* | D2 | D3 | D4 | D5 | D6 | <b>D7</b> | D8 | D9 | D10 | D11 | D12 | D13 | D14 | D15/<br>ET | D21<br>(+1d) | D28<br>(±3d) |
| Study Procedure | | | | | | | | | | | | | | | | | | |
| Informed Consent | X | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion | X | X | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | |
| Medical/Family History | X | | | | | | | | | | | | | | | | | |
| SCID-I | X | | | | | | | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | | | | | | | |
| Confinement | | | | | X | | | | | | | (X) | | | | | | |
| Physical Examination | X | | | | | | | | X | | | | | | | X | X | X |
| Body Weight/Height | X | | | | | | | | | | | | | | | X (wt<br>only) | X (wt<br>only) | X (wt<br>only) |
| Clinical Laboratory<br>Assessments | X | | | | | | | | X | | | | | | | X | X | X |
| Drug & Alcohol Screen | X | X | | | | | | | | | | | | | | | | |
| Pregnancy Test | X | X | | | | | | | | | | | | | | X | | X |
| Hepatitis & HIV Screen | X | | | | | | | | | | | | | | | | | |
| Blood Sample | О | | | | | | | | О | | | | | | | О | | |
| Genetic Sample | О | | | | | | | | | | | | | | | | | |
| Vital Signs | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pulse Oximetry | | X | X | X | X | X | X | X | X | | | | | | | | | |
| 12-Lead ECG | X | X | X | | | | | X | | | | | | | X | | X | |
| C-SSRS | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

| | <b>Screening Period</b> | | | | Doul | ole-Blin | d, Plac | ebo-Co | ntrolle | d Treat | ment P | eriod | | | | Foll | ow-up P | eriod |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visits | OUTPATIENT | | INPATIENT INPATIENT or OUTPATIENT a | | | | | | | | | | | | | OUTPATIENT | | |
| Visit Days | D-7 to D-1 | D1* | D2 | D3 | D4 | D5 | D6 | <b>D</b> 7 | D8 | D9 | D10 | D11 | D12 | D13 | D14 | D15/<br>ET | D21<br>(+1d) | D28<br>(±3d) |
| Study Procedure | | | | | | | | | | | | | | | | | | |
| CGI-S <sup>k</sup> | X | X | X | X | | | | | X | | | | | | | X | X | X |
| CGI-I <sup>k</sup> | | | X | X | | | | | X | | | | | | | X | X | X |
| HAM-A <sup>k</sup> | X | X | X | X | | | | | X | | | | | | | X | X | X |
| HAM-D <sup>k</sup> | X | X | X | X | X | X | X | X | X | | | | | | | X | X | X |
| MADRS <sup>k</sup> | X | X | X | X | X | X | X | X | X | | | | | | | X | X | X |
| SF-36 <sup>k</sup> | X | X | | | | | | | X | | | | | | | X | X | X |
| FAs-D <sup>k</sup> | X | X | | | | | | | X | | | | | | | X | X | X |
| SSS | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Plasma PK | | | X | X | X | X | X | X | X | | | | | | X | X | | |
| Study Drug<br>Administration | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | |
| Adverse Events | | | | | | | | | X | • | | | | | | | • | |
| Prior/Concomitant<br>Medications | | | | | | | | | X | | | | | | | | | |

CGI-I = Clinical Global Impression - Improvement; CGI-S - Clinical Global Impression - Severity; C-SSRS = Columbia Suicide Severity Rating Scale; D = day; ET = early termination; ECG = electrocardiogram; FAs-D = fatigue associated with depression; HAM-A = Hamilton Anxiety Rating Scale; HAM-D = Hamilton Rating Scale for Depression, 17-item; HIV = human immunodeficiency virus; MADRS = Montgomery-Åsberg Depression Rating Scale; PK = pharmacokinetic; SCID-I = Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Axis I Disorders; SF-36 = 36-item short form survey; SSS = Stanford Sleepiness Scale \*D1 procedures are to be completed prior to dosing

<sup>&</sup>lt;sup>a</sup> Outpatient visits may take place at the subject's residence or in the clinic.

<sup>&</sup>lt;sup>b</sup> Safety laboratory tests will include hematology, serum chemistry, coagulation, and urinalysis. Laboratory assessments are to be completed in the morning on Days 8 and 15 and during the follow-up visits on Day 21 and Day 28.

<sup>&</sup>lt;sup>c</sup> Urine toxicology for selected drugs of abuse and serum or breath test for alcohol.

<sup>&</sup>lt;sup>d</sup> Serum pregnancy test at screening and urine pregnancy test at Day 1 and Day 28.

<sup>&</sup>lt;sup>e</sup> Female subjects who prematurely discontinue will have a pregnancy test performed at the ET visit.

f An optional blood sample for hormone and exploratory biochemistry testing, where consent is given.

<sup>&</sup>lt;sup>g</sup> An optional genetic sample for biomarker testing, where consent is given.

- h Vital signs include oral temperature (°C), respiratory rate, heart rate, and blood pressure (supine and standing). Vital signs will be obtained within ±5 minutes of the scheduled time point through 0.5 hours after dosing and ±30 minutes of the scheduled time point from 1 hour after dosing and greater, unless the subject is asleep between the hours of 23:00 h and 06:00 h. From Day 1 through Day 7, vital signs will be completed at the following time points: predose, 0.25, 0.5, 1, 2, and 12 hours after dosing. During the outpatient treatment period, vital signs will be completed prior to dosing and 1 hour after dosing. Vital signs may be repeated at the discretion of the Investigator or Visiting Home Healthcare Provider as clinically indicated.
- Will be performed 1 hour ±15 minutes after dosing on Days 1, 2, 7, and 14, and during the follow-up visit on Day 21.
- <sup>j</sup> The "Baseline/Screening" C-SSRS form will be completed at screening. The "Since Last Visit" C-SSRS form will be completed at any time of day at all subsequent time points.
- k To be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28. The assessment timeframe for HAM-D and HAM-A scales will refer to the past 7 days (1 week) on Screening, Day 1, Day 15/ET, Day 21, and Day 28 visits, and the past 24 hours on visits occurring on Days 2 through 8.
- To be completed within ±5 minutes of the scheduled time point through 0.5 hours after dosing and ±15 minutes of the scheduled time point from 1 hour after dosing and greater, unless the subject is asleep between 23:00 h and 06:00 h during the inpatient treatment period. From Day 1 through Day 7, SSS will be completed at the following time points: predose, 0.25, 0.5, 1, and 2 hours after dosing. During the outpatient treatment period, SSS will be completed prior to dosing and 1 hour after dosing.
- m Plasma samples for PK analysis in Part A and Part B will be collected predose on Days 2, 3, 4, 5, and 6, predose and 0.25, 0.5, 1, 2, 10, and 12 hours postdose on Day 7 (within ±5 minutes of the scheduled time point through 0.5 hours after dosing and ±15 minutes of the scheduled time point from 1 hour after dosing and greater), prior to discharge on Day 8 for subjects being discharged or 16 hours postdose for subjects remaining as inpatients, predose on Day 14, and in the morning on Day 15. The time of study drug administration is time zero and all post-dosing sampling times are relative to this time. In the event of a dose adjustment, an unscheduled PK sample should be collected just prior to the dose change. Plasma samples for PK analysis will be collected per protocol and subjects may need to be awoken for sample collection.
- <sup>n</sup> To include those taken within 30 days prior to informed consent and throughout the study.

# 3. TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES

# **TABLE OF CONTENTS**

| 1. | TITLE PAGE | 1 |
|---|---|---|
| 2. | SYNOPSIS | 5 |
| 3. | TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES | 18 |
| 4. | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 23 |
| 5. | INTRODUCTION | 25 |
| 5.1. | Background of Major Depressive Disorders and Unmet Medical Need | 25 |
| 5.2. | SAGE-217 Oral Solution | 26 |
| 5.3. | Summary of Nonclinical and Clinical Experience with SAGE-217 | 26 |
| 5.3.1. | Nonclinical Studies with SAGE-217 | 26 |
| | | 26 |
| | | 28 |
| 5.5. | Dose Justification | 28 |
| 6. | STUDY OBJECTIVES AND PURPOSE | 29 |
| 6.1. | Part A | 29 |
| 6.1.1. | Primary Objective | 29 |
| 6.1.2. | Secondary Objective | 29 |
| 6.2. | Part B | 29 |
| 6.2.1. | Primary Objective | 29 |
| 6.2.2. | Secondary Objective | 29 |
| 6.3. | Pharmacokinetic Objective. | 29 |
| 6.4. | Endpoints | 29 |
| 6.4.1. | Part A | 29 |
| 6.4.1.1. | Primary | 29 |
| 6.4.1.2. | Secondary | 29 |
| 6.4.2. | Part B | 30 |
| 6.4.2.1. | Primary | 30 |
| 6.4.2.2. | Secondary | 30 |
| 7. | INVESTIGATIONAL PLAN | 31 |

| /.l. | Overall Study Design | 3 |
|---------|--------------------------------------------------------|----|
| 7.2. | Blinding and Randomization | 32 |
| 8. | SELECTION AND WITHDRAWAL OF SUBJECTS | 34 |
| 8.1. | Subject Inclusion Criteria | 32 |
| 8.2. | Subject Exclusion Criteria | 34 |
| 8.3. | Subject Withdrawal Criteria | 35 |
| 8.3.1. | Study Drug Withdrawal | 36 |
| 8.3.2. | Criteria for Study Termination | 36 |
| 9. | TREATMENT OF SUBJECTS | 37 |
| 9.1. | Number of Subjects | 37 |
| 9.2. | Treatment Assignment | 37 |
| 9.2.1. | Part A | 37 |
| 9.2.2. | Part B | 37 |
| 9.3. | Dose Adjustment Criteria | 37 |
| 9.4. | Prior/Concomitant Medications | 38 |
| 9.4.1. | Prior/Concomitant Medications | 38 |
| 9.4.2. | Restricted Medications | 38 |
| 9.5. | Treatment Compliance. | 39 |
| 10. | STUDY DRUG MATERIALS AND MANAGEMENT | 40 |
| 10.1. | Study Drug | 40 |
| 10.2. | Batch Formula for Stock SAGE-217 Oral Solution 6 mg/mL | 40 |
| 10.3. | Study Drug Packaging and Labeling | 40 |
| 10.4. | Study Drug Storage | 41 |
| 10.5. | Administration and Study Drug Accountability | 41 |
| 10.5.1. | Study Drug Administration | 42 |
| 10.5.2. | Study Drug Accountability | 42 |
| 10.6. | Study Drug Handling and Disposal | 42 |
| 11. | ASSESSMENT OF EFFICACY | 43 |
| 11.1. | Hamilton Rating Scale for Depression (HAM-D) | 43 |
| 11.2. | Montgomery-Åsberg Depression Rating Scale (MADRS) | 43 |
| 11.3. | Hamilton Anxiety Rating Scale (HAM-A) | 4 |
| 11.4. | Clinical Global Impression (CGI) | 44 |

| 11.5. | Short Form-36 (SF-36) | 45 |
|---|---|---|
| 11.6. | The Fatigue Associated With Depression (FAs-D) Patient-Reported Outcome (PRO) | 45 |
| 12. | PHARMACOKINETICS | 46 |
| 12.1. | Blood Sample Collection | 46 |
| 12.2. | Storage and Shipment of Pharmacokinetic Samples | 46 |
| 12.3. | Sample Analysis | 46 |
| 13. | ASSESSMENT OF SAFETY | 47 |
| 13.1. | Safety Parameters | 47 |
| 13.1.1. | Demographic/Medical History | 47 |
| 13.1.2. | Vital Signs | 47 |
| 13.1.3. | Weight and Height | 47 |
| 13.1.4. | Physical Examination | 47 |
| 13.1.5. | Electrocardiogram (ECG) | 47 |
| 13.1.6. | Laboratory Assessments | 47 |
| 13.1.6.1. | Hematology | 48 |
| 13.1.6.2. | Blood Chemistry | 48 |
| 13.1.6.3. | Urinalysis | 48 |
| 13.1.6.4. | Hormones and Exploratory Biochemistry | 48 |
| 13.1.6.5. | Virus Serology | 48 |
| 13.1.6.6. | Pregnancy Test | 49 |
| 13.1.6.7. | Genetic Testing | 49 |
| 13.1.6.8. | Drugs of Abuse and Alcohol | 49 |
| 13.1.7. | Columbia-Suicide Severity Rating Scale (C-SSRS) | 49 |
| 13.1.8. | Stanford Sleepiness Scale (SSS) | 50 |
| 13.2. | Adverse and Serious Adverse Events | 50 |
| 13.2.1. | Definition of Adverse Events | 50 |
| 13.2.1.1. | Adverse Event | 50 |
| 13.2.1.2. | Suspected Adverse Reaction. | 50 |
| 13.2.1.3. | Serious Adverse Event | 50 |
| 13.3. | Relationship to Study Drug | 51 |
| 13.4. | Recording Adverse Events | 51 |
| 13.5. | Reporting Adverse Events | 52 |

| 13.6. | Emergency Identification of Study Drug | 52 |
|---------|-------------------------------------------|----|
| 14. | STATISTICS | 54 |
| 14.1. | Data Analysis Sets | 52 |
| 14.1.1. | Analysis Populations and Methods | 54 |
| 14.2. | Handling of Missing Data | 52 |
| 14.3. | General Considerations | 52 |
| 14.4. | Demographics and Baseline Characteristics | 54 |
| 14.5. | Efficacy Analyses | 54 |
| 14.6. | Safety Analyses | 55 |
| 14.6.1. | Adverse Events | 56 |
| 14.6.2. | Clinical Laboratory Evaluations | 56 |
| 14.6.3. | Physical Examinations | 56 |
| 14.6.4. | Vital Signs | 56 |
| 14.6.5. | 12-Lead Electrocardiogram | 56 |
| 14.6.6. | Prior and Concomitant Medications | 56 |
| 14.6.7. | Columbia Suicide Severity Rating Scale | 57 |
| 14.6.8. | Stanford Sleepiness Scale | 57 |
| 14.7. | Pharmacokinetic Analyses | 57 |
| 14.8. | Determination of Sample Size | 57 |
| 14.9. | Changes From Protocol Specified Analyses | 57 |
| 15. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 58 |
| 15.1. | Study Monitoring | 58 |
| 15.2. | Audits and Inspections | 58 |
| 15.3. | Institutional Review Board (IRB) | 59 |
| 16. | QUALITY CONTROL AND QUALITY ASSURANCE | 60 |
| 17. | ETHICS | 61 |
| 17.1. | Ethics Review | 61 |
| 17.2. | Ethical Conduct of the Study | 61 |
| 17.3. | Written Informed Consent | 61 |
| 18. | DATA HANDLING AND RECORDKEEPING | 62 |
| 18.1. | Inspection of Records | 62 |
| 18.2 | Patention of Pacords | 60 |

| 18.3. | Confidentiality | 62 |
|---|---|---|
| 19. | PUBLICATION POLICY | 64 |
| 20. | LIST OF REFERENCES | 65 |
| 21. | APPENDICES | 67 |
| APPEND | IX 1. HAMILTON RATING SCALE FOR DEPRESSION, 17-ITEM (HAM-D) | 68 |
| APPEND | IX 2. MONTGOMERY-ÅSBERG DEPRESSION RATING SCALE (MADRS) | 85 |
| APPEND | IX 3. HAMILTON ANXIETY RATING SCALE (HAM-A) | 97 |
| APPEND | IX 4. CLINICAL GLOBAL IMPRESSION–IMPROVEMENT SCALE (CGI-I) AND SEVERITY SCALE (CGI-S) | 122 |
| APPEND | IX 5. SHORT-FORM 36 (SF-36) | 125 |
| APPEND | IX 6. THE FATIGUE ASSOCIATED WITH DEPRESSION (FAS-D) PATIENT-REPORTED OUTCOME (PRO) | 130 |
| APPEND | IX 7. COLUMBIA - SUICIDE SEVERITY RATING SCALE (C-SSRS) | 132 |
| APPEND | IX 8. STANFORD SLEEPINESS SCALE (SSS) | 140 |
| | LIST OF TABLES | |
| Table 1: | Emergency Contact Information | 4 |
| Table 2: | Schedule of Events (Part A) | 12 |
| Table 3: | Schedule of Events (Part B) | 15 |
| Table 4: | Abbreviations and Specialist Terms | 23 |
| Table 5: | Batch Formula for 125 mL of Stock SAGE-217 Oral Solution 6 mg/mL | 40 |

# 4. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

The following abbreviations and specialist terms are used in this study protocol.

**Table 4:** Abbreviations and Specialist Terms

| Abbreviation or Specialist Term | Explanation |
|---|---|
| AUC | area under the concentration-time curve |
| $\mathrm{AUC}_{\infty}$ | area under the concentration-time curve from time zero to infinity |
| BMI | body mass index |
| CGI-I | Clinical Global Impression - Improvement |
| CGI-S | Clinical Global Impression - Severity |
| C <sub>max</sub> | maximum (peak) plasma concentration |
| CS | clinically significant |
| $C_{ss}$ | steady-state drug concentration in the plasma during oral intake |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CYP450 | cytochrome P450 |
| DSM-5 | Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EP | European Pharmacopeia |
| FAs-D | fatigue associated with depression |
| GABA | γ-aminobutyric acid |
| GABA <sub>A</sub> | γ-aminobutyric acid-ligand gated chloride channel |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HAM-A | Hamilton Anxiety Rating Scale |
| HAM-D | 17-item Hamilton Rating Scale for Depression |
| HBsAg | hepatitis B surface antigen |
| HCV | hepatitis C virus |
| HIV | human immunodeficiency virus |
| НРβCD | hydroxypropyl-β-cyclodextrin |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |

| Abbreviation or Specialist Term | Explanation |
|---|---|
| IRB | Institutional Review Board |
| MAD | multiple-ascending dose |
| MADRS | Montgomery-Åsberg Depression Rating Scale |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MDD | major depressive disorders |
| MMRM | mixed effects model for reported measures |
| MTD | maximum tolerated dose |
| n | number |
| NCS | not clinically significant |
| NF | National Formulary |
| PK | pharmacokinetic(s) |
| PPD | postpartum depression |
| SAD | single-ascending dose |
| SCID-I | Structured Clinical Interview for DSM-5 Axis I Disorders |
| SD | standard deviation |
| SF-36 | 36-item short form survey |
| SOC | system organ class |
| SRC | Safety Review Committee |
| SSS | Stanford Sleepiness Scale |
| TEAE | treatment-emergent adverse event |
| t <sub>max</sub> | time at maximum (peak) plasma concentration |
| USP | United States Pharmacopeia |
| WHO | World Health Organization |
| WHO-DD | World Health Organization-Drug Dictionary |

## 5. INTRODUCTION

# 5.1. Background of Major Depressive Disorders and Unmet Medical Need

World Health Organization (WHO) has identified depression as the leading cause of disability worldwide, and a major contributor to the overall global burden of disease (<a href="http://www.who.int/mediacentre/factsheets/fs369/en/">http://www.who.int/mediacentre/factsheets/fs369/en/</a>). Globally, depression has been estimated to affect 350 million people.

In DSM-5, depression refers to an overarching set of diagnoses, including disruptive mood dysregulation disorder, major depressive disorder, persistent depressive disorder (dysthymia), premenstrual dysphoric disorder, substance/medication-induced depressive disorder, depressive disorder due to another medical condition, other specified depressive disorder, and unspecified depressive disorder.

In the US, the economic burden of depression, including workplace costs, direct costs and suicide-related costs, was estimated to be \$210.5 billion in 2010 (Greenberg 2015). As per WHO statistics, over 800,000 people die due to suicide every year, and suicide is the second leading cause of death in 15- to 29-year-olds. In the US, an estimated 10% to 15% of individuals with depression commit suicide (Angst 1999).

Antidepressants are mainstay of pharmacological treatment for depressive disorders. Selective serotonin reuptake inhibitors, serotonin and norepinephrine reuptake inhibitors, tricyclic antidepressants, monoamine oxidase inhibitors, and other compounds that affect monoaminergic neurotransmission, such as mirtrazapine and bupropion, represent the major classes of antidepressants. While antidepressants are widely used, large scale studies have demonstrated their limited efficacy. For example, in the STAR\*D trial where over 2800 patients were treated in "real world" settings, the HAM-D remission rate was 28% following 14 weeks of treatment with citalopram, a typical selective serotonin reuptake inhibitor (Trivedi 2006). Recent studies have shown a number of symptoms that remain untreated, such as cognitive impairment, sleep disturbances and anxiety, even in patients that are in remission over a long period of time after treatment (Conradi 2011; Romera 2013). A close examination of randomized placebo-controlled trials of antidepressants approved by the Food and Drug Administration in the treatment of both major or minor depressive disorders demonstrated Cohen's *d* effect sizes below 0.2 and high placebo response rates (Kirsch 2008; Fournier 2010), emphasizing the challenges in assessing antidepressant drug efficacy and the unmet need in the treatment of depression.

Converging preclinical and clinical evidence (Gerner 1981; Honig 1988; Drugan 1989; Luscher 2011; Mann 2014) implicates deficits in GABAergic neurotransmission in the pathophysiology of depressive disorders including MDD and PPD. Furthermore, several pieces of experimental data implicate deficiencies in the normal regulation of endogenous neuroactive steroids in depressive disorders (Maguire 2008; Maguire 2009). The neuroactive steroid class of compounds includes the endogenous neuroactive steroid, allopregnanolone. Allopregnanolone is a positive allosteric modulator of both synaptic and extrasynaptic GABA<sub>A</sub> receptors – the prominent inhibitory transmitter system in the brain. Depressed patients show low levels of GABA in the brain and of neurosteroids in the CSF and plasma, and antidepressant therapy

restores GABA levels in relevant animal models and neurosteroid concentrations in depressed patients (Luscher 2011; Schüle 2014).

# 5.2. SAGE-217 Oral Solution

The intended dosage form for oral administration is SAGE-217 Oral Solution to be compounded at the clinical pharmacy from components supplied by the Sponsor (SAGE-217 Drug Substance Powder in the Bottle, Excipients in the Bottle, and sucralose) and Sterile Water for Injection. SAGE-217 Oral Solution is a clear, colorless, aqueous hydroxypropyl-β-cyclodextrin (HPβCD) solution of SAGE-217 Drug Substance. One concentration, 6 mg/mL, is available for use in clinical studies. In addition to SAGE-217 Drug Substance, SAGE-217 Oral Solution contains HPβCD (MELLIC MELLIC MELLI

The SAGE-217 Oral Solution 6 mg/mL stock solution is compounded at point of use. This stock solution is for oral administration after dilution to the intended dose by the clinical pharmacy.

# 5.3. Summary of Nonclinical and Clinical Experience with SAGE-217

#### 5.3.1. Nonclinical Studies with SAGE-217

In nonclinical studies of SAGE-217, sedative-hypnotic effects were consistently observed at higher doses in both in vivo pharmacology studies and toxicology studies. The sedative-hypnotic impairments seen with SAGE-217 were typical for GABAA positive allosteric modulators, ranging from hyperexcitability and ataxia at the lower doses through deep sedation and ultimately anesthesia at higher doses. Depth and duration of sedation demonstrated a clear dose response over the range tested, with evidence of tolerance occurring with continued exposure. Tolerance to the effects of SAGE-217 on motor incoordination was not observed after 7 days of dosing.

The compound has been assessed in 14-day rat and dog toxicology studies with daily administration of SAGE-217 as a solution in HPβCD in dogs and Labrasol® in rats. The no-observed-adverse-effect-level was 3 mg/kg (females) and 22.5 mg/kg (males) in rats and 2.5 mg/kg in dogs. There were no adverse effects in dogs or rats in the main toxicology studies. A single observation of mortality occurred in one female rat at the high dose in a toxicokinetic study that was suspected to have been related to exaggerated pharmacology. Additional toxicology and pharmacology information is provided in the Investigator's Brochure.







# 5.5. Dose Justification

To date, the pharmacokinetics of SAGE-217 Oral Solution has been investigated in healthy volunteers within the context of the SAD and MAD studies (217-CLP-101 and 217-CLP-102, respectively). The MTD was determined to be 55 mg in the SAD study and 30 mg once daily (either AM or PM dosing) in the MAD study. Thus as a first step, while ensuring tolerability, a 30 mg dose has been chosen to maximize the potential therapeutic benefit in this first clinical study of MDD.

## 6. STUDY OBJECTIVES AND PURPOSE

## **6.1.** Part A

## 6.1.1. Primary Objective

The primary objective of the study is to evaluate the safety and tolerability of SAGE-217 Oral Solution 30 mg.

# **6.1.2.** Secondary Objective

The secondary objective of Part A is to determine if treatment with SAGE-217 Oral Solution 30 mg for 14 days reduces depressive symptoms.

# **6.2.** Part B

# **6.2.1.** Primary Objective

The primary objective of the study is to evaluate the safety and tolerability of SAGE-217 Oral Solution 30 mg.

# **6.2.2.** Secondary Objective

The secondary efficacy objective for Part B of the study is to determine if treatment with SAGE-217 Oral Solution 30 mg reduces depressive symptoms in subjects with moderate to severe MDD compared to matching placebo.

# 6.3. Pharmacokinetic Objective

The PK objective of Part A and Part B is to assess the PK profile of SAGE-217 Oral Solution in plasma samples.

# 6.4. Endpoints

#### 6.4.1. Part A

# **6.4.1.1.** Primary

The primary endpoint is the safety and tolerability of SAGE-217 as assessed by the frequency and severity of adverse events; changes from baseline in clinical laboratory measures, vital signs, and electrocardiograms (ECGs); Stanford Sleepiness Scale (SSS) score; physical examination; and suicidal ideation using the Columbia-Suicide Severity Rating Scale (C-SSRS).

## **6.4.1.2. Secondary**

Reduction in depressive symptoms as assessed by the following:

• Change from baseline in HAM-D total score at all time points;

- HAM-D response (defined as having a 50% or greater reduction from baseline in HAM-D total score);
- HAM-D remission (defined as having a HAM-D total score of  $\leq 7$ );
- Change from baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score at all time points;
- Change from baseline in HAM-D subscale and individual item scores at all time points;
- Change from baseline in Hamilton Anxiety Rating Scale (HAM-A) total score at all time points; and
- Clinical Global Impression Improvement (CGI-I) response (defined as a CGI-I score of "very much improved" or "much improved").

#### 6.4.2. Part B

# **6.4.2.1.** Primary

The primary endpoint is the safety and tolerability of SAGE-217 as assessed by the frequency and severity of adverse events; changes from baseline in clinical laboratory measures, vital signs, and ECGs; SSS score; physical examination; and suicidal ideation using the C-SSRS.

# **6.4.2.2.** Secondary

Reduction in depressive symptoms, compared to placebo, as assessed by the following:

- Change from baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D) total score at all time points;
- HAM-D response;
- HAM-D remission:
- Change from baseline in the MADRS total score at all time points;
- Change from baseline in HAM-D subscale and individual item scores at all time points;
- Change from baseline in HAM-A total score at all time points;
- CGI-I response; and
- 36-item short form survey (SF-36) and fatigue associated with depression (FAs-D) patient-reported outcome.

# 7. INVESTIGATIONAL PLAN

# 7.1. Overall Study Design

This study is a two-part, multicenter, Phase 2a study to evaluate the safety, tolerability, PK, and efficacy of SAGE-217 Oral Solution in approximately 62 adult subjects with MDD. Part A of the study is an open-label design with SAGE-217 Oral Solution dosing for 14 days. Part B of the study is a randomized, double-blind, parallel-group, placebo-controlled design with SAGE-217 Oral Solution or matching placebo dosing for 14 days. Separate cohorts of subjects will be enrolled in Part A and Part B; subjects participating in Part A cannot enroll in Part B.

Parts A and B of the study will consist of an up to 7-day Screening Period (Days -7 to -1), a 14-day Treatment Period, and a 2-week Follow-up Period (through Day 28).

During the Screening Period (Day -7 to Day -1), after signing the informed consent form (ICF), subjects will be assessed for study eligibility, and the severity of each subject's MDD will be evaluated using HAM-D. The Screening Period assessments will be conducted on an outpatient basis.

If applicable, standard of care data collected prior to obtaining informed consent may also be included as screening data, if appropriate, such as laboratory tests, ECG, physical examination, and vital signs conducted within the preceding 48 hours, as long as the requirement for the screening assessment to be collected retrospectively is met in full. If applicable, to ensure protocol compliance, any standard of care data eligible for inclusion as screening data must include the precise nature and timing of data collection.

During the 14-day study Treatment Period of Parts A and B, subjects must remain inpatient for the first 7 days at minimum and per Investigator's judgement thereafter. The Follow-up Period assessments will be conducted on an outpatient basis.

The study will be conducted in two parts:

- Part A: Beginning on Day 1, subjects will receive open-label SAGE-217 Oral Solution at 8:00 PM (±15 minutes) with food (as outlined in Section 9.2.1). Subjects will receive SAGE-217 Oral Solution 30 mg from Day 1 to Day 14 as tolerated.
- Part B: Based on the results of Part A, eligible subjects will be stratified based on use of antidepressant treatment (current/stable or not treated/withdrawn ≥30 days) and randomized within each stratum in a 1:1 fashion to receive SAGE-217 Oral Solution or matching placebo for 14 days beginning on Day 1 as tolerated. All doses of study drug will be administered at 8:00 PM (±15 minutes) with food as outlined in Section 9.2.2.

Enrollment into Part A may be stopped and Part B initiated if there is a clear signal of activity based on the HAM-D scores and/or other scales being assessed. Alternatively, upon completion of Part A, Part B may begin. The study may be terminated if there is clear lack of activity based on HAM-D scores during Part A.

In Part A and Part B, study drug (SAGE-217 Oral Solution or matching placebo) will be administered at the study center for at least the first 7 days of the Treatment Period, which

includes Day 1 of study drug administration through completion of study drug administration on Day 14. Subjects may be discharged after a minimum 7-day inpatient stay, following completion of the Day 7 assessments. If their clinical condition does not allow discharge, the Investigator may keep the subjects as inpatients for a longer period of time. Subjects discharged from the inpatient unit may receive treatment with study drug for the remainder of the 14-day Treatment Period as outpatients. For the outpatient phase, dosing will be done at the clinical site or, if suitable arrangements can be made, via home administration where local regulations allow. Home administration of study drug will be performed according to a site-specific plan by a healthcare professional trained on the protocol and delivery of the study drug.

Subjects will be monitored for safety during the Treatment and Follow-up Periods including monitoring for adverse events/serious adverse events, routine clinical laboratory assessments, physical examination, vital signs, and ECG.

During the Treatment Period, subjects will be able to receive study drug as long as there are no dose-limiting safety/tolerability concerns. Subjects who experience moderate or severe adverse events that according to the clinical judgement of the Investigator are related to study drug while receiving the 30 mg dose of study drug will receive 20 mg for the remaining of the Treatment Period. Subjects who experience moderate or severe related adverse events while receiving the 20 mg dose of study drug may not be able to continue receiving study drug based on the evaluation and clinical judgment of the Investigator, and may be terminated from the study.

Dosing may also be modified based on tolerability as assessed with SSS scores. Any SSS score of  $\geq 6$  will be reassessed within 10 minutes. If a subject is receiving the 30 mg dose of study drug and has an SSS score of  $\geq 6$  that is confirmed on repeat assessment during normal waking hours, the dose will be decreased to 20 mg for the rest of the Treatment Period. If a subject is receiving the 20 mg dose of study drug and has an SSS score of  $\geq 6$  that is confirmed on repeat assessment during normal waking hours, then study drug will be discontinued and the subject will be terminated from the study.

# 7.2. Blinding and Randomization

Part A is open-label with no control group; therefore, there will be no randomization or blinding.

Part B is a double-blind, placebo-controlled study. Subjects who meet the entrance criteria will be stratified based on use of antidepressant treatment (current/stable or not treated/withdrawn ≥30 days) and randomly assigned within each stratum in a 1:1 ratio to receive SAGE-217 Oral Solution or taste-matched placebo according to a computer-generated randomization schedule. Once it has been determined that a subject meets eligibility criteria, the subject will be sequentially assigned a subject number from the randomization schedule provided to the unblinded pharmacist. Subject identification numbers will consist of the site number (eg, "01") followed by numbering starting with double zero (eg, 01-001, 01-002, 01-003 through 01-062).

The randomization schedule will be generated using SAS V9.2 or later. Only the clinic pharmacist or designated pharmacy staff, who is responsible for preparing the solutions, will be given a copy of the randomization schedule. In the event of a medical emergency, the pharmacist may reveal actual solution contents to the Investigator, who should also alert Sage of the emergency (see Section 13.6 for more details related to unblinding). In all cases where the study drug allocation for a subject is unblinded, pertinent information (including the reason for

unblinding) must be documented in the subject's records and on the electronic case report form (eCRF). If the subject or study center personnel (other than pharmacist) have been unblinded, the subject will be terminated from the study. In addition, an unblinded Monitor will perform drug accountability during the study.

## 8. SELECTION AND WITHDRAWAL OF SUBJECTS

# 8.1. Subject Inclusion Criteria

The following inclusion criteria must be met for individuals to be eligible for the study.

- 1. Subject has signed an ICF prior to any study-specific procedures being performed.
- 2. Subject is an ambulatory male or female between 18 and 65 years of age, inclusive.
- 3. Subject is in good physical health and has no clinically significant findings, as determined by the Investigator, on physical examination, 12-lead ECG, or clinical laboratory tests.
- 4. Subject agrees to adhere to the study requirements.
- 5. Subject has a diagnosis of MDD that has been present for at least a 4-week period as diagnosed by Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Axis I Disorders (SCID-I).
- 6. Subject has a HAM-D total score of ≥22 at screening and Day 1 (prior to dosing).
- 7. Subject has a HAM-A total score of ≥20 at screening and Day 1 (prior to dosing) (Part B only).
- 8. Subject is willing to delay start of other antidepressant or antianxiety medications and any new pharmacotherapy regimens, including as-needed benzodiazepine anxiolytics, during the screening and treatment periods.
- 9. Subject agrees to practice an acceptable method of highly effective birth control at screening and throughout study participation. Highly effective methods of birth control include sexual abstinence (for males and females); vasectomy; or a condom with spermicide in combination with a highly effective female partner's method (for males); and hormonal methods of contraception (ie, established use of oral, implantable, injectable, or transdermal hormones); placement of an intrauterine device; placement of an intrauterine system; and mechanical/barrier method of contraception (ie, condom or occlusive cap [diaphragm or cervical/vault cap] in conjunction with spermicide [foam, gel, film, cream, or suppository]) (for females).

# 8.2. Subject Exclusion Criteria

Subjects will be excluded if they meet any of the following exclusion criteria.

- 1. Subject has a history of suicide attempt.
- 2. Subject has a recent history or active clinically significant manifestations of metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, musculoskeletal, dermatological, urogenital, neurological, or eyes, ears, nose, and throat disorders, or any other acute or chronic condition that, in the Investigator's opinion, would limit the subject's ability to complete or participate in this clinical study.

- 3. Subject has a history of treatment-resistant depression, defined as persistent depressive symptoms despite treatment with adequate doses of antidepressants from two different classes for an adequate amount of time (ie, at least 4 weeks of treatment).
- 4. Subject has a known allergy to SAGE-217, allopregnanolone, or related compounds.
- 5. Subject has a positive pregnancy test at screening or on Day 1 prior to the start of study drug administration.
- 6. Subject has detectable hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV), or human immunodeficiency virus (HIV) antibody at screening.
- 7. Subject has active psychosis per Investigator assessment.
- 8. Subject has a medical history of seizures.
- 9. Subject has a medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder.
- 10. Subject has a history of alcohol or drug dependence (including benzodiazepines) in the 12 months prior to screening.
- 11. Subject has had exposure to another investigational medication or device within 30 days prior to screening.
- 12. Subject has been treated or randomized in this study (eg, Part A) or any other study employing SAGE-217 previously (ie, subject may not have received study drug and then re-enroll).
- 13. Subject has had administration of psychotropics that have been initiated within 14 days prior to screening and/or are not being taken at a stable dose.
- 14. Use of any known strong inhibitors and/or inducers of CYP3A4 within the 14 days or five half-lives (whichever is longer) or consumed grapefruit juice, grapefruit, Seville oranges, or St. John's Wort or products containing these within 30 days prior to receiving the first dose of study drug.
- 15. Subject has a positive drug and/or alcohol screen at screening or on Day 1 prior to dosing.

# 8.3. Subject Withdrawal Criteria

If there is an adverse event or medical reason for the withdrawal, the subject should be followed medically until the condition has either resolved or is stable. Details of the reason for withdrawal should be recorded in the subject's eCRF.

Subjects who withdraw should, if possible, have a follow-up examination, including a physical examination, the appropriate investigations, vital signs, and clinical laboratory tests (including pregnancy tests), as outlined for the Day 15 visit (Table 2 and Table 3). All details of this follow-up examination should be recorded in the subject's medical source documents.

# 8.3.1. Study Drug Withdrawal

Participation in the study is strictly voluntary. Subjects are free to discontinue the study at any time without giving their reason(s).

A subject must be withdrawn from the study treatment in the event of any of the following:

- Withdrawal of the subject's consent;
- New onset of a condition that would have met exclusion criterion, is clinically relevant and affects the subject's safety, and discontinuation is considered necessary by the Investigators and/Sponsor;
- Occurrence of intolerable adverse events;
- Occurrence of pregnancy;
- Intake of nonpermitted concomitant medication;
- Subject noncompliance;
- Significant protocol deviation determined in consultation with the Medical Monitor.

If a subject failed to attend scheduled assessments during the course of the study, the Investigators must determine the reasons and the circumstances as completely and accurately as possible and document this in the subject's source documents.

Subjects may be withdrawn from the study if there is concern for the subject's safety or it is determined that the subject is no longer a qualified participant. Subjects who withdraw should, if possible, have a follow-up examination, including a physical examination, the appropriate investigations, vital signs, and clinical laboratory tests (including pregnancy tests), as outlined for the Day 15 visit (Table 2 and Table 3). All details of this follow-up examination should be recorded in the subject's medical source documents.

Subjects who withdraw or are withdrawn from the study will be replaced only if they withdraw prior to dosing. Subjects who are withdrawn from the study, fail to return or are no longer qualified will not be replaced.

## **8.3.2.** Criteria for Study Termination

Sage Therapeutics may terminate this study or any portion of the study at any time for safety reasons, including the occurrence of adverse events or other findings suggesting unacceptable risk to subjects, or for administrative reasons. In the event of study termination, Sage Therapeutics will provide written notification to the Investigator. Investigational sites must promptly notify their Institutional Review Board (IRB) and initiate withdrawal procedures for participating subjects.
#### 9. TREATMENT OF SUBJECTS

## 9.1. Number of Subjects

Approximately ten subjects with MDD will be enrolled into Part A of the study. Up to 52 subjects may be randomized in Part B to ensure at least 46 evaluable subjects for Part B. Evaluable subjects are defined as those subjects receiving study drug with at least one post-baseline HAM-D assessment.

# 9.2. Treatment Assignment

Study drug will be administered with food in both the inpatient and outpatient treatment periods. Food intake will be standardized as specified by the Sponsor.

#### 9.2.1. Part A

Subjects participating in Part A of the study will take study drug (SAGE-217) in an open-label manner. Subjects will be administered a 30 mg dose of study drug at 8:00 PM ( $\pm 15$  minutes) with food for 14 days (Day 1 to Day 14) as tolerated.

#### 9.2.2. Part B

Subjects participating in the randomized, double-blind, placebo-controlled portion of the study (Part B) will be randomly assigned to receive SAGE-217 Oral Solution 30 mg or matching placebo solution on a 1:1 basis according to a computer-generated randomization schedule; the randomization schedule will be stratified to allow for treatment balance within each use of antidepressant stratum.

Subjects, clinicians, and study team will be blinded to treatment allocation. The pharmacist, who will prepare the oral solutions according to the randomization schedule, and an unblinded Monitor, who will perform drug accountability during the study, will be unblinded.

# 9.3. Dose Adjustment Criteria

During the Treatment Period, subjects will be able to receive study drug as long as there are no dose-limiting safety/tolerability concerns.

In both Part A and Part B, subjects who experience moderate or severe adverse events that according to the clinical judgement of the Investigator are related to study drug while receiving the 30 mg dose of study drug will receive 20 mg for the remaining of the Treatment Period. Subjects who experience moderate or severe related adverse events while receiving the 20 mg dose of study drug may not be able to continue receiving study drug based on the evaluation and clinical judgment of the Investigator, and may be terminated from the study.

Dosing may also be modified based on tolerability as assessed with SSS scores. Any SSS score of  $\geq 6$  will be reassessed within 10 minutes. If a subject is receiving the 30 mg dose of study drug and has an SSS score of  $\geq 6$  that is confirmed on repeat assessment during normal waking hours, the dose will be decreased to 20 mg for the rest of the Treatment Period. If a subject is receiving the 20 mg dose of study drug and has an SSS score of  $\geq 6$  that is confirmed on repeat

assessment during normal waking hours, then study drug will be discontinued and the subject will be terminated from the study.

Enrollment into Part A may be stopped and Part B initiated if there is a clear signal of activity based on the HAM-D scores and/or other scales being assessed. The study may be terminated if there is clear lack of activity based on HAM-D scores during Part A. A Data Review Team will assess the HAM-D and other data on an ongoing basis during Part A.

#### 9.4. Prior/Concomitant Medications

#### 9.4.1. Prior/Concomitant Medications

Subjects will receive standard of care for adult patients diagnosed with moderate to severe MDD. Psychotropic medications, which must have been initiated at least 14 days prior to screening, must remain at a stable dose until completion of the Day 15 assessments (Parts A and B).

Eligible subjects will be stratified based on use of antidepressant treatment (current/stable or not treated/withdrawn ≥30 days) and randomly assigned within each stratum in a 1:1 ratio to receive SAGE-217 Oral Solution or taste-matched placebo.

In this study, psychotropic medications refer to central nervous system active medications taken to help depressive symptoms, and include antidepressants, benzodiazepines, and hypnotic agents. Subjects presenting to the study on antidepressants may be eligible to participate if they have been on a stable dose for at least 14 days. Those subjects on benzodiazepines and hypnotic agents may be considered for eligibility based on specific discussions between the Investigator and the Sponsor to ensure safety. Subjects on other psychotropic medications, including stimulants, antipsychotics, and mood stabilizers, are not eligible to participate in this study.

Any concomitant medication determined necessary for the welfare of the subject may be given at the discretion of the Investigator at any time during the study under the guidance outlined in Section 9.4.2. In both Part A and Part B, all medications should be documented throughout the study from 30 days prior to signing the ICF through Day 28 (±3 days) and recorded on the eCRF. Prior medications (ie, those taken prior to signing of ICF) that required washout for study entry will also be documented.

#### 9.4.2. Restricted Medications

Restrictions on specific classes of medications include the following:

- Initiation of new antidepressant therapy is prohibited upon admission to the study center for those eligible subjects who desire study participation. Those subjects already taking an antidepressant at the time of study entry (and meeting all study inclusion criteria) will be permitted to remain on the pre-existing antidepressant at their current dose if they were on this medication for at least 14 days prior to study enrollment.
- Benzodiazepines are to be avoided as much as possible. Eligible subjects taking a stable dose of benzodiazepine for at least 14 days prior to the study will be discussed on a case-by-case basis with the Sponsor to determine eligibility. Subjects may be permitted to continue to take their current dose of the benzodiazepine (to prevent

acute withdrawal), but no new benzodiazepine use will be permitted during the course of the study.

- The use of hypnotics for sleep/insomnia such as Ambien® and trazodone is to be avoided; use of hypnotics will be discussed on a case-by-case basis with the Sponsor.
- Anticonvulsants and atypical antipsychotics are prohibited.

## 9.5. Treatment Compliance

Investigational product will be prepared by the site pharmacist. The Investigator(s) or designee will record the time and dose of study drug administration in the source documents. Any reasons for noncompliance will also be documented, including:

- Missed visits;
- Interruptions in the schedule of administration; and
- Nonpermitted medications.

The time at which study procedures are conducted should follow the protocol timelines as closely as possible.

#### 10. STUDY DRUG MATERIALS AND MANAGEMENT

# 10.1. Study Drug

SAGE-217 Oral Solution is available as a 6 mg/mL stock aqueous solution of SAGE-217 Drug Substance containing 40% HPβCD and 0.0025% sucralose, which is further diluted with Sterile Water for Injection to achieve the selected dose. The 6 mg/mL stock SAGE-217 Oral Solution will be compounded from SAGE-217 Drug Substance Powder in the Bottle and Excipient (s) in the Bottle (manufactured under current Good Manufacturing Practice [GMP] conditions and further admixed at the clinical site in preparation for dosing.

A matching placebo oral solution will be prepared for administration without the active ingredient, but including the HP $\beta$ CD and sucralose, as well as three taste-masking components to preserve the blinding. Detailed instructions for study drug (SAGE-217 Oral Solution 30 mg and matching placebo) preparation will be provided in the Pharmacy Manual.

## 10.2. Batch Formula for Stock SAGE-217 Oral Solution 6 mg/mL

Each bottle of SAGE-217 Oral Solution 6 mg/mL will be compounded at the clinical pharmacy from components manufactured and supplied by the Sponsor per the directions provided in the Pharmacy Manual. The batch formula for a 125 mL solution of the 6 mg/mL stock solution is shown in Table 5.

| Table 5: | Batch Formula for 125 mL of Stock SAGE-217 Oral Solution 6 mg/mL |
|----------|------------------------------------------------------------------|
|----------|------------------------------------------------------------------|

| Ingredient | Compendia Specification | Concentration (mg/mL) | Amount (mg/Bottle) |
|---|---|---|---|
| SAGE-217 | not applicable | 6 | 750 |
| НРВСО | USP/EP | 457 | 57,100 |
| Sucralose | USP/NF | 0.025 | 3.124 |
| Water for Injection | USP | not applicable | 85,650 |

Abbreviations: EP = European Pharmacopeia; HPβCD = hydroxypropyl-β-cyclodextrin; NF = National Formulary; USP = United States Pharmacopeia

Additional excipients will be utilized in matching placebo to match the taste of SAGE-217 Oral Solution. They include sucrose octaacetate, tannic acid, and ammonium glycyrrhizate. The quantities of these excipients will vary depending on the dose of SAGE-217 to match the taste of each individual dose.

# 10.3. Study Drug Packaging and Labeling

The composition and pharmaceutical quality of the investigational product will be maintained according to the current GMP and Good Clinical Practice (GCP) guidelines and available for review in the study medication documentation. Study drug will be provided to the site as powder in the bottle and excipient(s) in the bottle units to be compounded in the pharmacy at a volume of 125 mL of a 6 mg/mL stock solution and then further diluted to approximately 40 mL at the identified doses. The taste-matching excipients will be provided to the clinical pharmacies via

suitable suppliers or can be ordered directly by the clinical pharmacies. Study drug labels with all required information and conforming to all applicable Code of Federal Regulations and GMP/GCP guidelines will be prepared by the clinical research organization.

## 10.4. Study Drug Storage

Upon receipt of study drug, the Investigator or designee will inspect the materials and complete and return the acknowledgment of receipt form enclosed with the parcel. A copy of the signed receipt will be kept in the study files.

The study drug materials must be carefully stored at the temperature specified in the Pharmacy Manual (eg, clinical dosing solutions stored at approximately 2 to 8°C for 11 days with room temperature excursions allowed for up to 24 hours after preparation), safely and separately from other drugs. The study drug may not be used for any purpose other than the present study. After the study is completed, all unused study drug must be retained, returned as directed, or destroyed on site per the Sponsor's instructions.

The Investigator or designee will be responsible for ensuring appropriate storage, compounding, dispensing, inventory, and accountability of all clinical supplies. An accurate, timely record of the disposition of all clinical supplies must be maintained. The supplies and inventory must be available for inspection by the designated representatives of the Sponsor or the Sponsor's representatives on request, and must include the information below:

- The identification of the subject to whom the drug was dispensed;
- The date(s) and quantity of the drug dispensed to the subject; and
- The product lot/batch number.

The preparation of the study drugs must be documented on a 'Drug Preparation and Dispensing Log Form' or similar form.

The drug inventory and any clinical supplies that have been destroyed must be documented. This documentation must include at least the information below or as agreed with the Sponsor:

- The number of prepared units;
- The number of administered units;
- The number of unused units;
- The number of units destroyed at the end of the study;
- The date, method, and location of destruction.

# 10.5. Administration and Study Drug Accountability

Doses will be prepared as an approximate 40 mL oral solution to be swallowed all at once, followed by approximately 200 mL of water that has been used to rinse the dosing bottle. The start time of swallowing the approximately 40 mL oral solution is time zero for all assessments. Subjects may have assistance from the clinic staff when taking the study drug.

#### 10.5.1. Study Drug Administration

While confined in the clinical unit (at least Day 1 through Day 7 of Part A and Part B), subjects will receive study drug at 8:00 PM (±15 minutes) with food.

Food intake will be standardized as specified by the Sponsor. Subjects who experience moderate or severe related adverse events while receiving study drug may not be able to continue receiving study drug based on the evaluation and clinical judgment of the Investigator, and may be terminated from the study.

Subjects may be discharged after a minimum 7-day inpatient stay, following completion of the Day 7 assessments. If their clinical condition does not allow discharge, the Investigator may keep the subjects as inpatients for a longer period of time.

For non-confinement days (Days 8 through 14 of Parts A and B), dosing will be done at the clinical site or, if suitable arrangements can be made, via home administration where local regulations allow. Home administration of study drug will be performed according to a site-specific plan by a healthcare professional trained on the protocol and delivery of the study drug.

### 10.5.2. Study Drug Accountability

The study drug provided is for use only as directed in this protocol.

The Investigator or designee must maintain a record of all study drug received, used, and discarded. It must be clear from the records which subject received which dose of active or matching placebo treatment.

The Sponsor will be permitted access to the study supplies at any time within usual business hours and with appropriate notice during or after completion of the study to perform drug accountability reconciliation. Only unblinded personnel will be able to access the study drug and accountability documentation from first dosing through database hard lock.

# 10.6. Study Drug Handling and Disposal

The pharmacist or designee for drug accountability is to document the date and time of initial compounding, subsequent admixture of dosing solutions, administration of test article, and for which subject the study drug was intended (ie, record subject initials and birth date or other unique identifier).

At the end of the study, any unused study drug will be retained or returned to the Sponsor for destruction or destroyed locally per the Sponsor's directions. The disposition of study drug will be documented.

#### 11. ASSESSMENT OF EFFICACY

# 11.1. Hamilton Rating Scale for Depression (HAM-D)

The primary outcome measure in Part B will be the change from baseline in 17-item HAM-D total score at the end of the Treatment Period (Day 15). The HAM-D will be administered before, during, and after the administration of open-label (Part A) and blinded (Part B) study drug.

The 17-item HAM-D will be used to rate the severity of depression in subjects who are already diagnosed as depressed (Williams 2013a; Williams 2013b). The 17-item HAM-D comprises individual ratings related to the following symptoms: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. The HAM-D assessments are to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28. Every effort should be made for the same rater to perform all HAM-D assessments for an individual subject.

The HAM-D total score will be calculated as the sum of the 17 individual item scores. Item 16 can be rated according to history (item 16A) or actual weight change (item 16B). The item 16 score is calculated as the item 16 response that is not equal to 3 (ie, "Not assessed").

In addition to the primary efficacy endpoint of change from baseline in HAM-D total score (Part B), several secondary efficacy endpoints will be derived for the HAM-D. Hamilton Rating Scale for Depression subscale scores will be calculated as the sum of the items comprising each subscale. Hamilton Rating Scale for Depression response will be defined as having a 50% or greater reduction from baseline in HAM-D total score. Hamilton Rating Scale for Depression remission will be defined as having a HAM-D total score of ≤7. A copy of the HAM-D is provided in Appendix 1.

# 11.2. Montgomery-Åsberg Depression Rating Scale (MADRS)

The MADRS is a 10-item diagnostic questionnaire that psychiatrists use to measure the severity of depressive episodes in subjects with mood disorders. It was designed as an adjunct to the HAM-D that would be more sensitive to the changes brought on by antidepressants and other forms of treatment than the Hamilton Scale.

The MADRS assessments are to be completed at 8:00 AM ( $\pm 30$  minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28.

Higher MADRS scores indicate more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60 (Williams 2008).

The questionnaire includes questions on the following symptoms:

- 1. Apparent sadness
- 2. Reported sadness

- 3. Inner tension
- 4. Reduced sleep
- 5. Reduced appetite
- 6. Concentration difficulties
- 7. Lassitude
- 8. Inability to feel
- 9. Pessimistic thoughts
- 10. Suicidal thoughts

The MADRS total score will be calculated as the sum of the 10 individual item scores. A copy of the MADRS is provided in Appendix 2.

## 11.3. Hamilton Anxiety Rating Scale (HAM-A)

The 14-item HAM-A will be used to rate the severity of symptoms of anxiety (Williams 2013c; Williams 2013d). Each of the 14 items is defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scoring for HAM-A is calculated by assigning scores of 0 (not present) to 4 (very severe), with a total score range of 0 to 56, where <17 indicates mild severity, 18 to 24 mild to moderate severity, and 25 to 30 moderate to severe severity.

The HAM-A assessments are to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28. Every effort should be made for the same rater to perform all HAM-A assessments for an individual subject.

The HAM-A total score will be calculated as the sum of the 14 individual item scores. A copy of the HAM-A is provided in Appendix 3.

# 11.4. Clinical Global Impression (CGI)

The CGI is a validated measure often utilized in clinical trials to allow clinicians to integrate several sources of information into a single rating of the subject's condition. The CGI scale consists of 3 items. Only the first 2 items are being used in this study.

The Clinical Global Impression - Severity (CGI-S) uses a 7-point Likert scale to rate the severity of the subject's illness at the time of assessment, relative to the clinician's past experience with subjects who have the same diagnosis. Considering total clinical experience, a subject is assessed on severity of mental illness at the time of rating as 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=extremely ill (Busner 2007a). The CGI-S assessments are to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28.

The CGI-I employs a 7-point Likert scale to measure the overall improvement in the subject's condition posttreatment. The Investigator will rate the subject's total improvement whether or

not it is due entirely to drug treatment. Response choices include: 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse (Busner 2007b). The CGI-I is only rated at posttreatment assessments. By definition, all CGI-I assessments are evaluated against baseline conditions. CGI-I response will be defined as having a CGI-I score of "very much improved" or "much improved." The CGI-I assessments are to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28. A copy of the CGI is provided in Appendix 4.

## 11.5. Short Form-36 (SF-36)

The SF-36® Health Survey is a subject-reported 36-item instrument for measuring functional health and well-being in eight dimensions (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health) (Ware 2007). Scores are provided for each of the eight dimensions and are totaled into a Physical Component Summary and a Mental Component Summary. Higher SF-36 scores indicate a better state of health. The SF-36 requires approximately 10 minutes to complete, and can be self-administered or completed by interview in person or by telephone. In Part B, the SF-36 assessments are to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28.

A copy of the SF-36 is provided in Appendix 5.

# 11.6. The Fatigue Associated With Depression (FAs-D) Patient-Reported Outcome (PRO)

Fatigue is one of the most common symptoms of MDD. The Fatigue Associated with Depression Questionnaire (FAs-D) was developed to assess fatigue and its impact in patients with MDD. The 13-item patient-reported questionnaire was designed to assess fatigue associated with depression in the past week. Three scores are computed: a six-item fatigue experience subscale (fatigued, tired, exhausted, lack of energy, physically weak, and feeling like everything requires too much effort), a seven-item fatigue impact subscale (impact on household chores; family relationships; enjoyable activities; social activities with friends; self-care; intimate relationships; and productivity at work or school), and a total score (all 13 items) (Matza 2015). Items 12 (impact on intimate relationships) and 13 (impact on productivity at work or school) are not applicable to all subjects, so these items are not answered in some cases. The fatigue experience items are rated on a five-point scale with response options of "never," "rarely," "sometimes," "often," and "always." The impact items are rated on a five-point scale with response options of "not at all," "a little," "somewhat," "quite a bit," and "very much." The two subscales and the total score are computed as the mean of all answered items within each scale, and each scale score has a possible range of 1 to 5, with higher scores representing greater fatigue. In Part B, the FAs-D assessments are to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and

A copy of the FAs-D is provided in Appendix 6.

#### 12. PHARMACOKINETICS

## **12.1.** Blood Sample Collection

Plasma samples for PK analysis in Part A and Part B will be collected predose on Days 2, 3, 4, 5, and 6, predose and 0.25, 0.5, 1, 2, 10, and 12 hours postdose on Day 7 (within ±5 minutes of the scheduled time point through 0.5 hours after dosing and ±15 minutes of the scheduled time point from 1 hour after dosing and greater), prior to discharge on Day 8 for subjects being discharged or 16 hours postdose for subjects remaining as inpatients, predose on Day 14, and in the morning on Day 15. The time of study drug administration is time zero and all post-dosing sampling times are relative to this time. The Investigator or designee will arrange to have the plasma samples processed, stored, and transported as directed for bioanalysis.

In the event of a dose adjustment, an unscheduled PK sample should be collected just prior to the dose change. An additional PK sample may be collected at any time if clinically indicated and at the discretion of the Investigator (eg, for unusual or severe adverse events).

Each sample will be marked with unique identifiers such as the study number, subject number, and the nominal sample time. The date and actual time that the blood sample was taken will be recorded on the CRF or electronically with a bar code or other method.

## 12.2. Storage and Shipment of Pharmacokinetic Samples

The plasma samples should be kept frozen at approximately -70 to -80°C until analyzed. They should be packed as directed to avoid breakage during transit and with sufficient dry ice to prevent thawing for at least 72 hours. A specimen-identification form must be completed and sent to the laboratory with each set of samples. The clinical site will arrange to have the plasma samples transported as directed for bioanalysis as detailed in the PK instructions.

# 12.3. Sample Analysis

Bioanalysis of plasma samples for the determination of SAGE-217 will be performed utilizing a validated liquid chromatography-tandem mass spectrometry method at a qualified laboratory.

#### 13. ASSESSMENT OF SAFETY

## 13.1. Safety Parameters

Safety and tolerability of study drug will be evaluated in Parts A and B by vital signs measurements, clinical laboratory measures, physical examination, ECGs, concomitant medication usage, C-SSRS, SSS, and adverse event reporting.

#### 13.1.1. Demographic/Medical History

Age, race, and ethnic origin will be recorded at the Screening visit. The diagnosis of MDD will be determined using the SCID-I.

#### 13.1.2. Vital Signs

Vital signs include respiratory rate, oral temperature, and supine (for at least 5 minutes prior to the measurement) and standing systolic and diastolic blood pressure and heart rate. Vital signs will be obtained within  $\pm 5$  minutes of the scheduled time point through 0.5 hours after dosing and  $\pm 30$  minutes of the scheduled time point from 1 hour after dosing and greater, unless the subject is asleep between the hours of 23:00 h and 06:00 h.

From Day 1 through Day 7, vital signs and pulse oximetry will be performed at screening (vital signs only) and at the following time points: predose, 0.25, 0.5, 1, 2, and 12 hours after dosing. During the outpatient treatment period, vital signs will be completed prior to dosing and 1 hour after dosing. Vital signs may be repeated at the discretion of the Investigator or Visiting Home Healthcare Provider as clinically indicated.

#### 13.1.3. Weight and Height

Body weight and height will be measured at the Screening visit; weight will also be measured on in the morning on Day 15, and during the follow-up visits on Days 21 and 28.

#### 13.1.4. Physical Examination

A physical examination of all major body systems will be undertaken and recorded at the Screening visit, Day 8, Day 15, and Day 21, with a brief physical examination on Day 28.

#### 13.1.5. Electrocardiogram (ECG)

A 12-lead ECG will be assessed at the Screening visit and 1 hour  $\pm 15$  minutes after dosing on Days 1, 2, 7, and 14 and during the follow-up visit on Day 21. All time points are relative to the time of dosing. The standard intervals as well as any abnormalities will be recorded.

#### 13.1.6. Laboratory Assessments

Blood and urine samples will be collected for hematology, serum chemistry, coagulation, select hormone parameters, and urinalysis at the Screening visit, and in the morning on Days 8 and 15 and during the follow-up visits on Days 21 and 28. Where consent is given, an optional blood sample for hormone and exploratory biochemistry testing will be collected at the Screening visit,

Day 8 and Day 15 and an optional genetic sample for biomarker testing will be collected at the Screening visit.

Serum and urine samples for pregnancy tests will also be collected. These assessments should be performed as outlined below.

All required samples in Part A will be analyzed at local laboratories. All samples in Part B will be analyzed at the central laboratory. Subjects may be considered eligible for the study based on local laboratory results; however, screening samples in Part B must also be sent to the central laboratory.

All clinical laboratory test results outside the reference range will be interpreted by the Investigator as abnormal, not clinically significant (NCS) or abnormal, clinically significant (CS). Screening results considered abnormal, CS recorded at the Screening visit may make the subject ineligible for the study pending review by the Medical Monitor. Clinical laboratory results that are abnormal, CS during the study but within normal range at baseline and/or indicate a worsening from baseline will be considered adverse events, assessed according to Section 13.2.1, and recorded in the eCRF.

#### **13.1.6.1.** Hematology

Hematology tests will include complete blood count, including red blood cells, white blood cells with differentiation, hemoglobin, hematocrit, reticulocytes, and platelets. The coagulation panel will include activated partial thromboplastin time, prothrombin time, and international normalized ratio.

#### 13.1.6.2. Blood Chemistry

Serum chemistry tests will include serum electrolytes; renal function tests, including creatinine, blood urea nitrogen, bicarbonate or total carbon dioxide; liver function tests, including alkaline phosphatase, total bilirubin, aspartate aminotransferase, and alanine aminotransferase; total protein; albumin; and thyroid stimulating hormone.

#### **13.1.6.3.** Urinalysis

Urinalysis will include assessment of protein, blood, glucose, ketones, bile, urobilinogen, hemoglobin, leukocyte esterase, nitrites, color, turbidity, pH, and specific gravity.

#### 13.1.6.4. Hormones and Exploratory Biochemistry

Optional blood samples will be collected and may be analyzed for stress hormone levels, kynurenine biochemistry, and markers of inflammation. Future research may suggest other biochemical pathways as candidates for influencing not only response to SAGE-217 but also susceptibility to disorders for which SAGE-217 may be evaluated. Thus, the exploratory biochemistry may involve study of additional unnamed molecular pathways, but only as related to disease susceptibility and drug action.

## 13.1.6.5. Virus Serology

Subjects will be screened for hepatitis (HBsAg and anti-HCV) and HIV prior to being enrolled in the study.

#### 13.1.6.6. Pregnancy Test

Females of childbearing potential will be tested for pregnancy by serum pregnancy test at the Screening visit and by urine pregnancy test on Day 1 (predose) and at the follow-up visit on Day 28. In addition, female subjects who prematurely discontinue before Day 28 will have a pregnancy test performed at the early termination visit.

#### 13.1.6.7. Genetic Testing

Where consent is given, an optional genetic sample for biomarker testing will be collected at the Screening visit.

The objective of this research is to collect and store blood samples for possible DNA extraction and exploratory research into how genes or specific genetic variation may influence response (ie, distribution, safety, tolerability, and efficacy) to SAGE-217. Specific genetic variations of interest include but are not limited to: classes of metabolizing enzymes (eg, cytochrome P450 supra-family genes), genes encoding enzymes involved in the production and metabolism of SAGE-217 (eg, AKR1C4 [3α-hydroxysteroid dehydrogenase]), genes associated with the γ-aminobutyric acid (GABA) receptor (eg, GABRA1-A6, GABRB1-B3, GABRD, GABRE, GABRG1-3), and genes associated with the production and degradation of GABA.

Future research may suggest other genes or gene categories as candidates for influencing not only response to SAGE-217 but also susceptibility to disorders for which SAGE-217 may be evaluated. Thus, the genetic research may involve study of additional unnamed genes or gene categories, but only as related to disease susceptibility and drug action.

#### 13.1.6.8. Drugs of Abuse and Alcohol

A urine sample for assessment of selected drugs of abuse (including amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates, phencyclidine, and propoxyphene) and a serum or breath sample for alcohol screen will be collected at screening and predose on Day 1. Use of benzodiazepines at screening is not necessarily exclusionary, as subjects will be allowed to take psychotropics that have been initiated at least 14 days prior to admission to the study center at a stable dose following discussion with the Sponsor (see Section 9.3).

### 13.1.7. Columbia-Suicide Severity Rating Scale (C-SSRS)

Suicidality will be monitored during the study using the C-SSRS. This scale consists of a baseline evaluation that assesses the lifetime experience of the subject with suicidal ideation and behavior (Posner 2008a), and a post-baseline evaluation that focuses on suicidality since the last study visit (Posner 2008b). The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe).

If, in the opinion of the Investigator, the subject is showing clinically meaningful changes in suicidality, no further study drug will be administered and the subject will be referred to a psychologist or psychiatrist for further evaluation. This information will be tracked.

The "Baseline/Screening" C-SSRS form will be completed at screening (lifetime history and past 24 months). The "Since Last Visit" C-SSRS form will be completed at any time of day at all

subsequent time points, as outlined in Table 2 and Table 3. The C-SSRS is provided in Appendix 7.

## 13.1.8. Stanford Sleepiness Scale (SSS)

The SSS is subject-rated scale designed to quickly assess how alert a subject is feeling. Degrees of sleepiness and alertness are rated on a scale of 1 to 7, where the lowest score of '1' indicates the subject is 'feeling active, vital, alert, or wide awake' and the highest score of '7' indicates the subject is 'no longer fighting sleep, sleep onset soon; having dream-like thoughts' (Hoddes 1973).

In both Part A and Part B, from Day 1 through Day 7, SSS will be completed at the following time points: predose, 0.25, 0.5, 1, and 2 after dosing. The scale is to be completed within  $\pm 5$  minutes of the scheduled time point through 0.5 hours after dosing and  $\pm 15$  minutes of the scheduled time point from 1 hour after dosing and greater, unless the subject is asleep between 23:00 h and 06:00 h during the inpatient treatment period. During the outpatient treatment period, SSS will be completed prior to dosing and 1 hour after dosing. All time points are relative to the time of dosing. The SSS is provided in Appendix 8.

#### 13.2. Adverse and Serious Adverse Events

#### 13.2.1. Definition of Adverse Events

#### **13.2.1.1.** Adverse Event

An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. In clinical studies, an adverse event can include an undesirable medical condition occurring at any time, including baseline or washout periods, even if no study treatment has been administered.

#### 13.2.1.2. Suspected Adverse Reaction

A suspected adverse reaction is any adverse event for which there is a reasonable possibility that the drug caused the adverse event. For the purposes of Investigational New Drug safety reporting, "reasonable possibility" means there is evidence to suggest a causal relationship between the drug and the adverse event. Suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any adverse event caused by a drug.

#### 13.2.1.3. Serious Adverse Event

A serious adverse event is an adverse event occurring during any study phase and at any dose of the investigational product, comparator or placebo, that fulfils one or more of the following:

- It results in death
- It is immediately life-threatening
- It requires inpatient hospitalization or prolongation of existing hospitalization
- It results in persistent or significant disability or incapacity

- It results in a congenital abnormality or birth defect
- It is an important medical event that may jeopardize the subject or may require medical intervention to prevent one of the outcomes listed above.

All serious adverse events that occur after any subject has been enrolled, whether or not they are related to the study, must be recorded for the duration of the study on forms provided by Sage Therapeutics or designee.

# 13.3. Relationship to Study Drug

An Investigator who is qualified in medicine must make the determination of relationship to the investigational product for each adverse event (unrelated, possibly related or probably related). The Investigator should decide whether, in his or her medical judgment, there is a reasonable possibility that the event may have been caused by the investigational product. If no valid reason exists for suggesting a relationship, then the adverse event should be classified as "unrelated." If there is any valid reason, even if undetermined, for suspecting a possible cause-and-effect relationship between the investigational product and the occurrence of the adverse event, then the adverse event should be considered "related."

| Not Related: | No relationship between the experience and the administration of study drug; related to other |
|---|---|
| | etiologies such as concomitant medications or subject's clinical state. |
| Possibly | A reaction that follows a plausible temporal sequence from administration of the study drug and |
| Related: | follows a known response pattern to the suspected study drug. |
| | The reaction might have been produced by the subject's clinical state or other modes of therapy |
| | administered to the subject, but this is not known for sure. |
| Probably | A reaction that follows a plausible temporal sequence from administration of the study drug and |
| Related: | follows a known response pattern to the suspected study drug. |
| | The reaction cannot be reasonably explained by the known characteristics of the subject's clinical |
| | state or other modes of therapy administered to the subject. |

If the relationship between the adverse event/serious adverse event and the investigational product is determined to be "possible" or "probable", the event will be considered to be related to the investigational product for the purposes of expedited regulatory reporting.

# **13.4.** Recording Adverse Events

Adverse events spontaneously reported by the subject and/or in response to an open question from the study personnel or revealed by observation will be recorded during the study at the investigational site. Clinically significant changes in laboratory values, blood pressure, and pulse need not be reported as adverse events unless they prompt corrective medical action by the Investigator, constitute a serious adverse event, or lead to discontinuation of administration of study drug.

Information about adverse events will be collected from the signing of the ICF until the final visit of the study for that subject. Adverse events that occur after the first administration of study drug will be denoted TEAEs.

All adverse events will be followed until they are resolved or have reached a clinical plateau with no expectation of future change.

The adverse event term should be reported in standard medical terminology when possible. For each adverse event, the Investigator will evaluate and report the onset (date and time), resolution or clinical plateau (date and time), severity, causality, action taken, outcome, and whether or not it caused the subject to discontinue the study.

Severity will be assessed according to the following scale:

- Mild (awareness of sign or symptom, but easily tolerated)
- Moderate (discomfort sufficient to cause interference with normal activities)
- Severe (incapacitating, with inability to perform normal activities)

## 13.5. Reporting Adverse Events

All serious adverse events (regardless of causality) will be recorded from the signing of the ICF until the Day 28 follow-up visit. Any serious adverse events considered possibly or probably related to the investigational product and discovered by the Investigator at any time after the study should be reported. All serious adverse events must be reported to the Sponsor or Sponsor's designee immediately by phone and in writing within 24 hours of the first awareness of the event. The Investigator must complete, sign and date the serious adverse event pages, verify the accuracy of the information recorded on the serious adverse event pages with the corresponding source documents, and send a copy to Sage Therapeutics or designee.

Additional follow-up information, if required or available, should be sent to Sage Therapeutics or designee within 24 hours of receipt; a follow-up serious adverse event form should be completed and placed with the original serious adverse event information and kept with the appropriate section of the study file.

Sage Therapeutics or designee is responsible for notifying the relevant regulatory authorities of certain events. It is the Principal Investigator's responsibility to notify the IRB of all serious adverse events that occur at his or her site if applicable per the IRB's requirements. Investigators will also be notified of all unexpected, serious, drug-related events (7-/15-Day Safety Reports) that occur during the clinical study. Each site is responsible for notifying its IRB of these additional serious adverse events.

# 13.6. Emergency Identification of Study Drug

Part B of the study is double-blind. The pharmacist responsible for preparing the solutions will be unblinded and will retain an official paper copy of the randomization schedule. In addition, an unblinded Monitor will perform drug accountability during the study.

During the study, the blind is to be broken only when the safety of a subject is at risk and the treatment plan is dependent on the study treatment received. Unless a subject is at immediate risk, the Investigator must make diligent attempts to contact the Sponsor prior to unblinding the study treatment administered to a subject. Any request from the Investigator about the treatment administered to study subjects must be discussed with the Sponsor. If the unblinding occurs without the Sponsor's knowledge, the Investigator must notify the Sponsor as soon as possible and no later than the next business morning. All circumstances surrounding a premature unblinding must be clearly documented in the source records. Unless a subject is at immediate

risk, any request for the unblinding of individual subjects must be made in writing to the Sponsor and approved by the appropriate Sponsor personnel, according to standard operating procedures. The blinding of the study will be broken after the database has been locked. Electronic copies of the randomization code will be made available to the laboratory performing the bioanalytical analyses in order to allow for limited analysis of samples from subjects receiving matching placebo.

In all cases where the study drug allocation for a subject is unblinded, pertinent information must be documented in the subject's records and on the eCRF. If the subject or study center personnel (other than pharmacist) have been unblinded, the subject will be terminated from the study.

#### 14. STATISTICS

## 14.1. Data Analysis Sets

#### 14.1.1. Analysis Populations and Methods

The Safety Population (for both Part A and Part B), defined as all subjects administered study drug, will be used to provide descriptive summaries of safety data.

The Efficacy Population (for both Part A and Part B), defined as all subjects in the Safety Population who complete at least 1 day of dosing of study drug and have at least one post-baseline efficacy evaluation, will be used to analyze efficacy data.

The PK Population will consist of all subjects in the Safety Population with sufficient plasma concentrations for PK evaluations, and will be used to summarize PK data.

## 14.2. Handling of Missing Data

Every attempt will be made to avoid missing data. All subjects will be used in the analyses, as per the analysis populations, using all non-missing data available. No imputation process will be used to estimate missing data. A sensitivity analysis will be used to investigate the impact of missing data if  $\geq$ 5% of subjects have missing data.

### 14.3. General Considerations

For the purpose of all safety and efficacy analyses where applicable, baseline is defined as the last measurement prior to the start of study drug administration.

Continuous endpoints will be summarized with n, mean, standard deviation (SD), median, minimum and maximum. In addition, change from baseline values will be calculated at each time point and summarized descriptively. For categorical endpoints, descriptive summaries will include counts and percentages.

# 14.4. Demographics and Baseline Characteristics

Demographic data, such as age, race, and ethnicity, and baseline characteristics, such as height, weight, and body mass index (BMI), will be summarized using the Safety Population.

Hepatitis, HIV, drug and alcohol, and pregnancy screening results will be listed, but not summarized as they are considered part of the inclusion/exclusion criteria.

Medical/family history will be listed by subject.

# 14.5. Efficacy Analyses

Efficacy data will be summarized using appropriate descriptive statistics and other data presentation methods where applicable; subject listings will be provided for all efficacy data. For (the open-label) Part A, efficacy data will be summarized descriptively. For Part B, subjects will be analyzed according to randomized treatment.

An analysis of ten subjects completing Part A is planned to inform Part B study conduct.

For Part B of the study, change from baseline to each assessment in HAM-D total score will be analyzed using a mixed effects model for repeated measures (MMRM); the model will include center, treatment, baseline HAM-D total score, antidepressant use strata, assessment time point, and time point-by-treatment as explanatory variables. Center will be treated as a random effect while all other explanatory variables will be treated as fixed effects. All post-baseline time points will be included in the model. The main comparison will be between SAGE-217 Oral Solution and matching placebo at the 15-day time point. Model-based point estimates (ie, least squares [LS] means), 95% confidence intervals, and p-values) will be reported where applicable. An unstructured covariance structure will be used to model the within-subject errors. Compound symmetry covariance structure will be used if there is a convergence issue with the unstructured covariance model.

Descriptive statistics for HAM-D total score and change from baseline values will be presented by assessment time point for Part A. Summaries will include n, mean, SD, median, minimum, and maximum.

Similar to those methods described above for Part B, an MMRM will be used for the analysis of the following variables: changes from baseline in MADRS total score and HAM-A total score, and select individual item and subscale scores. For each model, the comparison of interest will be between SAGE-217 Oral Solution and matching placebo at the 15-day time point. Model-based point estimates (ie, LS means), 95% confidence intervals, and p-values will be reported.

Logistic regression methods will be used for the analysis of the following binary variables: HAM-D response (defined as ≥50% reduction from baseline in HAM-D total score), HAM-D remission (defined as HAM-D total score of ≤7.0), and CGI-I response. Logistic regression models will include terms for center, treatment, antidepressant use strata, and baseline score. The comparison of interest will be the difference between SAGE-217 Oral Solution and matching placebo at the 15-day time point in Part B. Model-based point estimates (ie, odds ratios), 95% confidence intervals, and p-values will be reported. For the CGI-I response analysis, baseline CGI-S score will be included in the model.

For all scores, descriptive statistics, change from baseline values, and response variables will be presented by treatment and assessment time point. Summaries will include n, mean, SD, median, minimum, and maximum.

Similar to the main comparison of HAM-D total score in Part B, descriptive summary statistics will be provided and an MMRM model will be used to analyze the change from baseline in SF-36 and FAs-D.

# 14.6. Safety Analyses

Safety and tolerability of study drug will be evaluated by adverse events, concomitant medication usage, changes from baseline in physical examination, vital signs, clinical laboratory evaluations, and 12-lead ECG. Suicidality will be monitored by the C-SSRS. Sedation will be assessed using the SSS. Safety data will be listed by subject and summarized by treatment group. All safety summaries will be performed on the Safety Population.

#### 14.6.1. Adverse Events

The analysis of adverse events will be based on the concept of TEAEs. A TEAE is defined as an adverse event with onset after the start of study drug, or any worsening of a pre-existing medical condition/adverse event with onset after the start of study drug and until 7 days after the last dose. The incidence of TEAEs will be summarized overall and by Medical Dictionary for Regulatory Activities (MedDRA) Version 18.1 or higher System Organ Class (SOC) and preferred term. Incidences will be presented in order of decreasing frequency for the SAGE-217 Oral Solution treatment group. In addition, summaries will be provided by severity (mild, moderate, severe) and by causality (related, not related) to study drug (see Section 13.3).

Treatment-emergent adverse events leading to discontinuation and serious adverse events (see Section 13.2.1.3 for definition) with onset after the start of randomized study drug will also be summarized.

All adverse events and serious adverse events (including those with onset or worsening before the start of study drug) through the Day 28 follow-up visit will be listed.

## 14.6.2. Clinical Laboratory Evaluations

Clinical laboratory results will be listed by subject and timing of collection. Mean changes from baseline in clinical laboratory measures will be summarized.

#### 14.6.3. Physical Examinations

Physical examinations in Parts A and B will be summarized at the Screening visit, Day 8, Day 15, Day 21, and Day 28 visits. Any clinically significant change in physical examination compared to those observed at screening should be noted as an adverse event.

#### 14.6.4. Vital Signs

Vital sign results will be listed by subject and timing of collection. Mean changes from randomization in vital signs will be summarized by time point.

#### 14.6.5. 12-Lead Electrocardiogram

The following ECG parameters will be listed for each subject: heart rate, PR, QRS, QT, QTc, and QT interval calculated using the Fridericia method (QTcF). Any clinically significant abnormalities or changes in ECGs should be listed as an adverse event. Electrocardiogram findings will be listed by subject and visit.

#### 14.6.6. Prior and Concomitant Medications

Medications will be recorded at each study visit during the study and will be coded using World Health Organization-Drug dictionary (WHO-DD) September 2015, or later.

Medications will be presented according to whether they are being taken prior to and/or during the study (concomitant). Prior medications are defined as those taken during the 30 days prior to informed consent. Concomitant medications are defined as those with a start date on or after the first dose of study drug, or those with a start date before the first dose of study drug that are ongoing or with a stop date on or after the first dose of study drug. If medication dates are

incomplete and it is not clear whether the medication was concomitant, it will be assumed to be concomitant.

Details of prior and concomitant medications will be listed by subject, start date, and verbatim term.

#### 14.6.7. Columbia Suicide Severity Rating Scale

Suicidality data collected on the C-SSRS at baseline and by visit during the Treatment Period will be listed for all subjects. Listings will include behavior type and/or category for Suicidal Ideation and Suicidal Behavior of the C-SSRS.

#### 14.6.8. Stanford Sleepiness Scale

Sedation data collected on the SSS will be listed for all subjects. Changes in score over time will be represented graphically, and change from Day 1 will be measured.

## 14.7. Pharmacokinetic Analyses

Pharmacokinetic parameters will be summarized using appropriate descriptive statistics. Time at maximum (peak) plasma concentration ( $t_{max}$ ) will be summarized using n, mean, SD, median, minimum, and maximum. All other PK parameters will be summarized using n, geometric mean, coefficient of variation, median, minimum, and maximum and listed by subject.

Plasma concentrations and PK parameters will be listed by subject.

In addition to typical descriptive statistics, summaries should include geometric mean, coefficient of variation, and geometric coefficient of variation.

# **14.8.** Determination of Sample Size

The sample size of ten subjects for Part A was selected based on clinical and not statistical considerations.

For Part B, assuming a two-sided t-test at an alpha level of 0.10, a sample size of 23 subjects per group would provide 80% power to detect an effect size of 0.75 between the SAGE-217 Oral Solution and matching placebo groups with regard to the secondary efficacy outcome variable of change from baseline in HAM-D total score. An effect size of 0.75 corresponds to a matching placebo-adjusted difference of 7.5 points in the change from baseline in HAM-D total score at 15 days with an assumed SD of 10 points. By including two treatment groups and using a 1:1 randomization, a total of 46 subjects are required. Assuming a non-evaluability rate of 10%, up to 52 subjects will be randomized.

# 14.9. Changes From Protocol Specified Analyses

Any changes from the analytical methods outlined in the protocol will be documented in the final statistical analysis plan.

#### 15. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

# 15.1. Study Monitoring

Before an investigational site can enter a subject into the study, a representative of Sage Therapeutics or designee will visit the investigational study site to:

- Determine the adequacy of the facilities; and
- Discuss with the Investigator(s) and other personnel their responsibilities with regard to protocol adherence, and the responsibilities of Sage Therapeutics or designee or its representatives. This will be documented in a Clinical Study Agreement between Sage Therapeutics and the Investigator.

During the study, a monitor from Sage Therapeutics or designee will have regular contacts with the investigational site for the following:

- Provide information and support to the Investigator(s);
- Confirm that facilities remain acceptable;
- Confirm that the investigational team is adhering to the protocol, that data are being accurately recorded in the eCRFs, and that investigational product accountability checks are being performed;
- Perform source data verification. This includes a comparison of the data in the eCRFs with the subject's medical records at the hospital or practice, and other records relevant to the study. This will require direct access to all original records for each subject (eg, clinic charts);
- Record and report any protocol deviations not previously sent to Sage Therapeutics or designee; and
- Confirm adverse events and serious adverse events have been properly documented on eCRFs and confirm any serious adverse events have been forwarded to Sage Therapeutics or designee and those serious adverse events that met criteria for reporting have been forwarded to the IRB.

The monitor will be available between visits if the Investigator(s) or other staff needs information or advice.

# 15.2. Audits and Inspections

Authorized representatives of Sage Therapeutics, a regulatory authority, an Independent Ethics Committee (IEC) or an IRB may visit the site to perform audits or inspections, including source data verification. The purpose of a Sage Therapeutics or designee audit or inspection is to systematically and independently examine all study-related activities and documents to determine whether these activities were conducted, and data were recorded, analyzed, and accurately reported according to the protocol, GCP guidelines of the International Council for

Harmonisation (ICH), and any applicable regulatory requirements. The Investigator should contact Sage Therapeutics immediately if contacted by a regulatory agency about an inspection.

## 15.3. Institutional Review Board (IRB)

The Principal Investigator must obtain IRB approval for the investigation. Initial IRB approval and all materials approved by the IRB for this study, including the subject consent form and recruitment materials, must be maintained by the Investigator and made available for inspection.

### 16. QUALITY CONTROL AND QUALITY ASSURANCE

The Investigator and institution will permit study-related monitoring, audits, IRB review, and regulatory inspections as requested by the Food and Drug Administration, the Sponsor, or the Sponsor's designee, including direct access to source data/documents (ie, original medical records, laboratory reports, hospital documents, progress reports, signed ICFs) in addition to eCRFs.

Quality assurance and quality-control systems with written standard operating procedures will be followed to ensure this study will be conducted and data will be generated, documented (recorded), and reported in compliance with the protocol, GCP, and the applicable regulatory requirements.

The site's dedicated study monitor will arrange to visit the Investigator at regular intervals during the study. The monitoring visits must be conducted according to the applicable ICH and GCP guidelines to ensure protocol adherence, quality of data, drug accountability, compliance with regulatory requirements, and continued adequacy of the investigational site and its facilities.

During these visits, eCRFs and other data related to the study will be reviewed and any discrepancies or omissions will be identified and resolved. The study monitor will be given access to study-relevant source documents (including medical records) for purposes of source data verification.

During and/or after completion of the study, quality-assurance officers named by Sage Therapeutics or the regulatory authorities may wish to perform on-site audits. The Investigator is expected to cooperate with any audit and provide assistance and documentation (including source data) as requested.

Quality control will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly.

Agreements made by the Sponsor with the Investigator/institution and any other parties involved with the clinical study will be in writing in a separate agreement.

#### 17. ETHICS

#### 17.1. Ethics Review

The final study protocol, including the final version of the ICF, must be approved or given a favorable opinion in writing by an IRB or IEC as appropriate. The Investigator must submit written approval to Sage Therapeutics or designee before he or she can enroll any subject into the study.

The Principal Investigator is responsible for informing the IRB or IEC of any amendment to the protocol in accordance with local requirements. In addition, the IRB or IEC must approve all advertising used to recruit subjects for the study. The protocol must be re-approved by the IRB or IEC upon receipt of amendments and annually, as local regulations require.

The Principal Investigator is also responsible for providing the IRB with reports of any reportable serious adverse drug reactions from any other study conducted with the investigational product. Sage Therapeutics or designee will provide this information to the Principal Investigator.

Progress reports and notifications of serious adverse drug reactions will be provided to the IRB or IEC according to local regulations and guidelines.

## 17.2. Ethical Conduct of the Study

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and its most recent amendment (2008) and are consistent with ICH/GCP and other applicable regulatory requirements.

#### 17.3. Written Informed Consent

The Principal Investigator will ensure that the subject is given full and adequate oral and written information about the nature, purpose, possible risk, and benefit of the study. Subjects must also be notified that they are free to discontinue from the study at any time. The subject should be given the opportunity to ask questions and allowed time to consider the information provided before signing the ICF.

As additional assessments, the ICF will contain provisions for optional consent for the collection of blood samples for biochemistry during screening, Day 8, and Day 15 and biomarker testing during screening. The ICF, as specified by the clinical site's IRB, must follow the Protection of Human Subjects regulations listed in the Code of Federal Regulations, Title 21, Part 50.

The subject's signed and dated informed consent must be obtained before conducting any study procedures.

The Principal Investigator(s) must maintain the original, signed ICF. A copy of the signed ICF must be given to the subject.

#### 18. DATA HANDLING AND RECORDKEEPING

Procedures for data handling (including electronic data) used in this protocol will be documented in a Data Management Plan.

Electronic CRFs will be completed for each study subject. It is the Investigator's responsibility to ensure the accuracy, completeness, and timeliness of the data reported in the subject's eCRF. Source documentation supporting the eCRF data should indicate the subject's participation in the study and should document the dates and details of study procedures, adverse events, and subject status.

The Investigator will have access to the electronic data capture system and will receive a copy of the subject eCRF data at the end of the study. For subjects who discontinue or terminate from the study, the eCRFs will be completed as much as possible, and the reason for the discontinuation or termination clearly and concisely specified on the appropriate eCRF.

# 18.1. Inspection of Records

Sage Therapeutics or designee will be allowed to conduct site visits to the investigational facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the monitor to inspect the drug storage area, study drug stocks, drug accountability records, subject charts and study source documents, and other records related to study conduct.

#### 18.2. Retention of Records

The Principal Investigator must maintain all documentation relating to the study for a period of 2 years after the last marketing application approval or, if not approved, 2 years following the discontinuation of the test article for investigation. If it becomes necessary for Sage Therapeutics or the Regulatory Authority to review any documentation relating to the study, the Investigator must permit access to such records.

# 18.3. Confidentiality

To maintain subject privacy, all eCRFs, study reports, and communications will identify the subject by the assigned subject number. The Investigator will grant monitor(s) and auditor(s) from the Sponsor or its designee and regulatory authority(ies) access to the subject's original medical records for verification of data gathered on the eCRFs and to audit the data collection process. The subject's confidentiality will be maintained and will not be made publicly available to the extent permitted by the applicable laws and regulations.

Subjects will be notified that registration information, results, and other information about this study will be submitted to ClinicalTrials.gov, a publicly available trial registry database; however, protected health information of individual subjects will not be used.

All information regarding the investigational product supplied by Sage Therapeutics to the Investigator is privileged and confidential information. The Investigator agrees to use this information to accomplish the study and will not use it for other purposes without consent from the Sponsor. It is understood that there is an obligation to provide the Sponsor with complete data obtained during the study. The information obtained from the clinical study will be used towards the development of the investigational product and may be disclosed to regulatory authorities, other Investigators, corporate partners, or consultants, as required.

# 19. PUBLICATION POLICY

All information concerning SAGE-217 is considered confidential and shall remain the sole property of Sage Therapeutics. The Investigator agrees to use this information only in conducting the study and shall not use it for any other purposes without written approval from Sage Therapeutics. No publication or disclosure of study results will be permitted except as specified in a separate, written, agreement between Sage Therapeutics and the Investigator.

#### 20. LIST OF REFERENCES

Angst J, Angst F, Stassen HH. Suicide risk in patients with major depressive disorder. J Clin Psychiatry. 1999;60 Suppl 2:57-62; discussion 75-6, 113-6.

Busner J, Targum S. CGI-S. (2007a), as adapted from Kay, Stanley R, Positive and Negative Symptoms in Schizophrenia: Assessment and Research. Clinical and Experimental Psychiatry, Monograph No. 5. Brunner/Mazel, 1991. Modified from Guy W. Clinical Global Impressions: In ECDEU Assessment Manual for Psychopharmacology. 1976; 218-22. Revised DHEW Pub. (ADM) Rockville, MD: National Institute for Mental Health.

Busner J, Targum S. CGI-I. (2007b), as adapted from Spearing, et al. Psychiatry Research, 1997;73:159-71. Modified from Guy W. Clinical Global Impressions: In ECDEU Assessment Manual for Psychopharmacology. 1976; 218-22. Revised DHEW Pub. (ADM) Rockville, MD: National Institute for Mental Health.

Conradi HJ, Ormel J, de Jonge P. Presence of individual (residual) symptoms during depressive episodes and periods of remission: a 3-year prospective study. Psychol Med. 2011 Jun;41(6):1165-74.

Drugan RC, Morrow AL, Weizman R, et al. Stress-induced behavioral depression in the rat is associated with a decrease in GABA receptor-mediated chloride ion flux and brain benzodiazepine receptor occupancy. Brain Res. 1989;487: 45–51.

DSM-5. Diagnostic and statistical manual of mental disorders (5th ed.). American Psychiatric Association 2013. Arlington, VA: American Psychiatric Publishing.

Fournier JC, DeRubeis RJ, Hollon SD, et al. Antidepressant drug effects and depression severity—a patient-level meta-analysis. JAMA. 2010;303:47-53.

Gerner RH, Hare TA. GABA in normal subjects and patients with depression, schizophrenia, mania, and anorexia nervosa. Am J Psychiatry. 1981;138:1098–101.

Greenberg PE, Fournier AA, Sisitsky T, Pike CT, Kessler RC. The economic burden of adults with major depressive disorder in the United States (2005 and 2010). J Clin Psychiatry. 2015 Feb;76(2):155-62.

Hoddes E, Zarcone V, Smythe H, Phillips R, Dement WC. Quantification of sleepiness: a new approach. Psychophysiology. 1973 Jul;10(4):431-6.

Honig A, Bartlett JR, Bouras N, Bridges PK. Amino acid levels in depression: a preliminary investigation. J Psychiatr Res. 1988; 22:159–64.

Kirsch I, Deacon BJ, Huedo-Medina TB, et al. Initial severity and antidepressant benefits: A meta-analysis of data submitted to the Food and Drug Administration. PLoS Med. 2008;5(2):e45.

Luscher B, Shen Q, Sahir N. The GABAergic deficit hypothesis of major depressive disorder. Mol Psychiatry. 2011;16(4):383-406.

Maguire J, Mody I. GABA(A)R plasticity during pregnancy: Relevance to postpartum depression. Neuron. 2008;59(2);207-13.

Maguire J, Ferando I, Simonsen C, Mody I. Excitability changes related to GABAA receptor plasticity during pregnancy. J Neurosci. 2009;29(30):9592-601.

Mann JJ, Oguendo MA, Watson KT, et al. Anxiety in major depression and cerebrospinal fluid free gamma-aminobutyric acid. Depress Anxiety. 2014;31(10):814-21.

Matza LS, Murray LT, Phillips GA, et al. Qualitative Research on Fatigue Associated with Depression: Content Validity of the Fatigue Associated with Depression Questionnaire (FAsD-V2). Patient. 2015 Oct;8(5):433-43.

Posner K, Brent D, Lucas C, et al. C-SSRS BL/Scr: 2008a Research Foundation for Mental Hygiene, Inc.C-SSRS—Baseline/Screening (Version 1/14/09).

Posner K, Brent D, Lucas C, et al. C-SSRS SLV: 2008b Research Foundation for Mental Hygiene, Inc.C-SSRS—Since Last Visit (Version 1/14/09).

Romera I, Pérez V, Ciudad A, et al. Residual symptoms and functioning in depression, does the type of residual symptom matter? A post-hoc analysis. BMC Psychiatry. 2013 Feb 11;13:51.

Schüle C, Nothdurfter C, Rupprecht R. The role of allopregnanolone in depression and anxiety. Prog Neurobiol. 2014 Feb;113:79-87.

Trivedi MH, Rush AJ, Wisniewski SR, et al. (STAR\*D Study Team). Evaluation of outcomes with citalopram for depression using measurement-based care in STAR\*D: implications for clinical practice. Am J Psychiatry. 2006 Jan;163(1):28-40.

Ware JE Jr, Kosinski M, Bjorner JB, et al. User's Manual for the SF-36v2 Health Survey. 2nd ed. Lincoln, RI: QualityMetric Incorporated; 2007.

Williams JBW, Kobak KA. Development and reliability of a structured interview guide for the Montgomery-Asberg Depression Rating Scale (SIGMA). Br J Psychiatry. 2008;192:52-8.

Williams JBW. SIGH-D 24hr: V1.3 – 24 HR Version. 2013a.

Williams JBW. SIGH-D Past week: - Past Week Version. 2013b.

Williams JBW. SIGH-A 24hr: V1.3 – 24 HR Version. 2013c.

Williams JBW. SIGH-A Past week: - Past Week Version. 2013d.

# 21. APPENDICES

# Appendix 1. HAMILTON RATING SCALE FOR DEPRESSION, 17-ITEM (HAM-D)

# STRUCTURED INTERVIEW GUIDE FOR THE HAMILTON DEPRESSION RATING SCALE – 17 ITEM VERSION (SIGH-D-17) – 24 HR TWENTY-FOUR HOUR ASSESSMENT VERSION

Janet B.W. Williams, PhD

#### INTERVIEWER

The first question for each item, in bold type, should be asked exactly as written. Often this question will elicit enough information about the severity and frequency of a symptom for you to rate the item with confidence. Follow-up questions are provided for use when further exploration or additional clarification of symptoms is necessary. The specified questions should be asked until you have enough information to rate the item confidently. In some cases, you may also have to add your own follow-up questions to obtain necessary information. You should ask for examples for any symptoms acknowledged as present (e.g., "Can you give me an example of that?"). For some of the HAM-D items, you may find you have already asked about some of the symptoms (for a previous item). You do not need to repeat questions about these symptoms unless you need additional information to rate their severity.

<u>Time period</u>. In this 24 hour version, the interview questions indicate that the ratings should be based on the subject's condition over the past 24 hours..

Referent of "usual" or "normal" condition. In the HAM-D, most items are rated positive only if they represent a change from usual functioning. In most cases, this version of the SIGH-D will be used at some time after the original Past Week version of the scale, during which a euthymic baseline (the most recent 2-month period of non-depressed functioning) was established. This euthymic baseline should be the referent for determining change. When no clear euthymic baseline can be established, one should rate symptomatic behavior as one sees it, even if it is not a change from the patient's usual dysphoric self.

Administration method. This version includes interview questions to help the clinician rate psychomotor agitation and psychomotor retardation when the interview is administered by telephone. Several research studies have demonstrated that depression scale scores are equivalent whether the scale is administered face-to-face, by telephone, or by video (Williams JBW and Kobak KA: Development and Reliability of a Structured Interview Guide for the Montgomery-Asberg Depression Rating Scale. Br J Psychiatry 192, 52-58, 2008; Kobak KA: A comparison of face-to-face and remote administration of the Hamilton Depression Rating Scale via videoconferencing. J Telemed Telecare 10, 231-235, 2004).

This instrument provides an interview guide for the Hamilton Depression Scale (Hamilton, Max: A rating scale for depression. J Neurol Neurosurg Psychiat 23:56-81, 1960). The anohor point descriptions for all items except Helplessness, Hopelessness, and Worthlessness, in the 25-item version with very minor modifications, have been taken from the ECDEU Assessment Manual (GV, William, ECDEU Assessment Manual for Psychopharmacology, Revised 1976, DHEW Publication No. (ADM) 78-338). The loss of weight item has been simplified to eliminate the section for ratings by ward staff and the "Not assessed" anohor point. A reliability study of the SIGH-D (interview guide for the HAM-D slone) was published in the Archives of General Psychiatry (1983;45:742-747). Additional designators were added in parentheses to the anohor points by Kobak, Lipsitz and Williams to further standardize ratings.

For further information and permission to use or translate the SIGH-D, contact Dr. Williams at jbwwny@gmail.com

| STRUCTURED INTERVIEW GUIDE FOR THE HAMILTON DEPRESSION RATING SCALE – 17 ITEM VERSION (SIGH-D-17) – 24 HR TWENTY-FOUR HOUR ASSESSMENT VERSION | |
|---|---|
| PT'S INITIALS:TIME BEGAN SIGH-D: _ | INTERVIEWER: |
| DATE TODAY:/ | DATE OF LAST EVALUATION: / / |
| OVERVIEW: How have you been feeling since yeste working? IF NOT: Why not? | rday at this time? IF OUTPATIENT: Have you been |
| What's your mood been like since this time yesterday (compared to when you feel okay)? | DEPRESSED MOOD (sadness, hopeless, helpless, worthless): |
| Have you been feeling down or depressed? | 0 Absent |
| IF YES: Can you describe what this feeling has been like for you? How bad is the feeling? | Indicated only on questioning (occasional, mild depression) Spontaneously reported verbally (persistent, mild to moderate depression) |
| Does the feeling lift at all if something good happens? How are you feeling about the future? | Communicated non-verbally, i.e., facial expression, posture, voice, tendency to weep (persistent, moderate to severe depression) |
| IF UNKNOWN: Have you been feeling discouraged or pessimistic since this time yesterday? | VIRTUALLY ONLY those feeling states reported in spontaneous verbal and non-verbal communication (persistent, very severe) |
| IF YES: What have your thoughts been? | depression, with extreme hopelessness or tearfulness) |
| Since this time yesterday, how often have you felt (OWN EQUIVALENT FOR DEPRESSED MOOD)? For how much of the time? | |
| Have you been crying at all? How often? | |
| INTERVIEWER: IF SCORED 1-4 ABOVE, | |
| REVIEW DATE OF EUTHYMIC BASELINE: How long have you been feeling this way (OWN EQUIVALENT FOR DEPRESSED MOOD)? (When was the last time you were feeling well, that is, not depressed at all, for at least 2 | |
| months?) | |

 $\otimes$  2013, v 1.2 – 24 HR Version. Janet B.W. Williams, PhD  

# How have you been spending your time since yesterday at this time (when not at work)?

Have you felt interested in doing (THOSE THINGS), or do you feel you have to push yourself to do them?

How much less interested in these things have you been, since this time yesterday, compared to when you're not depressed? How hard to do you have to push yourself to do them?

Have you stopped doing anything you used to do? (What about hobbies?) IF YES: Why?

About how many hours a day have you spent doing things that interest you, since this time yesterday?

Is there anything you look forward to?

IF WORKING (IN OR OUT OF THE HOME): Since this time yesterday, have you been able to get as much (work) done as you usually do?

How much less productive or efficient are you compared to before you were depressed?

#### 2. WORK AND ACTIVITIES:

| 0 | No difficulty |
|---|---|
| 1 | Thoughts and feelings of incapacity, fatigue or weakness related to activities, work or hobbies (mild reduction in interest or pleasure; no clear impairment in functioning) |
| 2 | Loss of interest in activity, hobbies or work -<br>by direct report of the patient or indirect in<br>listlessness, indecision and vacillation (feels<br>he has to push self to work or activities) (clear<br>reduction in interest, pleasure or functioning) |
| 3 | Decrease in actual time spent in activities or decrease in productivity. In hosp., pt. spends less than 3 hirs./day in activities (hospital job or hobbies) exclusive of ward chores (profound reduction in interest, pleasure, or functioning) |
| 4 | Stopped working because of present illness.<br>In hospital, no activities except ward chores,<br>or fails to perform ward chores unassisted<br>(unable to work or fulfill primary role because |

of illness, and total loss of interest)

Now let's talk about your sleep. What were your usual hours of going to sleep and waking up, before this began?

When have you fallen asleep and awakened since this time yesterday?

Have you had any trouble falling asleep at the beginning of your sleep time, over the past 24 hours? (Right after you went to bed, how long did it take you to fall asleep?)

Did you change the time at which you tried to get to sleep, compared to before you became depressed?

#### 3. INSOMNIA EARLY (INITIAL INSOMNIA):

| 0 | No difficulty falling asleep |
|---|---|
| 1 | Complains of occasional difficulty falling asleep (i.e., 30 minutes or more, 2-3 nights) |
| 2 | Complains of nightly difficulty falling asleep (i.e., 30 minutes or more, 4 or more nights) |

© 2013, v 1.2 – 24 HR Version. Janet B.W. Williams, PhD  

Since this time yesterday, did you wake up in the middle of your sleep time? IF YES: Did you get out of bed? What did you do? (Only go to the bathroom?)

When you got back in bed, were you able to fall right back asleep? How long did it take you to fall back asleep?

Did you wake up more than once during your sleep time in the past 24 hours? (IF YES: How long did it take for you to fall back to sleep each time?)

Have you felt your sleeping has been restless or disturbed since this time yesterday?

#### 4. INSOMNIA MIDDLE:

| 0 | No difficulty |
|---|---|
| 1 | Complains of being restless and disturbed during the night (or occasional difficulty, i.e., 2-3 nights, 30 minutes or more) |
| 2 | Waking during the night; any getting out of bed (except to void) (often, i.e., 4 or more nights of difficulty, 30 minutes or more) |

# What time did you wake up for the last time, since this time yesterday?

IF EARLY: Is that with an alarm clock, or did you just wake up yourself? What time do you usually wake up (that is, when you feel well)?

#### 5. INSOMNIA LATE (TERMINAL INSOMNIA):

| 0 | No difficulty |
|---|---|
| 1 | Waking in early hours of morning but goes back to sleep (occasional, i.e., 2-3 nights difficulty) |
| 2 | Unable to fall asleep again if gets out of bed (often, i.e., 4 or more nights difficulty) |

Sometimes, along with depression or anxiety, people might lose interest in sex. Since this time yesterday, how has your interest in sex been? (I'm not asking about actual sexual activity, but about your interest in sex.)

Has there been any change in your interest in sex (from when you were feeling OK)?

IF YES: How much less interest have you had in the past 24 hours, compared to when you're not depressed? (Is it a little less or a lot less?)

How has your appetite been since this time yesterday? (What about compared to your usual appetite?)

IF LESS: How much less than usual?

Have you had to force yourself to eat?

Have other people had to urge you to eat? (Have you skipped meals?)

GENITAL SYMPTOMS (such as loss of libido, menstrual disturbances):

| Absent |
|------------------------------------------|
| Mild (somewhat less interest than usual) |
| Severe (a lot less interest than usual) |

#### 7. SOMATIC SYMPTOMS GASTROINTESTINAL:

| 0 | None |
|---|---|
| 1 | Loss of appetite but eating without encouragement (appetite somewhat less than usual) |
| 2 | Difficulty eating without urging (appetite significantly less than usual) |

© 2013, v 1.2 = 24 HR Version. Janet B.W. Williams, PhD 


| Have you lost any weight since this (DEPRESSION) | 0 10 | SS OF WEIGHT |
|---|---|---|
| began? | 8. LO | SS OF WEIGHT |
| IF YES: Do you think you lost any weight in the last 24 | Rate b | by history: |
| hours? (Was it because of feeling depressed or | 0 | No weight loss |
| down?) How much do you think you lost? | 1 | Probable weight loss due to current |
| IF NOT SURE: Do you think your clothes are any | 2 | depression Definite (according to patient) weight loss due |
| looser on you? | * | to depression |
| FOLLOW-UP: Have you gained back any of the weight you've lost since this (DEPRESSION) began? IF YES: How much? | | |
| How has your energy been since this time vesterday? | 9. <b>S</b> O | MATIC SYMPTOMS GENERAL: |
| | 0 | None |
| IF LOW ENERGY: Have you felt tired? (How much of the time? How bad has it been?) | 1 | Heaviness in limbs, back, or head. |
| | | Backaches, muscle aches. Loss of energy and fatigability (somewhat less energy than |
| Since this time yesterday, have you had any aches or pains? (What about backaches or muscle aches?) | | usual, mild, intermittent loss of energy or |
| (How much of the time? How bad has it been?) | 2 | muscle aches/heaviness) Any clear-cut symptoms (persistent, |
| Have you felt any heaviness in your limbs, back, or | 1 | significant loss of energy or muscle |
| head? | | aches/heaviness) |
| Since this time yesterday, have you been putting yourself down, feeling you've done things wrong, | 10. FI | EELINGS OF GUILT: |
| or let others down? | 0 | Absent |
| IF YES: What have your thoughts been? | 1 | Self-reproach; feels he has let people down |
| I land the second secon | 2 | Ideas of guilt or rumination over past errors |
| Have you been feeling guilty about anything that you've done or not done? | | or sinful deeds (feelings of guilt, remorse or shame) |
| IF YES: What have your thoughts been? | 3 | Present illness is a punishment; delusions of guilt (severe, pervasive feelings of guilt) |
| What about things that happened a long time ago? | 4 | Hears accusatory or denunciatory voices and/or experiences threatening visual |
| Have you thought that you've brought (THIS<br>DEPRESSION) on yourself in some way? | | hallucinations |
| (Have you been hearing voices or seeing visions since this time yesterday? IF YES: Tell me about that.) | | |

 $\ \odot$  2013, v 1.2 – 24 HR Version. Janet B.W. Williams, PhD  

| Since this time yesterday, have you had thoughts that life is not worth living? | 11. SU | ICIDE: |
|---|---|---|
| | | Absent |
| What about thinking you'd be better off dead? | 1 | Feels life is not worth living |
| Have you had thoughts of hurting or killing yourself? | 2 | Wishes he were dead or any thoughts of possible death to self |
| IF YES: What have you thought about? Have you | 3 | Suicidal ideas or gesture |
| actually done anything to hurt yourself? | 4 | Attempts at suicide |
| | | O, |
| Have you been feeling anxious or tense since this | 12. AN | XIETY PSYCHIC: |
| time yesterday? IF YES: Is this more than is normal for you? | 0 | No difficulty |
| in 120. Is the more startle hornarier year. | 1 | Subjective tension and irritability (mild. |
| Have you been feeling irritable since this time | | occasional) |
| yesterday? (IF YES): Can you give me some examples? How | 2 | Worrying about minor matters (moderate, causes some distress) |
| bad has it been? | 3 | Apprehensive attitude apparent in face or<br>speech (severe; significant impairment in<br>functioning due to anxiety) |
| Have you been worrying a lot about little things, things you don't ordinarily worry about? IF YES: Like what, for example? | 4 | Fears expressed without questioning (symptoms incapacitating) |
| How about worrying about big problems more than you need to? | | |
| How much of the time has that happened since this time yesterday? | | |
| Has this caused you any problems or difficulties? | | |
| IF YES: Like what, for example? | | |

© 2013, v 1.2 – 24 HR Version. Janet B.W. Williams, PhD  

# Tell me if you've had any of the following physical symptoms since this time yesterday. (READ LIST)

FOR EACH SX ACKNOWLEDGED AS PRESENT: How much has (THE SX) been bothering you since this time yesterday? [How bad has it gotten? How much of the time, or how often, have you had it? Did (the symptom) interfere at all with your functioning or your usual activities?]

NOTE: DO NOT RATE SXS THAT ARE CLEARLY RELATED TO A DOCUMENTED PHYSICAL CONDITION.

13. ANXIETY SOMATIC (physiologic concomitants of

anxiety, such as

GI - dry mouth, gas, indigestion, diarrhea,

stomach cramps, belching
CV - heart palpitations, headaches
Resp - hyperventilating, sighing

Urinary frequency

Sweating):

| Not present |
|---|
| Mild (symptom(s) present only infrequently, no impairment, minimal distress) |
| Moderate (symptom(s) more persistent, or<br>some interference with usual activities,<br>moderate distress) |
| Severe (significant impairment in functioning) |
| Incapacitating |

Since this time yesterday, how much have your thoughts been focused on your physical health or how your body is working (compared to your normal thinking)? (Have you worried a lot about being or becoming physically ill? Have you really been preoccupied with this?)

Have you worried a lot that you have a specific medical illness?

Do you complain much about how you feel physically?

Have you seen a doctor about these problems since this time yesterday? IF YES: What did the doctor say?

# RATING BASED ON OBSERVATION DURING INTERVIEW

# 14. HYPOCHONDRIASIS:

| ľ | 0 | Not present |
|---|---|---|
| | 1 | Self-absorption (bodily) (some inappropriate<br>worry about his/her health OR slightly<br>concerned despite reassurance) |
| | 2 | Preoccupation with health (often has<br>excessive worries about his/her health OR<br>definitely concerned has specific illness<br>despite medical reassurance) |
| | 3 | Frequent complaints, requests for help, etc. (is certain there is a physical problem which the doctors cannot confirm; exaggerated or unrealistic concerns about body and physical health) |
| | 4 | Hypochondriacal delusions |

## 15. INSIGHT:

| Ι. | | |
|---|---|---|
| | 0 | Acknowledges being depressed and ill OR not currently depressed |
| | 1 | Acknowledges illness but attributes cause to bad food, overwork, virus, need for rest, etc. |
| | 2 | Denies being ill at all |

© 2013, v 1.2 – 24 HR Version. Janet B.W. Williams, PhD  

| RATING BASED ON OBSERVATION DURING INTERVIEW | 16. AGITATION: |
|---|---|
| | 0 None |
| IF INTERVIEWING BY PHONE: | Fidgetiness (slight agitation or mild restlessness) |
| During this interview have you been fidgeting a lot or moving around a lot in your chair? | Playing with hands, hair, etc. (moderate to marked restlessness or agitation) |
| Have you had trouble sitting still? | Moving about, can't sit still (cannot remain seated) |
| Have you been shaking your legs or playing with your hair or your hands? | Hand-wringing, nail biting, hair-pulling, biting of lips (interview cannot be conducted; severe agitation) |
| RATING BASED ON OBSERVATION DURING INTERVIEW | RETARDATION (slowness of thought and speech; impaired ability to concentrate; decreased motor activity): |
| IF INTERVIEWING BY PHONE: | delivity). |
| | Normal speech and thought |
| During this interview have you been moving slowly, reacting slowly, or speaking more slowly than usual | Slight retardation at interview (mild psychomotor retardation) |
| for you? | Obvious retardation at interview (moderate; some difficulty with interview, noticeable pauses and slowness of thought) |
| | 3 Interview difficult (severe psychomotor<br>retardation; very long pauses) |
| | Complete stupor (extreme retardation; interview barely possible) |
| $\sim$ | |

| TIME ENDED SIGH-D-17: | AM / PM |
|-----------------------|---------|
| TOTAL HAM-D-17 SCORE: | |

© 2013, v 1.2 – 24 HR Version. Janet B.W. Williams, PhD  

| SIGH-D-17 Feb. 2013

# STRUCTURED INTERVIEW GUIDEFOR THE HAMILTON DEPRESSION RATING SCALE – 17 ITEM VERSION (SIGH-D-17)

Janet B.W. Williams, PhD

### INTERVIEWER

The first question for each item should be asked exactly as written. Often this question will elicit enough information about the severity and frequency of a symptom for you to rate the item with confidence. Follow-up questions are provided for use when further exploration or additional clarification of symptoms is necessary. The specified questions should be asked until you have enough information to rate the item confidently. In some cases, you may also have to add your own follow-up questions to obtain necessary information. You should ask for examples for any symptoms acknowledged as present (e.g., "Can you give me an example of that?"). For some of the HAM-D items, you may find you have already asked about some of the symptoms (for a previous item). You do not need to repeat questions about these symptoms unless you need additional information to rate their severity.

<u>Time period</u>. The interview questions indicate that the ratings should be based on the subject's condition in the past week.

Administration method. This version includes interview questions to help the clinician rate psychomotor agitation and psychomotor retardation, when the interview is administered by telephone. Several research studies have demonstrated that depression scale scores are equivalent whether the scale is administered face-to-face, by telephone, or by video (Williams JBW and Kobak KA: Development and Reliability of a Structured Interview Guide for the Montgomery-Asberg Depression Rating Scale. Br J Psychiatry 192, 52-58, 2008; Kobak KA: A comparison of face-to-face and remote administration of the Hamilton Depression Rating Scale via videoconferencing. J Telemed Telecare 10, 231-235, 2004).

Referent of "usual" or "normal" condition. In the HAM-D, most items are rated positive only if they represent a change from usual functioning. For this reason, several of the interview questions in the HAM-D refer to the subject's usual or normal functioning. The referent should be to the last time they felt okay (i.e., not depressed or high and normal interest in things) for at least two months. When no clear euthymic baseline can be established, one should rate symptomatic behavior as one sees it, even if it is not a change from the subject's usual dysphoric self.

This instrument provides an interview guide for the Hamilton Depression Scale (Hamilton, Max. A rating scale for depression. 
J Neurol Neurosung Psychiat 23:68-61, 1960). The anchor point descriptions for all items except Helplessness, Hopelessness, and Worthlessness, with very minor modifications, have been taken from the ECDEU Assessment Manual (Guy, William, ECDEU Assessment Manual for Psychopharmacology, Revised 1976, DHEW Publication No. (ADM) 76-338). The loss of weight item has been simplified to eliminate the section for ratings by ward staff. A reliability study of the SiGH-D (interview guide for the HAM-D alone) was published in the Archives of General Psychiatry (1988;45:742-747). Additional designators were added in parentheses to the anchor points by Kobak, Lipsitz and Williams to further standardize ratings.

For further information and permission to use or translate the SIGH-D, contact Dr. Williams at jbwwny@gmail.com.

© Janet B.W. Williams, PhD Version 2013.1 

| | ERVIEW GUIDE FOR THE<br>SCALE – 17 ITEM VERSION (SIGH-D-17) |
|---|---|
| SUBJECT'S INITIALS: TI | ME BEGAN SIGH-D: |
| INTERVIEWER: DA | TE:/ |
| OVERVIEW: I'd like to ask you some questions at last (DAY OF WEEK)? IF OUTPATIENT: Have you | pout the past week. How have you been feeling sind been working? IF NOT: Why not? |
| What's your mood been like this past week (compared to when you feel okay)? | DEPRESSED MOOD (sadness, hopeless, helpless, worthless): |
| Have you been feeling down or depressed? | 0 Absent |
| IF YES: Can you describe what this feeling has been like for you? How bad is the feeling? | Indicated only on questioning (occasional, mindepression) Spontaneously reported verbally (persistent, in the control of the control |
| Does the feeling lift at all if something good happens? | to moderate depression) 3 Communicated non-verbally, i.e., facial expression, posture, voice, tendency to weep |
| How are you feeling about the future? | (persistent, moderate to severe depression) |
| IF UNKNOWN: Have you been feeling discouraged or pessimistic? | VIRTUALLY ONLY those feeling states report in spontaneous verbal and non-verbal communication (persistent, very severe) |
| IF YES: What have your thoughts been? | depression, with extreme hopelessness or tearfulness) |
| In the last week, how often have you felt (OWN EQUIVALENT FOR DEPRESSED MOOD)? On how many days? For how long each day? | |
| Have you been crying at all? How often? | |
| <.O, | |
| IF CORED A A POWE ACK, How less have | |
| IF SCORED 1-4 ABOVE, ASK: How long have you been feeling this way (OWN EQUIVALENT FOR DEPRESSED MOOD)? | |

| SIGH-D-17 Feb. 2013

# How have you been spending your time this past week (when not at work)?

Have you felt interested in doing (THOSE THINGS), or do you feel you have to push yourself to do them?

How much less interested in these things have you been this past week compared to when you're not depressed? How hard to do you have to push yourself to do them?

Have you stopped doing anything you used to do? (What about hobbies?) IF YES: Why?

About how many hours a day do you spend doing things that interest you?

Is there anything you look forward to?

IF WORKING (IN OR OUT OF THE HOME): Have you been able to get as much (work) done as you usually do?

How much less productive or efficient are you compared to before you were depressed?

## 2. WORK AND ACTIVITIES:

| 0 | No difficulty |
|---|---|
| 1 | Thoughts and feelings of incapacity, fatigue or weakness related to activities, work or hobbies (mild reduction in interest or pleasure; no clear impairment in functioning) |
| 2 | Loss of interest in activity, hobbies or work -<br>by direct report of the patient or indirect in<br>listlessness, indecision and vacillation (feels<br>he has to push self to work or activities) (clear<br>reduction in interest, pleasure or functioning) |
| 3 | Decrease in actual time spent in activities or decrease in productivity. In hosp., pt. spends less than 3 hrs. (day in activities (hospital job |

- decrease in actual time spent in activities of decrease in productivity. In hosp., pt. spends less than 3 hrs./day in activities (hospital job or hobbies) exclusive of ward chores (profound reduction in interest, pleasure, or functioning)
- Stopped working because of present illness. In hospital, no activities except ward chores, or fails to perform ward chores unassisted (unable to work or fulfill primary role because of illness, and total loss of interest.)

Now let's talk about your sleep. What were your usual hours of going to sleep and waking up, before this began?

When have you been falling asleep and waking up over the past week?

Have you had any trouble falling asleep at the beginning of the night? (Right after you go to bed, how long has it been taking you to fall asleep?)

How many nights this week have you had trouble falling asleep?

Have you changed the time at which you try to get to sleep since you've been depressed?

# 3. INSOMNIA EARLY (INITIAL INSOMNIA):

| ı | 0 | No difficulty falling asleep |
|---|---|---|
| | 1 | Complains of occasional difficulty falling asleep (i.e., 30 minutes or more, 2-3 nights) |
| | 2 | Complains of nightly difficulty falling asleep (i.e., 30 minutes or more, 4 or more nights) |

© Janet B.W. Williams, PhD Version 2013.1


### SIGH-D-17 Feb. 2013

During the past week, have you been waking up in the middle of the night? IF YES: Do you get out of bed? What do you do? (Only go to the bathroom?)

When you get back in bed, are you able to fall right back asleep? How long does it take you to fall back asleep?

Do you wake up more than once during the night? (IF YES: How long does it take for you to fall back to sleep each time?)

Have you felt your sleeping has been restless or disturbed some nights?

How many nights this week have you had that kind of trouble?

### 4. INSOMNIA MIDDLE:

| L | 0 | No difficulty |
|---|---|---|
| | 1 | Complains of being restless and disturbed during the night (or occasional difficulty, i.e., 2-3 nights, 30 minutes or more) |

Waking during the night, any getting out of bed (except to void) (often, i.e., 4 or more nights of difficulty, 30 minutes or more)

# What time have you been waking up in the morning for the last time, this past week?

IF EARLY: Is that with an alarm clock, or do you just wake up yourself? What time do you usually wake up (that is, when you feel well)?

How many mornings this past week have you awakened early?

## 5. INSOMNIA LATE (TERMINAL INSOMNIA):

| 0 | No difficulty |
|---|---|
| 1 | Waking in early hours of morning but goes back to sleep (occasional, i.e., 2-3 nights difficulty) |
| 2 | Unable to fall asleep again if gets out of bed (often, i.e., 4 or more nights difficulty) |

Sometimes, along with depression or anxiety, people might lose interest in sex. This week, how has your interest in sex been? (I'm not asking about actual sexual activity, but about your interest in sex.)

Has there been any change in your interest in sex (from when you were feeling OK)?

IF YES: How much less interest do you have compared to when you're not depressed? (Is it a little less or a lot less?)

How has your appetite been this past week? (What about compared to your usual appetite?)

IF LESS: How much less than usual?

Have you had to force yourself to eat?

Have other people had to urge you to eat? (Have you skipped meals?)

GENITAL SYMPTOMS (such as loss of libido, menstrual disturbances):

| 0 | Absent |
|---|------------------------------------------|
| 1 | Mild (somewhat less interest than usual) |
| 2 | Severe (a lot less interest than usual) |

# 7. SOMATIC SYMPTOMS GASTROINTESTINAL:

| 0 | None |
|---|---|
| 1 | Loss of appetite but eating without encouragement (appetite somewhat less than usual) |
| 2 | Difficulty eating without urging (appetite significantly less than usual) |

© Janet B.W. Williams, PhD Version 2013.1 

| Have you lost any weight since this (DEPRESSION) | 8. LC | DSS OF WEIGHT |
|---|---|---|
| began? IF YES: Did you lose any weight this last week? (Was | | by history: |
| if 1E3. Did you lose any weight this last week? (Was<br>it because of feeling depressed or down?) How much<br>did you lose? | 0 | No weight loss |
| IF NOT SURE: Do you think your clothes are any | 1 | Probable weight loss due to current depression |
| looser on you? | 2 | Definite (according to patient) weight loss du<br>to depression |
| FOLLOW-UP: Have you gained any of the weight back? IF YES: How much? | | -013 |
| How has your energy been this past week? | 9. \$0 | OMATIC SYMPTOMS GENERAL: |
| IF LOW ENERGY: Have you felt tired? (How much of | 0 | None |
| the time? How bad has it been?) This week, have you had any aches or pains? (What about backaches or muscle aches?) (How much of the time? How bad has it been?) | 1 | Heaviness in limbs, back, or head. Backaches, muscle aches. Loss of energy and fatigability (somewhat less energy than usual; mild, intermittent loss of energy or muscle aches/heaviness) |
| Have you felt any heaviness in your limbs, back, or head? | 2 | Any clear-cut symptoms (persistent,<br>significant loss of energy or muscle<br>aches/heaviness) |
| | 1 | |
| Have you been putting yourself down this past week, feeling you've done things wrong, or let | 10. F | FEELINGS OF GUILT: |
| others down? | 0 | Absent |
| IF YES: What have your thoughts been? | 1 | Self-reproach; feels he has let people down |
| Have you been feeling guilty about anything that you've done or not done? | 2 | Ideas of guilt or rumination over past errors<br>or sinful deeds (feelings of guilt, remorse or<br>shame) |
| IF YES: What have your thoughts been? | 3 | Present illness is a punishment; delusions of guilt (severe, pervasive feelings of guilt) |
| What about things that happened a long time ago? | 4 | Hears accusatory or denunciatory voices and/or experiences threatening visual |
| Have you thought that you've brought (THIS | 11 | hallucinations |

 Janet B.W. Williams, PhD Version 2013.1


| SIGH-D-17 Feb. 2013

| This past week, have you had thoughts that life is not worth living? | 11. SUICIDE: | |
|---|---|---|
| not worth nying. | 0 | Absent |
| What about thinking you'd be better off dead? | 1 | Feels life is not worth living |
| Have you had thoughts of hurting or killing vourself? | 2 | Wishes he were dead or any thoughts of possible death to self |
| IF YES: What have you thought about? Have you | 3 | Suicidal ideas or gesture |
| actually done anything to hurt yourself? | 4 | Attempts at suicide |
| Have you been feeling anxious or tense this past<br>week? | 12. AN | XIETY PSYCHIC: |
| IF YES: Is this more than is normal for you? | 0 | No difficulty |
| Have you have feeling instable this past week? | 1 | Subjective tension and irritability (mild, occasional) |
| Have you been feeling irritable this past week? (IF YES): Can you give me some example? How bad has it been? | 2 | Worrying about minor matters (moderate, causes some distress) |
| Have you been worrying a lot about little things, things | 3 | Apprehensive attitude apparent in face or<br>speech (severe; significant impairment in<br>functioning due to anxiety) |
| you don't ordinarily worry about? IF YES: Like what, for example? | | Fears expressed without questioning (symptoms incapacitating) |
| How about worrying about big problems more than you need to? | | |
| How much of the time has that happened this week? | | |
| Has this caused you any problems or difficulties? IF YES: Like what, for example? | | |

© Janet B.W. Williams, PhD Version 2013.1 

#### | SIGH-D-17 Feb. 2013 Tell me if you've had any of the following physical 13. ANXIETY SOMATIC (physiologic concomitants of symptoms in the past week. (READ LIST) anxiety, such as GI dry mouth, gas, indigestion, diarrhea, FOR EACH SX ACKNOWLEDGED AS PRESENT: stomach cramps, belching How much has (THE SX) been bothering you this CV heart palpitations, headaches past week? [How bad has it gotten? How much of Resp hyperventilating, sighing the time, or how often, have you had it? Did (the Urinary frequency symptom) interfere at all with your functioning or your Sweating): Not present 0 NOTE: DO NOT RATE SXS THAT ARE CLEARLY Mild (symptom(s) present only infrequently, RELATED TO A DOCUMENTED PHYSICAL no impairment, minimal distress) CONDITION. Moderate (symptom(s) more persistent, or 2 some interference with usual activities, moderate distress) Severe (significant impairment in 3 functioning) 4 Incapacitating 14. HYPOCHONDRIASIS: In the last week, how much have your thoughts been focused on your physical health or how your body is working (compared to your normal 0 Not present thinking)? (Have you worried a lot about being or Self-absorption (bodily) (some inappropriate becoming physically ill? Have you really been worry about his/her health OR slightly preoccupied with this?) concerned despite reassurance) Have you worried a lot that you have a specific Preoccupation with health (often has medical illness? excessive worries about his/her health OR definitely concerned has specific illness Do you complain much about how you feel physically? despite medical reassurance) Frequent complaints, requests for help, etc. Have you seen a doctor about these problems? (is certain there is a physical problem which IF YES: What did the doctor say? the doctors cannot confirm; exaggerated or unrealistic concerns about body and physical health) Hypochondriacal delusions 4 RATING BASED ON OBSERVATION DURING 15. INSIGHT: INTERVIEW Acknowledges being depressed and ill OR not currently depressed Acknowledges illness but attributes cause to bad food, overwork, virus, need for rest, Denies being ill at all

@ Janet B.W. Williams, PhD Version 2013.1


| RATING BASED ON OBSERVATION DURING INTERVIEW | 16. AGITATION: |
|---|---|
| | 0 None |
| IF INTERVIEWING BY PHONE: | Fidgetiness (slight agitation or mild restlessness) |
| During this interview have you been fidgeting a lot or moving around a lot in your chair? | Playing with hands, hair, etc. (moderate to marked restlessness or agitation) |
| Have you had trouble sitting still? | Moving about, can't sit still (cannot remain seated) |
| Have you been shaking your legs or playing with your hair or your hands? | 4 Hand-wringing, nail biting, hair-pulling, biting of lips (interview cannot be conducted; severe agitation) |
| RATING BASED ON OBSERVATION DURING INTERVIEW | 17. RETARDATION (slowness of thought and speech;<br>impaired ability to concentrate; decreased motor<br>activity): |
| IF INTERVIEWING BY PHONE: | |
| | Normal speech and thought |
| During this interview have you been moving slowly,<br>reacting slowly, or speaking more slowly than usual<br>for you? | Slight retardation at interview (mild psychomotor retardation) |
| tor you? | Obvious retardation at interview (moderate; some difficulty with interview, noticeable pauses and slowness of thought) |
| | 3 Interview difficult (severe psychomotor retardation; very long pauses) |
| | Complete stupor (extreme retardation; interview barely possible) |

| TIME ENDED SIGH-D-17: | AM / PM |
|-----------------------|---------|
| TOTAL HAM-D-17 SCORE: | |

© Janet B.W. Williams, PhD Version 2013.1 

# Appendix 2. MONTGOMERY-ÅSBERG DEPRESSION RATING SCALE (MADRS)

## STRUCTURED INTERVIEW GUIDE FOR THE MONTGOMERY AND ASBERG DEPRESSION RATING SCALE (SIGMA) – 24 HR TWENTY-FOUR HOUR ASSESSMENT VERSION

Janet B.W. Williams, Ph.D. and Kenneth A. Kobak, Ph.D.

INTERVIEWING GUIDELINES: The questions in bold for each item should be asked exactly as written unless the information has been previously obtained, in which case it is appropriate to restate the information for confirmation. Follow-up questions are provided for use when further exploration or additional clarification of symptoms is necessary. The specified questions should be asked until you have enough information to rate the item confidently. In some cases, you may also have to add your own follow-up questions to obtain necessary information. Note that questions in parentheses are optional, for use, for example, if information is unknown. Statements in ALL CAPITALS are interviewer instructions and should not be read to the subject.

RATING GUIDELINES: Ratings should be based on the subject's condition as observed over the past 24 hours. As specified in the item descriptions, three of the items, Reduced Sleep, Reduced Appetite, and Inability to Feel, are rated as present only when they reflect a change from before the depression began (EUTHYMIC BASELINE). In most cases, this version will be used after the original Past Week version of the scale, during which a euthymic baseline (the most recent 2-month period of non-depressed functioning) was established. The interviewer for this 24-hour version should use this euthymic baseline as a reference point for the Reduced Sleep, Reduced Appetite, and Inability to Feel items. When a clear euthymic baseline has not been established because of chronic depressive symptoms, these three items should be rated as observed over the past 24 hours instead of as compared to a previous time point.

This interview guide is based on the Montgomery-Asberg Depression Rating Scale (MADRS) (Montgomery SA, Asberg M: A new depression scale designed to be sensitive to change. *Br J Psychiatry*; 1979 **134:** 382-9). The scale itself has been retained in its original form, except for reversing the order of the first two items. This guide adds interview questions to aid in the assessment and application of the MADRS. Previous versions of this guide appeared in 1988, 1992, 1996, 2005 and 2008. This version of the SIGMA has been designed for assessments that capture a 24-hour time frame. A 4-hour version and a Since Last Evaluation version have also been designed for studies needing to capture assessments over those time periods.

©2008, 2011 The Royal College of Psychiatrists. The SIGMA may be copied by individual researchers or clinicians for their own use without seeking permission from the publishers. The scale must be copied in full and all copies must acknowledge the following source: Williams JBW, Kobak KA. Development and reliability of a structured interview guide for the Montgomery-Asberg Depression Rating Scale (SIGMA). Br J Psychiatry 2008;192:52-58. Brianne Brown, PsyD, contributed to this revision. Written permission must be obtained from the Royal College of Psychiatrists for copying, distribution to others, for replication (in print, online or by any other medium), and translations. Scientific correspondence should be addressed to Dr. Janet Williams at <a href="mailto:jbwwny@gmail.com">jbwwny@gmail.com</a>. To inform an ongoing survey, researchers and clinicians are asked to notify Dr. Williams of their intention to use the SIGMA.

# STRUCTURED INTERVIEW GUIDE FOR THE MONTGOMERY AND ASBERG DEPRESSION RATING SCALE (SIGMA) – 24 HR TWENTY-FOUR HOUR ASSESSMENT VERSION

| TWENTY-FOUR HOUR ASSESSMENT VERSION | |
|---|---|
| PT'S INITIALS: PT'S ID: | TIME BEGAN SIGMA: AM / PM |
| INTERVIEWER: | DATE: |
| OVERVIEW: I'd like to ask you some questions about the past 24 hours. How have you been feeling since this time yesterday? IF OUTPATIENT: Have you been working? (What kind of work do you do? Have you been able to work your normal hours?) IF NOT WORKING OR WORKING LESS, CLARIFY WHY. | |
| Since this time yesterday, have you been feeling sad or<br>unhappy? (Depressed at all?) IF YES: Can you describe<br>what this has been like for you? (IF UNKNOWN: How<br>bad has that been?) | <ol> <li>REPORTED SADNESS. Representing reports of depressed<br/>mood, regardless of whether it is reflected in appearance or not.<br/>Includes low spirits, despondency or the feeling of being beyond<br/>help and without hope. Rate according to intensity, duration, and<br/>the extent to which the mood is reported to be influenced by</li> </ol> |
| IF DEPRESSED: Does the feeling lift at all if something good happens? How much does your mood lift? Does the feeling ever go away completely? (How often have you had lifts in your mood since this time yesterday? What things have made you feel better?) How often did you feel (depressed/OWN EQUIVALENT) since this time yesterday? (IF UNKNOWN: How much of the time have you felt that way since this time yesterday?) Since this time yesterday, how have you been feeling | events. 0 - Occasional sadness in keeping with the circumstances. 1 - 2 - Sad or low but brightens up without difficulty. 3 - 4 - Pervasive feelings of sadness or gloominess. The mood is still influenced by external circumstances. 5 - 6 - Continuous or unvarying sadness, misery, or despondency. |
| about the future? (Have you been discouraged or pessimistic?) What have your thoughts been? How (discouraged or pessimistic) have you been? How often have you felt that way since this time yesterday? Do you think things will ever get better for you? | |
| INTERVIEWER: REVIEW DATE OF EUTHYMIC BASELINE (When was the last time you were well, not depressed at all, for at least 2 months?) | |

© 2011, v.1.2 - 24 hr. version. The Royal College of Psychiatrists  

# RATING BASED ON OBSERVATION DURING INTERVIEW AND THE FOLLOWING QUESTIONS.

Since this time yesterday, do you think you have looked sad or depressed to other people? Did anyone say you looked sad or down?

How about when you've looked in the mirror - did you look gloomy or depressed?

IF YES: How sad or depressed do you think you have looked? How much of the time since this time yesterday do you think you have looked depressed or down?

Has it been hard for you to laugh or smile since this time yesterday?

- APPARENT SADNESS. Representing despondency, gloom and despair. (More than just ordinary transient low spirits) reflected in speech, facial expressions, and posture. Rate by depth and inability to brighten up.
- 0 No sadness
- 1 –
- 2 Looks dispirited but does brighten up without difficulty.
- 3 -
- 4 Appears sad and unhappy most of the time.
- 5 -
- 6 Looks miserable all the time. Extremely despondent

# Have you felt tense or edgy over the past 24 hours, since yesterday at this time? Have you felt anxious or nervous?

IF YES: Can you describe what that has been like for you? How bad has it been?

What about feeling fearful that something bad is about to happen?

How much of the time have you felt (anxious/tense/OWN EQUIVALENT) since this time yesterday?

Have you felt panicky since this time yesterday? IF YES: Can you describe this feeling? How often have you felt this way since yesterday at this time?

IF YES TO ANY TENSION SYMPTOM: How hard has it been to control these feelings? (What has it taken to help you feel calmer? Has anything worked to calm you down?)

INNER TENSION. Representing feelings of ill-defined discomfort, edginess, inner turmoil, mental tension mounting to either panic, dread, or anguish. Rate according to intensity, frequency, duration and the extent of reassurance called for.

- 0 Placid. Only fleeting inner tension.
- 2 Occasional feelings of edginess and ill-defined discomfort.
- 4 Continuous feelings of inner tension or intermittent panic
- which the patient can only master with some difficulty.
- 6 Unrelenting dread or anguish. Overwhelming panic.

# How has your sleeping been in the past 24 hours? (How many hours did you sleep, compared to usual?)

Did you have trouble falling asleep since this time yesterday? (How long did it take you to fall asleep in the past 24 hours? How does that compare to your usual pattern?)

In the past 24 hours were you able to stay asleep through the night? (Did you wake up at all in the middle of the night? How long did it take you to fall back to sleep? How does that compare to EUTHYMIC BASELINE?)

In the past 24 hours did you awaken earlier than (EUTHYMIC BASELINE)?

IF UNKNOWN: Has your sleeping been restless or disturbed since this time yesterday?

- REDUCED SLEEP. Representing the experience of reduced duration or depth of sleep compared to the subject's own normal pattern when well.
- 0 Sleeps as usual.
- 1 -
- Slight difficulty dropping off to sleep or slightly reduced, light, or fitful sleep.
- 4 Sleep reduced or broken by at least 2 hours.
- 6 Less than 2 or 3 hours sleep.

© 2011, v.1.2 – 24 hr. version. The Royal College of Psychiatrists 


How has your appetite been since this time yesterday? (What about compared to your usual appetite?)

IF NOT REDUCED: Have you been less interested in food compared to (EUTHYMIC BASELINE)? (How much less?)

Does food taste as good as usual (compared to EUTHYMIC BASELINE)? IF LESS: How much less? Does it have any taste at all?

(Have you had to push yourself to eat or have other people had to urge you to eat over the past 24 hours?)

5. REDUCED APPETITE. Representing the feeling of a loss of appetite compared with when well. Rate by loss of desire for food or the need to force oneself to eat.

- 0 Normal or increased appetite.
- \_
- 2 Slightly reduced appetite.
- 4 No appetite. Food is tasteless.
  - 110 appente. 1 cou is
- 6 Needs persuasion to eat at all.

Have you had trouble concentrating or collecting your thoughts since this time yesterday? (How about at home or at work?) IF YES: Can you give me some examples? (Have you been able to concentrate on reading a book or on the computer? Do you need to read things over and over again? Are you able to follow movies or television?)

How often has that happened since this time yesterday? Has this caused any problems for you?

Have you had any trouble following a conversation? (IF YES: How bad has that been? How often has that happened since this time yesterday?)

NOTE: ALSO CONSIDER BEHAVIOR DURING INTERVIEW.

 CONCENTRATION DIFFICULTIES. Representing difficulties in collecting one's thoughts mounting to incapacitating lack of concentration. Rate according to intensity, frequency, and degree of incapacity produced.

- 0 No difficulties in concentration.
- 1 -
- 2 Occasional difficulties in collecting one's thoughts.
- 4 Difficulties in concentrating and sustaining thought which
- reduces ability to read or hold a conversation.
- 6 Unable to read or converse without great difficulty.

Have you had any trouble getting started at things since this time yesterday? IF YES: What things? How bad has that been?

Have you had difficulty getting started at simple routine everyday things (like getting dressed, brushing your teeth, showering)?

Since this time yesterday, have you been OK once you get started at things or has it still been more of an effort to get something done?

Has there been anything that you needed to do in the past 24 hours that you were unable to do? Have you needed help to do things? IF YES: What things? How often?

Have you done everyday things more slowly than usual since this time yesterday? IF YES: Like what, for example? How bad has that been?

- LASSITUDE. Representing a difficulty getting started, or slowness initiating and performing everyday activities.
- 0 Hardly any difficulty in getting started. No sluggishness.
- Difficulties in starting activities.
- 3 –
- $4-\mbox{Difficulties}$  in simple routine activities, which are carried out with effort.
- \_
- 6 Complete lassitude. Unable to do anything without help.

© 2011, v.1.2 – 24 hr. version. The Royal College of Psychiatrists  

89

Over the last 24 hours, have you been less interested in things around you, or in activities you used to enjoy, compared to (EUTHYMIC BASELINE)? IF YES: What things? How much less interested are you in (those things), compared to (EUTHYMIC BASELINE)?

What things have you enjoyed over the past 24 hours? How much did you enjoy them?

Has there been any change in your ability to feel emotions since (EUTHYMIC BASELINE)? (Do you feel things less intensely than you used to, things like anger, grief, pleasure?) IF YES: Can you tell me more about that? (IF UNKNOWN: Are you able to feel any emotions at all?)

Have your feelings towards family and friends changed at all since (EUTHYMIC BASELINE)? IF YES: Do you feel less towards them than you used to (AT EUTHYMIC BASELINE)?

8. INABILITY TO FEEL. Representing the subjective experience of reduced interest in the surroundings, or activities that normally give pleasure. The ability to react with adequate emotion to circumstances or people is reduced.

- 0 Normal interest in the surroundings and in other people.
- 2 Reduced ability to enjoy usual interests.
- 4 Loss of interest in the surroundings. Loss of feelings for friends and acquaintances.
- 6 The experience of being emotionally paralyzed, inability to feel anger, grief or pleasure, and a complete or even painful failure to feel for close relatives and friends.

Have you been putting yourself down, or feeling that you're a failure in some way, since this time yesterday? (Have you been blaming yourself for things that you've done, or not done?) IF YES: What have your thoughts been? How often have you felt that way?

Since this time yesterday have you been feeling guilty about anything? What about feeling as if you have done something bad or sinful? IF YES: What have your thoughts been? How often have you felt that way over the

ALSO CONSIDER RESPONSES TO QUESTIONS ABOUT PESSIMISM FROM ITEM 1.

9. PESSIMISTIC THOUGHTS. Representing thoughts of guilt, inferiority, self-reproach, sinfulness, remorse, and ruin.

- 0 No pessimistic thoughts.
- 2 Fluctuating ideas of failure, self-reproach, or self-depreciation.
- 4 Persistent self-accusations, or definite but still rational ideas of guilt or sin. Increasingly pessimistic about the future.

Delusions of ruin, remorse, or unredeemable sin. Selfaccusations which are absurd and unshakeable.

© 2011, v.1.2 - 24 hr. version. The Royal College of Psychiatrists  

Since this time yesterday, have you felt like life isn't worth living? (IF NO: What about feeling as if you're tired

of living?)
IF YES: Tell me about that. How often have you felt that way since this time yesterday?

Since this time yesterday, have you thought that you would be better off dead? IF YES: Tell me about that. How often have you felt that way since this time yesterday?

Have you had thoughts of hurting or even killing yourself since this time yesterday? IF YES: What have you thought about? How often have you had these thoughts since this time yesterday? How long have they lasted? Have you actually made plans? IF YES: What are these plans? Have you made any preparations to carry out these plans? (Have you told anyone about it?)

10. SUICIDAL THOUGHTS. Representing the feeling that life is not worth living, that a natural death would be welcome, suicidal thoughts, and preparation for suicide. Suicidal attempts should not in themselves influence this rating.

- 0 Enjoys life or takes it as it comes.
- 2 Weary of life. Only fleeting suicidal thoughts.
- 3 4 Probably better off dead. Suicidal thoughts are common, and suicide is considered as a possible solution, but without specific plans or intention.
- 6 Explicit plans for suicide when there is an opportunity. Active preparations for suicide.

| TIME ENDED SIGMA: | AM / PM |
|--------------------------|---------|
| TOTAL MADRS SCALE SCORE: | |

© 2011, v.1.2 - 24 hr. version. The Royal College of Psychiatrists  

COL

# STRUCTURED INTERVIEW GUIDE FOR THE MONTGOMERY AND ASBERG DEPRESSION RATING SCALE (SIGMA)

Janet B.W. Williams, Ph.D. and Kenneth A. Kobak, Ph.D.

INTERVIEWING GUIDELINES: The questions in bold for each item should be asked exactly as written unless the information has been previously obtained, in which case it is appropriate to restate the information for confirmation. Follow-up questions are provided for use when further exploration or additional clarification of symptoms is necessary. The specified questions should be asked until you have enough information to rate the item confidently. In some cases, you may also have to add your own follow-up questions to obtain necessary information. Note that questions in parentheses are optional, for use, for example, if information is unknown. Statements in ALL CAPITALS are interviewer instructions and should not be read to the subject.

RATING GUIDELINES: Ratings should be based on the subject's condition as observed in the past week (past 7 days). As specified in the item descriptions, three of the items, Reduced Sleep, Reduced Appetite, and Inability to Feel, are rated as present only when they reflect a change from before the depression began (EUTHYMIC BASELINE). The interviewer should attempt to identify the most recent 2-month period of non-depressed functioning and use this as a reference point. In some cases, such as when the subject has dysthymia, the referent should be to the last time the subject felt alright (i.e., not depressed or high) for at least a few weeks. When a clear euthymic baseline cannot be established because of chronic depressive symptoms, these items should be rated as observed over the past 7 days instead of comparing to a previous time point.

This interview guide is based on the Montgomery-Asberg Depression Rating Scale (MADRS) (Montgomery SA, Asberg M: A new depression scale designed to be sensitive to change. <u>Br J Psychiatry</u>; 1979 **134**: 382-9). The scale itself has been retained in its original form, except for reversing the order of the first two items. This guide adds interview questions to aid in the assessment and application of the MADRS. Previous versions of this guide appeared in 1988, 1992, 1996, 2005 and 2008.

©2008, 2011v1.2 The Royal College of Psychiatrists. The scale must be copied in full and all copies must acknowledge the following source: Williams JBW, Kobak KA. Development and reliability of a structured interview guide for the Montgomery-Asberg Depression Rating Scale (SIGMA). Br J Psychiatry 2008; 192: 52-58. Brianne Brown, PsyD, contributed to this revision. Written permission must be obtained from the Royal College of Psychiatrists for copying, distribution to others, for replication (in print, online or by any other medium), and translations. Scientific correspondence should be addressed to Dr. Janet Williams at <a href="https://documbia.edu">https://documbia.edu</a>. To inform an ongoing survey, researchers and clinicians are asked to notify Dr. Williams of their intention to use the SIGMA.

## STRUCTURED INTERVIEW GUIDE FOR THE MONTGOMERY AND ASBERG DEPRESSION RATING SCALE (SIGMA)

| MONTGOMERY AND ASBERG DEPRESSION RATING SCALE (SIGMA) | |
|---|---|
| PT'S INITIALS: PT'S ID: | TIME BEGAN SIGMA: AM / PM |
| INTERVIEWER: | DATE: |
| OVERVIEW: I'd like to ask you some questions about the past week. Ho IF OUTPATIENT: Have you been working? (What kind of w NOT WORKING OR WORKING LESS, CLARIFY WHY. | ork do you do? Have you been able to work your normal hours?) IF |
| In the past week, have you been feeling sad or unhappy? (Depressed at all?) IF YES: Can you describe what this has been like for you? (IF UNKNOWN: How bad has that been?) IF DEPRESSED: Does the feeling lift at all if something good happens? How much does your mood lift? Does the feeling ever go away completely? (How often have you had lifts in your mood this week? What things have made you feel better?) How often did you feel (depressed/OWN EQUIVALENT) this past week? (IF UNKNOWN: How many days this week did you feel that way? How much of each day?) In the past week, how have you been feeling about the future? (Have you been discouraged or pessimistic?) What have your thoughts been? How (discouraged or pessimistic) have you been? How often have you felt that way? Do you think things will ever get better for you? ESTABLISH EUTHYMIC BASELINE: When was the last time you were well, not depressed at all, for at least 2 months? | 1. REPORTED SADNESS. Representing reports of depressed mood, regardless of whether it is reflected in appearance or not. Includes low spirits, despondency or the feeling of being beyond help and without hope. Rate according to intensity, duration, and the extent to which the mood is reported to be influenced by events. 0 - Occasional sadness in keeping with the circumstances. 1 - 2 - Sad or low but brightens up without difficulty. 3 - 4 - Pervasive feelings of sadness or gloominess. The mood is still influenced by external circumstances. 5 - 6 - Continuous or unvarying sadness, misery, or despondency. |

© 2011, v.1.2, The Royal College of Psychiatrists  

### RATING BASED ON OBSERVATION DURING INTERVIEW AND THE FOLLOWING QUESTIONS.

In the past week, do you think you have looked sad or depressed to other people? Did anyone say you looked sad or down?

How about when you've looked in the mirror; did you look gloomy or depressed?

IF YES: How sad or depressed do you think you have looked? How much of the time over the past week do you think you have looked depressed or down?

Has it been hard for you to laugh or smile in the past week?

- 2. APPARENT SADNESS. Representing despondency, gloom and despair. (More than just ordinary transient low spirits) reflected in speech, facial expressions, and posture. Rate by depth and inability to brighten up.
- 0 No sadness
- 2 Looks dispirited but does brighten up without difficulty. 3 -
- 4 Appears sad and unhappy most of the time.
- 6 Looks miserable all the time. Extremely despondent.

### Have you felt tense or edgy in the last week? Have you felt anxious or nervous?

IF YES: Can you describe what that has been like for you? How bad has it been?

What about feeling fearful that something bad is about

How much of the time have you felt (anxious/tense/OWN EQUIVALENT) over the past week?

Have you felt panicky in the past week? IF YES: Can you describe this feeling? How often have you felt this

IF YES TO ANY TENSION SYMPTOM: How hard has it been to control these feelings? (What has it taken to help you feel calmer? Has anything worked to calm you down?)

3. INNER TENSION. Representing feelings of ill-defined discomfort, edginess, inner turmoil, mental tension mounting to either panic, dread, or anguish. Rate according to intensity, frequency, duration and the extent of reassurance called for.

- 0 Placid. Only fleeting inner tension.
- 2 Occasional feelings of edginess and ill-defined discomfort.
- 4 Continuous feelings of inner tension or intermittent panic which the patient can only master with some difficulty.
- 6 Unrelenting dread or anguish. Overwhelming panic.

# How has your sleeping been in the last week? (How many hours have you been sleeping, compared to

Have you had trouble falling asleep? (How long has it been taking you to fall asleep this past week? How many

Have you been able to stay asleep through the night? (Have you been waking up at all in the middle of the night? How long does it take you to fall back to sleep? How many

Have there been any mornings this past week when you have awakened earlier than (EUTHYMIC BASELINE)?

IF UNKNOWN: Has your sleeping been restless or disturbed?

- 4. REDUCED SLEEP. Representing the experience of reduced duration or depth of sleep compared to the subject's own normal pattern when well.
- 0 Sleeps as usual.
- 2 Slight difficulty dropping off to sleep or slightly reduced, light, or fitful sleep. 3 -
- 4 Sleep reduced or broken by at least 2 hours.
- 6 Less than 2 or 3 hours sleep.

© 2011, v.1.2, The Royal College of Psychiatrists  

How has your appetite been this past week? (What about compared to your usual appetite?)

IF NOT REDUCED: Have you been less interested in food? (How much less?)

Does food taste as good as usual? IF LESS: How much less? Does it have any taste at all?

(Have you had to push yourself to eat or have other people had to urge you to eat?)

5. REDUCED APPETITE. Representing the feeling of a loss of appetite compared with when well. Rate by loss of desire for food or the need to force oneself to eat.

- 0 Normal or increased appetite.
- 1 -
- 2 Slightly reduced appetite.
- 4 No appetite. Food is tasteless.
- 5 -
- 6 Needs persuasion to eat at all.

Have you had trouble concentrating or collecting your thoughts in the past week? (How about at home or at work?) IF YES: Can you give me some examples? (Have you been able to concentrate on reading a book or on the computer? Do you need to read things over and over again? Are you able to follow movies or television?)

How often has that happened in the past week? Has this caused any problems for you?

Have you had any trouble following a conversation? (IF YES: How bad has that been? How often has that happened this past week?)

NOTE: ALSO CONSIDER BEHAVIOR DURING INTERVIEW.

 CONCENTRATION DIFFICULTIES. Representing difficulties in collecting one's thoughts mounting to incapacitating lack of concentration. Rate according to intensity, frequency, and degree of incapacity produced.

- 0 No difficulties in concentration.
- 2 Occasional difficulties in collecting one's thoughts.
  - 5-mm 10-1
- 4 Difficulties in concentrating and sustaining thought which reduces ability to read or hold a conversation.
- 6 Unable to read or converse without great difficulty.

Have you had any trouble getting started at things in the past week? IF YES: What things? How bad has that been? Have you had difficulty getting started at simple routine everyday things (like getting dressed, brushing your teeth, showering)?

Are you OK once you get started at things or is it still more of an effort to get something done?

Has there been anything that you needed to do that you were unable to do? Have you needed help to do things? IF YES: What things? How often?

Have you done everyday things more slowly than usual? IF YES: Like what, for example? How bad has that been?

LASSITUDE. Representing a difficulty getting started, or slowness initiating and performing everyday activities.

- 0 Hardly any difficulty in getting started. No sluggishness.
- 2 Difficulties in starting activities.
- 3 –
- 4 Difficulties in simple routine activities, which are carried out with effort.
  - \_
- 6 Complete lassitude. Unable to do anything without help.

© 2011, v.1.2, The Royal College of Psychiatrists  

Have you been less interested in things around you, or in activities you used to enjoy? IF YES: What things? How much less interested in (those things) are you now compared to (EUTHYMIC BASELINE)?

What things have you enjoyed this week? How much did you enjoy them?

Has there been any change in your ability to feel emotions? (Do you feel things less intensely than you used to, things like anger, grief, pleasure?) IF YES: Can you tell me more about that? (IF UNKNOWN: Are you able to feel any emotions at all?)

Have your feelings towards family and friends changed at all? IF YES: Do you feel less towards them than you used to?

- 8. INABILITY TO FEEL. Representing the subjective experience of reduced interest in the surroundings, or activities that normally give pleasure. The ability to react with adequate emotion to circumstances or people is reduced
- 0 Normal interest in the surroundings and in other people.
- 2 Reduced ability to enjoy usual interests.
- 3 -
- 4 Loss of interest in the surroundings. Loss of feelings for friends and acquaintances.
- 6 The experience of being emotionally paralyzed, inability to feel anger, grief or pleasure, and a complete or even painful failure to feel for close relatives and friends.

Have you been putting yourself down, or feeling that you're a failure in some way, over the past week? (Have you been blaming yourself for things that you've done, or not done?) IF YES: What have your thoughts been? How often have you felt that way?

In the past week have you been feeling guilty about anything? What about feeling as if you have done something bad or sinful? IF YES: What have your thoughts been? How often have you felt that way?

ALSO CONSIDER RESPONSES TO QUESTIONS ABOUT PESSIMISM FROM ITEM 1.

9. PESSIMISTIC THOUGHTS. Representing thoughts of guilt, inferiority, self-reproach, sinfulness, remorse, and ruin.

- 0 No pessimistic thoughts
- 2 Fluctuating ideas of failure, self-reproach, or self-depreciation.
- 4 Persistent self-accusations, or definite but still rational ideas of guilt or sin. Increasingly pessimistic about the future.
- 6 Delusions of ruin, remorse, or unredeemable sin. Selfaccusations which are absurd and unshakeable.

This past week, have you felt like life isn't worth living? (IF NO: What about feeling as if you're tired of living?) IF YES: Tell me about that. How often have you felt that

This week, have you thought that you would be better off dead? IF YES: Tell me about that. How often have you felt that way?

Have you had thoughts of hurting or even killing yourself this past week? IF YES: What have you thought about? How often have you had these thoughts? How long have they lasted? Have you actually made plans? IF YES: What are these plans? Have you made any preparations to carry out these plans? (Have you told anyone about it?)

10. SUICIDAL THOUGHTS. Representing the feeling that life is not worth living, that a natural death would be welcome, suicidal thoughts, and preparation for suicide. Suicidal attempts should not in themselves influence this rating.

- 0 Enjoys life or takes it as it comes.
- 2 Weary of life. Only fleeting suicidal thoughts.
- 4 Probably better off dead. Suicidal thoughts are common, and suicide is considered as a possible solution, but without specific plans or intention.

6 - Explicit plans for suicide when there is an opportunity. Active preparations for suicide.

| TIME ENDED SIGMA: | AM / PM |
|--------------------------|---------|
| TOTAL MADRS SCALE SCORE: | |

© 2011, v.1.2, The Royal College of Psychiatrists  

# APPENDIX 3. HAMILTON ANXIETY RATING SCALE (HAM-A)

# STRUCTURED INTERVIEW GUIDE FOR THE HAMILTON ANXIETY SCALE (SIGH-A) – 24 HR TWENTY-FOUR HOUR ASSESSMENT VERSION

Janet B.W. Williams, PhD

INTERVIEWER: The first question for each item, in bold type, should be asked exactly as written. For each symptom endorsed, use the additional probes at the top of each page to determine the frequency and severity of the symptom, including how bad it's been, how much distress it has caused, and if the symptom has caused any impairment. Follow-up questions are provided for use when further exploration or additional clarification of symptoms is necessary. The specified questions should be asked until you have enough information to rate the item confidently. In some cases, you may also have to add your own follow-up questions to obtain necessary information. You should ask for examples for any symptoms acknowledged as present (e.g., "Can you give me an example of that?"). For some of the HAM-A items, you may find you have already asked about some of the symptoms (for a previous item). You do not need to repeat questions about these symptoms unless you need additional information to rate their severity.

All of the items have the same anchor points. The following may be useful as a guide to rating item severity:

ABSENT Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety

MILD Score 1 if symptom is infrequent, with no impairment and

no more than mild distress

MODERATE Score 2 if symptom is more frequent, with moderate distress or limited interference with usual activities

SEVERE Score 3 if symptom is severe and persistent or results in severe distress or marked impairment in functioning

VERY SEVERE Score 4 if symptom is incapacitating

For each symptom, ask:

- Tell me what that was like. Can you give me some examples?
- · How bad has this been over the past week?
- How much has it bothered you? Has it caused you any problems?
- . How much of the time or how often have you had this over the past week?

# NOTES

<u>Time period</u>. For this 24 hour version, the ratings should be based on the patient's condition over the past 24 hours. Unlike the HAMD, change from usual self is not required for most items to be rated positively on the HAMA. However, symptoms should not be rated positively if they are clearly due to a cause unrelated to anxiety, e.g., respiratory symptoms due to pneumonia.

<u>Panic attacks</u>. If the patient has panic attacks, this could affect the ratings of many of the symptoms. It is recommended that you consider the total amount of time during the past 24 hours that the panic attack symptoms occurred, as well as their severity. For example, a patient who has several severe but short-lived panic attacks during the past 24 hours, even if they otherwise do not have many anxiety symptoms, would probably have a high total HAM-A score.

This instrument provides an interview guide for the Hamilton Anxiety Scale (Hamilton M: The assessment of anxiety states by rating. Brit J Med Psychol 32:60-56, 1959; Hamilton M: The diagnosis and rating of anxiety. In Studies of Anxiety. MH Lader, Ed., Headley Bros., Kent, 1969). The anchor point descriptions for the scale have been taken from the ECDEU Assessment Manual (Guy, William, ECDEU Assessment Manual for Psychopharmacology, Revised 1976, DHEW Publication No. (ADM) 76-339), except that "sighing" and "dyspnea," which appear twice in that version, have been taken out of the item "cardiovascular symptoms," and remain under "respiratory symptoms." Kenneth A. Kobak, PhD and Joshua D. Lipsitz, PhD contributed to revisions of this interview guide.

For further information and permission to use or translate the SIGH-A, contact Dr. Williams at <a href="mailto:jbwwny@gmail.com">jbwwny@gmail.com</a>. SIGH-A 2013, v1.2 – 24 HR Version. Janet B.W. Williams, PhD  

# STRUCTURED INTERVIEW GUIDE FOR THE HAMILTON ANXIETY SCALE (SIGH-A) – 24 HR TWENTY-FOUR HOUR ASSESSMENT VERSION

| PT'S INITIALS: PT'S ID: | TIME BEGAN SIGH-A: | AM / PM |
|-------------------------|--------------------|--------------|
| | | ET / CT / PT |
| INTERVIEWER: | DATE:// | |

**OVERVIEW**: I'd like to ask you some questions about the past 24 hours. How have you been feeling since this time yesterday? IF OUTPATIENT: Have you been working? IF NOT: Why not?

Suggested follow-up questions:

- Tell me what that was like. Can you give me some examples?
- How bad has this been since this time yesterday?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this since this time yesterday?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent or<br>results in severe distress or marked impairment<br>in functioning |
| VERY SEVERE | Symptom is incapacitating |

Since this time yesterday, how much have you been worrying? (What have you been worried about? How hard has it been to stop worrying?)

(IF UNKNOWN): How much have you been afraid that the worst is going to happen?

Have you been feeling nervous or anxious since this time yesterday?

Have you been feeling irritable since this time yesterday?

# 1. ANXIOUS MOOD

(worries, anticipation of the worst, fearful anticipation, irritability):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

IF SCORED 1-4 ABOVE, FOR CONTEXT, ASK: How long have you been feeling this way?

 $\ \odot$  SIGH-A 2013, v1.2 – 24 HR Version. Janet B.W. Williams, PhD 


| Sugo | rested | follow | up ( | questions: |
|------|--------|--------|------|------------|

- Tell me what that was like. Can you give me some examples?
- How bad has this been since this time yesterday?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this since this time yesterday?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

# Since this time yesterday, how much have you felt tense, keyed up, or on edge?

### Have you gotten tired easily?

How much have you been bothered by any of these things:

- · being startled easily?
- crying easily?
- trembling?
- feeling restless?
- not being able to relax?

# 2. TENSION

(feelings of tension, fatigability, startle response, moved to tears easily, trembling, feelings of restlessness, inability to relax):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

# Since this time yesterday, have you been afraid of . . .

- the dark?
- · of strangers?
- of being left alone?
- of animals?
- of traffic?
- of crowds?

Have you had any other specific fears since this time yesterday?

# 3. FEARS

(of dark, of strangers, of being left alone, of animals, of traffic, of crowds):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

# NOTE: INCLUDE ANY IRRATIONAL ANXIETY ABOUT

© SIGH-A 2013, v1.2 – 24 HR Version. Janet B.W. Williams, PhD  

- Tell me what that was like. Can you give me some examples?
- How bad has this been since this time yesterday?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this since this time yesterday?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

| ATION: |
|--------|

## Now let's talk about your sleep.

Since this time yesterday, have you had trouble falling asleep?

How long has it taken you to fall asleep? IF MORE THAN 30 MINUTES: How many times since this time yesterday did this happen?

Since this time yesterday, did you wake up in the middle of your sleep time? IF YES: How long were you awake? How often did this happen?

IF UNKNOWN: Since this time yesterday, has your sleep been restless or disturbed? IF YES: For how much of your sleep time has this been the case?

Did you feel tired when you woke up because you felt you didn't have a good sleep?

How about having bad dreams or nightmares?

## 4. INSOMNIA

(difficulty in falling asleep, broken sleep, unsatisfying sleep and fatigue on waking, dreams, nightmares, night terrors):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe


- Tell me what that was like. Can you give me some examples?
- How bad has this been since this time yesterday?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this since this time yesterday?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

| Since this time yesterday have you had trouble concentrating? | 5. INTELLECTUAL (difficulty in concentrating, poor memory): |
|---|---|
| IF YES: Can you give me some examples? | 0 - not present |
| | 1 - mild |
| However the state of the state | 2 - moderate |
| How about trouble reading – like a book or a newspaper? Do you need to read things over and over again? | 3 - severe |
| , | 4 - very severe |
| Have you had any trouble following a conversation? | |
| Have you had trouble remembering things since this | |
| time yesterday? | 3 |
| IF UNKNOWN: What about remembering appointments or errands you have to do? | |


- Tell me what that was like. Can you give me some examples?
- How bad has this been since this time yesterday?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this since this time yesterday?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

Since this time yesterday, have you felt sad, depressed, or down?

Can you describe the feeling? How bad has it been?

IF YES: Does the feeling lift if something good happens?

How have you been feeling about the future, since this time yesterday?

Have you been feeling discouraged or pessimistic?

What have your thoughts been?

Have you been crying since this time yesterday?

Have you been less interested in things, or not enjoying things you usually enjoy doing?

Have you awakened earlier than usual, when you have slept since this time yesterday? (Is that with an alarm clock, or did you just wake up yourself?)

Since this time yesterday, have you been feeling better or worse at any particular time of day - morning or evening? IF VARIATION: How much worse?

## 6. DEPRESSED MOOD

(loss of interest, lack of pleasure in hobbies depression, early waking, diurnal swing):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe


| Suggest | ted fo | ollow | up q | uestic | ons: |
|---------|--------|-------|------|--------|------|

- Tell me what that was like. Can you give me some examples?
- How bad has this been since this time yesterday?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this since this time yesterday?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

## Since this time yesterday, have you had any ...

- muscle aches or pains?
- muscle twitching?
- tight or stiff muscles?
- sudden muscle jerks?
- grinding of your teeth?
- an unsteady voice?

# 7. SOMATIC (MUSCULAR)

(pains and aches, twitching, stiffness, myoclonic jerks, grinding of teeth, unsteady voice, increased muscular tone):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

# Since this time yesterday, have you had ...

- · ringing in your ears?
- blurred vision?
- hot or cold flashes?
- feelings of physical weakness (not just feeling tired)?
- How about pricking sensations?

# 8. SOMATIC (SENSORY)

(tinnitus, blurring of vision, hot and cold flushes, feelings of weakness, pricking sensation):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe


- Tell me what that was like. Can you give me some examples?
- How bad has this been since this time yesterday?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this since this time yesterday?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

# Since this time yesterday, has . . .

- · your heart raced, skipped or pounded?
- · Have you had pain in your chest?
- · Had any throbbing blood vessels?
- Any fainting feelings?

# 9. CARDIOVASCULAR SYMPTOMS

(tachycardia, palpitations, pain in chest, throbbing vessels, fainting feelings):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

# Since this time yesterday, have you had . . .

- · pressure or tightness in your chest?
- choking feelings?
- · What about sighing?
- · Have you had shortness of breath?

# 10. RESPIRATORY SYMPTOMS

(pressure or constriction in chest, choking feelings, sighing, dyspnea):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe


- Tell me what that was like. Can you give me some examples?
- How bad has this been since this time yesterday?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this since this time yesterday?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

## Since this time yesterday, have you had ...

- · trouble swallowing?
- · stomach pain or fullness?
- gas?
- nausea?
- vomiting?
- · burning or rumbling in your stomach?
- loose bowels?
- constipation?
- Have you lost weight since this time yesterday? IF YES: How much? (Have you been trying to lose weight?) DO NOT RATE LOSS OF WEIGHT DUE TO DIETING.

# 11. GASTROINTESTINAL SYMPTOMS

(difficulty in swallowing, wind, abdominal pain, burning sensations, abdominal fullness, nausea, vomiting, borborygmi, looseness of bowels, loss of weight, constipation):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe


- Tell me what that was like. Can you give me some examples?
- How bad has this been since this time yesterday?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this since this time yesterday?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

Since this time yesterday, have you had to urinate frequently? IF NO: Have you had the urge to?

How has your interest in sex been since this time yesterday? I'm not asking about performance, but about your interest in sex.

Is this a change for you? IF YES: How much of a change?

FOR WOMEN: When some women feel nervous or anxious, they have trouble having an orgasm, although they have had them in the past. Have you had difficulty with orgasm since this time yesterday?
IF YES: How much trouble have you had?

Have you had your period in the last month or so? IF YES: Has it been especially heavy? IF NOT: Do you know why not?

FOR MEN: Sometimes when men feel nervous or anxious, they have trouble with premature ejaculation, or they have trouble keeping an erection. Has that happened to you since this time yesterday? IF YES: How much trouble have you had?

## 12. GENITOURINARY SYMPTOMS

(frequency of micturition, urgency of micturition, amenorrhea, menorrhagia, development of frigidity, premature ejaculation, loss of libido, impotence):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe

© SIGH-A 2013, v1.2 - 24 HR Version. Janet B.W. Williams, PhD  

- Tell me what that was like. Can you give me some examples?
- How bad has this been since this time yesterday?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this since this time yesterday?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

Since this time yesterday, has your mouth been dry?

Have you had any flushing in your face?

Have you been pale?

Have you felt lightheaded?

Have you had headaches?

How about feeling the hair rise on your arms, the back of your neck, or your head?

Have you tended to sweat a lot since this time yesterday?

## 13. AUTONOMIC SYMPTOMS

(dry mouth, flushing, pallor, tendency to sweat, giddiness, tension headache, raising of hair):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe


108
- Tell me what that was like. Can you give me some examples?
- How bad has this been since this time yesterday?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this since this time yesterday?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

RATING BASED ON OBSERVATION DURING INTERVIEW (CIRCLE SYMPTOMS PRESENT).

#### FOR TELEPHONE ASSESSMENT:

During this interview, have you been fidgeting at all, or having trouble sitting still? Have you been doing anything like playing with your hands or hair, or tapping your foot?

IF YES: How bad has that been?

Have your hands been shaky?

What about swallowing or feeling the need to swallow?

If you looked in a mirror right now, would your face look relaxed? IF NO: Would it look strained or tight?

Do you think you look pale?

#### 14. BEHAVIOR AT INTERVIEW

(fidgeting, restlessness or pacing, tremor of hands, furrowed brow, strained face, sighing or rapid respiration, facial pallor, swallowing, belching, brisk tendon jerks, dilated pupils, exophthalmos, etc.):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

| TIME ENDED SIGH-A: | <br>AM / PM | ET / CT / PT |
|--------------------|-------------|--------------|
| TOTAL HAM-A SCORE: | | |


#### STRUCTURED INTERVIEW GUIDE FOR THE HAMILTON ANXIETY SCALE (SIGH-A)

Janet B.W. Williams, PhD

INTERVIEWER: The questions for each item that appear in bold type should be asked exactly as written. Follow-up questions are provided for further exploration of symptoms. For each symptom endorsed, use the additional probes at the top of each page to determine the frequency and severity of the symptom, including how bad it's been, how much distress it has caused, and if the symptom has caused any impairment. These questions should be asked until you have enough information to rate the item confidently. You may also have to add your own follow-up questions to obtain necessary information. For some of the HAM-A items, you may find you have already asked about some of the symptoms (for a previous item). You do not need to repeat questions about these symptoms unless you need additional information to rate their severity.

All of the items have the same anchor points. The following may be useful as a guide to rating item severity:

ABSENT Score 0 if symptoms are absent, insignificant, or clearly

due to causes other than anxiety

MILD Score 1 if symptom is infrequent, with no impairment and

no more than mild distress

MODERATE Score 2 if symptom is more frequent, with moderate

distress or limited interference with usual activities

SEVERE Score 3 if symptom is severe and persistent or results in severe distress or marked impairment in functioning

severe distress of marked impairment in function

VERY SEVERE Score 4 if symptom is incapacitating

For each symptom, ask:

- Tell me what that was like. Can you give me some examples?
- How bad has this been over the past week?
- . How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this over the past week?

#### NOTES

<u>Time period</u>. The ratings should be based on the patient's condition during the past week. Unlike the HAMD, change from usual self is not required for most items to be rated positively on the HAMA. However, symptoms should not be rated positively if they are clearly due to a cause unrelated to anxiety, e.g., respiratory symptoms due to pneumonia.

<u>Panic attacks</u>. If the patient has panic attacks, this could affect the ratings of many of the symptoms. It is recommended that you consider the total amount of time during the past week that the panic attack symptoms occurred, as well as their severity. For example, a patient who has a few severe but short-lived panic attacks during the week, but who otherwise does not have many anxiety symptoms, would probably not have a very high total HAM-A score.

This instrument provides an interview guide for the Hamilton Anxiety Scale (Hamilton M: The assessment of anxiety states by rating. Brit J Med Psychol 32:50-55, 1959; Hamilton M: The disgnosis and rating of anxiety, in Studies of Anxiety, MH Lader, Ed., Headley Bros., Kent, 1969). The anchor point descriptions for the scale have been taken from the ECDEU Assessment Manual (Guy, William, ECDEU Assessment Manual for Psychopharmacology, Revised 1976, DHEW Publication No. (ADM) 76-338), except that "sighing" and "dyspnea," which appear twice in that version, have been taken out of the item "cardiovascular symptoms," and left under "respiratory symptoms." Kenneth A. Kobak, PhD and Joshua D. Lipsitz, PhD contributed to revisions of this interview guide. Dr. Williams' degree was changed to PhD; no other changes have been made to the interview guide since the date of this revision.

For further information and permission to use or translate the SIGH-A, contact Dr. Williams at <a href="mailto:ibwwny@gmail.com">ibwwny@gmail.com</a>.

2008 © Janet B. W. Williams, PhD Revision 15Jan08 

| TIME BEGAN SIGH-A: AM / PM ET / CT DATE: / / st week. How have you been feeling since last u been working? IF NOT: Why not? Score 0 if symptoms are absent, |
|---|
| st week. How have you been feeling since last u been working? IF NOT: Why not? Score 0 if symptoms are absent, |
| u been working? IF NOT: Why not? Score 0 if symptoms are absent, |
| ABSENT insignificant, or clearly due to causes other<br>than anxiety |
| MILD Symptom is infrequent, with no impairment and no more than mild distress |
| Symptom is more frequent, with moderate distress or limited interference with usual |
| activities Score 3 if symptom is severe and persister SEVERE or results in severe distress or marked |
| impairment in functioning SEVERE Symptom is incapacitating |
| 1. ANXIOUS MOOD (worries, anticipation of the worst, fearful anticipation, irritability): 0 - not present 1 - mild 2 - moderate 3 - severe |
| 4 - very severe |
| lave you been feeling this way? |

| Suggest | ted | follow | up | quest | ions: |
|---------|-----|--------|----|-------|-------|

- Tell me what that was like. Can you give me some examples?
- How bad has this been over the past week?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this over the past week?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

#### In the past week, how much have you felt tense, keyed up, or on edge?

Have you gotten tired easily?

How much have you been bothered by any of these things:

- · being startled easily?
- crying easily?
- trembling?
- feeling restless?
- not being able to relax?

#### 2. TENSION

(feelings of tension, fatigability, startle response, moved to tears easily, trembling, feelings of restlessness, inability to relax):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

#### This past week, have you been afraid of . . .

- the dark?
- · of strangers?
- of being left alone?
- of animals?
- of traffic?
- · of crowds?

Have you had any other specific fears this past week?

NOTE: INCLUDE ANY IRRATIONAL ANXIETY ABOUT OBJECTS OR SITUATIONS.

#### 3. FEARS

(of dark, of strangers, of being left alone, of animals, of traffic, of crowds):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

2008 © Janet B. W. Williams, PhD Revision 15Jan08 

- Tell me what that was like. Can you give me some examples?
- How bad has this been over the past week?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this over the past week?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

#### Now let's talk about your sleep.

In the last week, have you had trouble falling asleep?

How long has it been taking you to fall asleep? IF MORE THAN 30 MINUTES: How many nights this past week did this happen?

In the past week have you been waking up in the middle of the night? IF YES: How long are you awake? How many nights this past week did this happen?

IF UNKNOWN: In the past week, has your sleep been restless or disturbed? IF YES: How many nights this past

Have you felt tired when you woke up because you felt you didn't get a good night's sleep? IF YES: How many times?

How about having bad dreams or nightmares?

#### 4. INSOMNIA

(difficulty in falling asleep, broken sleep, unsatisfying sleep and fatigue on waking, dreams, nightmares, night terrors):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

2008 © Janet B. W. Williams, PhD Revision 15Jan08 

- Tell me what that was like. Can you give me some examples?
- How bad has this been over the past week?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this over the past week?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate<br>distress or limited interference with usual<br>activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

| n the last week, have you had trouble | 5. INTELLECTUAL |
|---|---|
| oncentrating? | (difficulty in concentrating, poor memory): |
| F YES: Can you give me some examples? | 0 - not present |
| | 1 - mild |
| | 2 - moderate |
| How about trouble reading – like a book or a newspaper? Do you need to read things over and over again? | 3 - severe |
| Do you need to read things over and over again: | 4 - very severe |
| Have you had any trouble following a conversation? | |
| Have you had trouble remembering things this past week? | |
| week? | |
| * ( | |
| IF UNKNOWN: What about remembering appointments | <b> </b> |
| or errands you have to do? | |

2008 © Janet B. W. Williams, PhD Revision 15Jan08 

- Tell me what that was like. Can you give me some examples?
- How bad has this been over the past week?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this over the past week?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

In the past week, have you felt sad, depressed, or down?

Can you describe the feeling? How bad has it been?

IF YES: Does the feeling lift if something good happens?

How have you been feeling about the future?

Have you been feeling discouraged or pessimistic? .

What have your thoughts been?

Have you been crying this past week?

Have you been less interested in things, or not enjoying things you usually enjoy doing?

Have there been times this past week when you have awakened earlier than usual? (Is that with an alarm clock, or did you just wake up yourself?)

IF EARLY WAKING: How many times?

This past week, have you been feeling better or worse at any particular time of day - morning or evening? IF VARIATION: How much worse? How many days has this been the pattern?

#### 6. DEPRESSED MOOD

(loss of interest, lack of pleasure in hobbies, depression, early waking, diurnal swing):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

2008 © Janet B. W. Williams, PhD Revision 15Jan08 

- Tell me what that was like. Can you give me some examples?
- How bad has this been over the past week?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this over the past week?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

#### In the last week, have you had any ...

- · muscle aches or pains?
- · muscle twitching?
- · tight or stiff muscles?
- sudden muscle jerks?
- · grinding of your teeth?
- · Having an unsteady voice?

#### 7. SOMATIC (MUSCULAR)

(pains and aches, twitching, stiffness, myoclonic jerks, grinding of teeth, unsteady voice, increased muscular tone):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

#### In the past week, have you had ...

- · ringing in your ears?
- · blurred vision?
- · hot or cold flashes?
- feelings of physical weakness (not just feeling tired)?
- How about pricking sensations?

#### 8. SOMATIC (SENSORY)

(tinnitus, blurring of vision, hot and cold flushes, feelings of weakness, pricking sensation):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

2008 © Janet B. W. Williams, PhD Revision 15Jan08 

- Tell me what that was like. Can you give me some examples?
- How bad has this been over the past week?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this over the past week?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

#### In the past week, has . . .

- · your heart raced, skipped or pounded?
- · Have you had pain in your chest?
- · Had any throbbing blood vessels?
- · Any fainting feelings?

#### 9. CARDIOVASCULAR SYMPTOMS

(tachycardia, palpitations, pain in chest, throbbing vessels, fainting feelings):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

#### In the last week, have you had . . .

- · pressure or tightness in your chest?
- choking feelings?
- What about sighing?
- · Have you had shortness of breath?

#### 10. RESPIRATORY SYMPTOMS

(pressure or constriction in chest, choking feelings, sighing, dyspnea):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

2008 © Janet B. W. Williams, PhD Revision 15Jan08 

- Tell me what that was like. Can you give me some examples?
- How bad has this been over the past week?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this over the past week?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

#### In the last week, have you had ...

- · trouble swallowing?
- · stomach pain or fullness?
- gas?
- nausea?
- vomiting?
- · burning or rumbling in your stomach?
- loose bowels?
- constipation?
- Have you lost weight in the past week? IF YES: How much? (Have you been trying to lose weight?) DO NOT RATE LOSS OF WEIGHT DUE TO DIETING.

#### 11. GASTROINTESTINAL SYMPTOMS

(difficulty in swallowing, wind, abdominal pain, burning sensations, abdominal fullness, nausea, vomiting, borborygmi, looseness of bowels, loss of weight, constipation):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

2008 © Janet B. W. Williams, PhD Revision 15Jan08 

- Tell me what that was like. Can you give me some examples?
- How bad has this been over the past week?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this over the past week?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

In the past week, have you had to urinate frequently? IF NO: Have you had the urge to?

How has your interest in sex been this past week? I'm not asking about performance, but about your interest in sex.

Is this a change for you? IF YES: How much of a change?

FOR WOMEN: When some women feel nervous or anxious, they have trouble having an orgasm, although they have had them in the past. Have you had difficulty with orgasm in the past week?

IF YES: How much trouble have you had?

Have you had your period in the last month or so?
IF YES: Has it been especially heavy?
IF NOT: Do you know why not?

FOR MEN: Sometimes when men feel nervous or anxious, they have trouble with premature ejaculation, or they have trouble keeping an erection. Has that happened to you in the past week? IF YES: How much trouble have you had?

#### 12. GENITOURINARY SYMPTOMS

(frequency of micturition, urgency of micturition, amenorrhea, menorrhagia, development of frigidity, premature ejaculation, loss of libido, impotence):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

2008 © Janet B. W. Williams, PhD Revision 15Jan08 

- Tell me what that was like. Can you give me some examples?
- How bad has this been over the past week?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this over the past week?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

In the past week, has your mouth been dry?

Have you had any flushing in your face?

Have you been pale?

Have you felt lightheaded?

Have you had headaches?

How about feeling the hair rise on your arms, the back of your neck, or your head?

Have you tended to sweat a lot in the past week?

#### 13. AUTONOMIC SYMPTOMS

(dry mouth, flushing, pallor, tendency to sweat, giddiness, tension headache, raising of hair):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

2008 © Janet B. W. Williams, PhD Revision 15Jan08 

| Suggested | follow | LID A | au oci | tione |
|-----------|--------|-------|--------|-------|

- Tell me what that was like. Can you give me some examples?
- How bad has this been over the past week?
- How much has it bothered you? Has it caused you any problems?
- How much of the time or how often have you had this over the past week?

| ABSENT | Score 0 if symptoms are absent, insignificant, or clearly due to causes other than anxiety |
|---|---|
| MILD | Symptom is infrequent, with no impairment and no more than mild distress |
| MODERATE | Symptom is more frequent, with moderate distress or limited interference with usual activities |
| SEVERE | Score 3 if symptom is severe and persistent<br>or results in severe distress or marked<br>impairment in functioning |
| VERY SEVERE | Symptom is incapacitating |

#### RATING BASED ON OBSERVATION DURING INTERVIEW (CIRCLE SYMPTOMS PRESENT):

#### FOR TELEPHONE ASSESSMENT:

During this interview, have you been fidgeting at all, or having trouble sitting still? Have you been doing anything like playing with your hands or hair, or tapping your foot?

IF YES: How bad has that been?

Have your hands been shaky?

What about swallowing or feeling the need to swallow?

If you looked in a mirror right now, would your face look relaxed? IF NO: Would it look strained or tight?

Do you think you look pale?

#### 14. BEHAVIOR AT INTERVIEW

(fidgeting, restlessness or pacing, tremor of hands, furrowed brow, strained face, sighing or rapid respiration, facial pallor, swallowing, belching, brisk tendon jerks, dilated pupils, exophthalmos, etc.):

- 0 not present
- 1 mild
- 2 moderate
- 3 severe
- 4 very severe

TIME ENDED SIGH-A: \_\_\_\_\_ AM / PM ET / CT / PT

TOTAL HAM-A SCORE: \_\_\_\_\_

2008 © Janet B. W. Williams, PhD Revision 15Jan08 

## APPENDIX 4. CLINICAL GLOBAL IMPRESSION–IMPROVEMENT SCALE (CGI-I) AND SEVERITY SCALE (CGI-S)

#### Clinical Global Impression - Improvement (CGI-I) Scale

Rate total improvement whether or not in your judgment it is due entirely to drug treatment. Compared to his/her condition at baseline, how much has patient changed? (Note that subject's illness is the disease under study; in this case, Major Depressive Disorder – NOT other conditions/co-morbidities.)

| 1 | Very much improved | Nearly all better; good level of functioning; minimal symptoms; represents a very substantial change |
|---|---|---|
| 2 | Much<br>improved | Notably better with significant reduction of symptoms; increase in the level of functioning but some symptoms remain |
| 3 | Minimally<br>improved | Slightly better with little or no clinically meaningful reduction of symptoms. Represents very little change in basic clinical status, level of care, or functional capacity |
| 4 | No change | Symptoms remain essentially unchanged |
| 5 | Minimally<br>worse | Slightly worse but may not be clinically meaningful, may represent very little change in basic clinical status or functional capacity |
| 6 | Much worse | Clinically significant increase in symptoms and diminished functioning |
| 7 | Very much<br>worse | Severe exacerbation of symptoms and loss of functioning |

| Rater Signature: | Date (DD/MMM/YYYY): |
|------------------|---------------------|

Busner, J., Targum, S. (2007), as adapted from Spearing, et al. Psychiatry Research, 1997. 73:159-171.

Modified from Guy W. Clinical Global Impressions: In ECDEU Assessment Manual for Psychopharmacology. 1976; 218-222. Revised DHEW Pub. (ADM) Rockville, MD: National Institute for Mental Health

Page 1 of 1

#### Clinical Global Impression - Severity of Illness (CGI-S) Scale

Considering your total clinical experience with this particular population, how mentally ill is the patient at this time? (Note that subject's illness is the disease under study; in this case, Major Depressive Disorder – NOT other conditions/co-morbidities.)

| 1 | Normal, not at all ill | Symptoms of disorder not present during the timeframe |
|---|---|---|
| 2 | Borderline ill | Subtle or suspected pathology |
| 3 | Mildly ill | Clearly established symptoms with minimal, if any, distress or difficulty in social and occupational function |
| 4 | Moderately ill | Overt symptoms causing noticeable, but modest, functional impairment or distress; symptom level may warrant medication |
| 5 | Markedly ill | Intrusive symptoms that distinctly impair social/occupational function or cause intrusive levels of distress |
| 6 | Severely ill | Disruptive pathology; behavior and function are frequently influenced by symptoms; may require assistance from others |
| 7 | Among the most extremely ill patients | Pathology drastically interferes in many life functions; may be hospitalized |

| Rater Signature: | Date (DD/MMM/YYYY): |
|------------------|---------------------|

Busner, J., Targum, S. (2007), as adapted from Kay, Stanley R., Positive and Negative Symptoms in Schizophrenia:Assessment and Research. Clinical and Experimental Psychiatry, Monograph No. 5. Brunner/Mazel, 1991.

Modified from Guy W. Clinical Global Impressions: In ECDEU Assessment Manual for Psychopharmacology. 1976; 218-222. Revised DHEW Pub. (ADM) Rockville, MD: National Institute for Mental Health

Page 1 of 1

#### **APPENDIX 5. SHORT-FORM 36 (SF-36)**

#### SF-36 QUESTIONNAIRE

| Name: | Ref. Dr: | | Date: | |
|---|---|---|---|---|
| D#: Gender: M / F | | | | |
| Please answer the 36 questions of | the Health Survey com | pletely, honestly, | and without intern | uptions. |
| GENERAL HEALTH: | | | | |
| In general, would you say your I | nealth is: | _ | _ | |
| C Excellent CV | ery Good | Good | OFair | Poor |
| Compared to one year ago, how Much better now than one year | | ealth in general | now? | |
| Somewhat better now than one | vear ago | | | |
| CAbout the same | ,5- | | | |
| Somewhat worse now than one | year ago | | | |
| OMuch worse than one year ago | | | | |
| LIMITATIONS OF ACTIVITIES:<br>The following items are about activities? If so, how much? | ties you might do during | a typical day. Do | es your health now | v limit you in the |
| Vigorous activities, such as runn | ing, lifting heavy object | ts, participating | in strenuous spo | rts. |
| CYes, Limited a lot | Yes, Limited a Little | | ONo, Not Limited | at all |
| Moderate activities, such as movi | ing a table, pushing a v | acuum cleaner, | bowling, or playi | ng golf |
| CYes, Limited a Lot | Yes, Limited a Little | | ONo, Not Limited | |
| Lifting or carrying groceries | | | | |
| CYes, Limited a Lot | Yes, Limited a Little | | ONo, Not Limited | at all |
| Climbing several flights of stairs | | | | |
| Yes, Limited a Lot | Yes, Limited a Little | | No, Not Limited | at all |
| Climbing one flight of stairs | | | | |
| Yes, Limited a Lot | Yes, Limited a Little | | ONo, Not Limited | at all |
| Bending, kneeling, or stooping | | | | |
| CYes, Limited a Lot | Yes, Limited a Little | | CNo, Not Limited | at all |
| Walking more than a mile | | | 0 | |
| CYes, Limited a Lot | Yes, Limited a Little | | CNo, Not Limited | at all |
| Walking several blocks | | | | |
| CYes, Limited a Lot | OYes, Limited a Little | | CNo, Not Limited | at all |
| Walking one block | | | 0 | |
| Yes, Limited a Lot | Yes, Limited a Little | | No, Not Limited | at all |

| 0.0000000 | 50 VIII | | | |
|---|---|---|---|---|
| Bathing or dress | | | 0 | |
| CYes, Limited | a Lot | Yes, Limited a Little | CNo, No | t Limited at all |
| | | any of the following probl | lems with your work or | other regular daily activities as |
| Cut down the ar | mount of time you sp | ent on work or other act | ivities | |
| CYes | CNo | | | |
| Accomplished I | ess than you would li | ike | | |
| CYes | CNo | | | |
| 141 | 0 - 1: - 1 - f 1 | | | |
| CYes | the kind of work or o | ther activities | | |
| Cics | CINO | | | |
| | | other activities (for exa | mple, it took extra ef | ffort) |
| CYes | CNo | | | |
| a result of any e | motional problems (suc | any of the following prob<br>th as feeling depressed or<br>ent on work or other act | anxious)? | other regular daily activities as |
| A | | de- | | |
| CYes | ess than you would li | Ke | | |
| 0100 | Cito | | | |
| Didn't do work o<br>⊖Yes | or other activities as | carefully as usual | | |
| SOCIAL ACTIVI<br>Emotional probl | Control to the Control of the Contro | our normal social activi | ities with family, frien | nds, neighbors, or groups? |
| CNot at all | Cslightly | OModerately | OSevere | CVery Severe |
| PAIN:<br>How much bodi | ly pain have you had | during the past 4 week | s? | |
| CNone ( | Very Mild | Mild CModerate | OSevere | OVery Severe |
| During the past<br>home and hous | | did pain interfere with y | our normal work (inc | luding both work outside the |
| CNot at all | OA little bit | OModerately ( | Cquite a bit | Extremely |

CA good Bit of the Time
Some of the time
CA little bit of the time
None of the Time

#### ENERGY AND EMOTIONS: These questions are about how you feel and how things have been with you during the last 4 weeks. For each question, please give the answer that comes closest to the way you have been feeling. Did you feel full of pep? All of the time Most of the time CA good Bit of the Time Some of the time CA little bit of the time None of the Time Have you been a very nervous person? CAll of the time Most of the time CA good Bit of the Time Some of the time CA little bit of the time ONone of the Time Have you felt so down in the dumps that nothing could cheer you up? CAll of the time Most of the time CA good Bit of the Time Some of the time A little bit of the time None of the Time Have you felt calm and peaceful? CAll of the time Most of the time CA good Bit of the Time Some of the time A little bit of the time None of the Time Did you have a lot of energy? CAll of the time Most of the time

| Have you felt downhearted and blue? |
|---|
| CAll of the time CMost of the time |
| CA good Bit of the Time CSome of the time |
| CA little bit of the time |
| CNone of the Time |
| Did you feel worn out? |
| CAll of the time |
| CMost of the time |
| CA good Bit of the Time |
| Csome of the time |
| CA little bit of the time |
| CNone of the Time |
| Have you been a happy person? |
| CAll of the time |
| CMost of the time |
| CA good Bit of the Time |
| Some of the time |
| CA little bit of the time |
| CNone of the Time |
| Did you feel tired? |
| CAll of the time |
| CMost of the time |
| CA good Bit of the Time |
| CSome of the time |
| CA little bit of the time |
| CNone of the Time |
| COCIAL ACTIVITIES |
| SOCIAL ACTIVITIES: During the past 4 weeks, how much of the time has your physical health or emotional problems interfered with |
| your social activities (like visiting with friends, relatives, etc.)? |
| CAll of the time |
| CMost of the time |
| Some of the time |
| CA little bit of the time |
| None of the Time |

#### Sage Therapeutics

| How true or false is ea | ch of the following | g statements for you | ? | |
|---|---|---|---|---|
| I seem to get sick a litt<br>Opefinitely true | tle easier than oth | er people<br>CDon't know | OMostly false | Opefinitely false |
| I am as healthy as anylopefinitely true | body I know<br>Mostly true | CDon't know | OMostly false | Opefinitely false |
| I expect my health to g | et worse<br>Mostly true | Opon't know | Mostly false | Opefinitely false |
| My health is excellent<br>Definitely true | Mostly true | CDon't know | OMostly false | Opefinitely false |

### APPENDIX 6. THE FATIGUE ASSOCIATED WITH DEPRESSION (FAs-D) PATIENT-REPORTED OUTCOME (PRO)

Some people experience fatigue when they are depressed. The following items ask you to rate fatigue you have experienced that you think may be related to depression.

| In the PAST WEEK, how often have you felt | Never | Rarely | Sometimes | Often | Always |
|---|---|---|---|---|---|
| 1. Fatigued | 1 | 2 | 3 | 4 | 5 |
| 2. Tired | 1 | 2 | 3 | 4 | 5 |
| 3. Exhausted | 1 | 2 | 3 | 4 | 5 |
| 4. Like you had no energy | 1 | 2 | 3 | 4 | 5 |
| 5. Physically weak | 1 | 2 | 3 | 4 | 5 |
| 6. Slowed down | 1 | 2 | 3 | 4 | 5 |
| 7. Like everything requires too much effort | 1 | 2 | 3 | 4 | 5 |

Now think about the impact of this fatigue that is related to depression. The following items ask about the impact of this fatigue on various aspects of your life.

| In the PAST WEEK, how much has your fatigue | Not at all | A little | Somewhat | Quite a bit | Very much |
|---|---|---|---|---|---|
| Limited your ability to complete daily household chores | 1 | 2 | 3 | 4 | 5 |
| <ol> <li>Interfered with family activities or relationships</li> </ol> | 1 | 2 | 3 | 4 | 5 |
| 10. Interfered with doing things you enjoy | 1 | 2 | 3 | 4 | 5 |
| 11. Interfered with social activities, like spending time with friends | 1 | 2 | 3 | 4 | 5 |
| 12. Interfered with taking care of yourself (e.g., bathing, dressing, brushing your teeth) | 1 | 2 | 3 | 4 | 5 |
| 13. Kept you from getting out of bed | 1 | 2 | 3 | 4 | 5 |

| Do you have a spouse or significant other? | $\Box$ Y | es 🗆 | No | | |
|---|---|---|---|---|---|
| If no, leave item 14 blank. | | | | | |
| If yes, please answer item 14. | | | | | |
| In the PAST WEEK, how much has your fatigue | Not at all | A little | Somewhat | Quite a bit | Very muci |
| 14. Interfered with your intimate relationship (i.e., with a spouse or significant other) | 1 | 2 | 3 | 4 | 5 |

**Do you have a job or go to school?**  $\Box$  Yes

If no, leave items 15 and 16 blank.

If yes, please answer items 15 and 16.

| In the past week, how much has your fatigue | Not at all | A little | Somewhat | Quite a bit | Very much |
|---|---|---|---|---|---|
| 15. Prevented you from going to work or school | 1 | 2 | 3 | 4 | 5 |
| Limited your productivity at work or school | 1 | 2 | 3 | 4 | 5 |

 $\square$  No

## APPENDIX 7. COLUMBIA - SUICIDE SEVERITY RATING SCALE (C-SSRS)

COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

#### Baseline/Screening Version

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <u>The Columbia Suicide</u> <u>History Form</u>, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103 -130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

© 2008 The Research Foundation for Mental Hygiene, Inc.

C-SSRS Baseline Screening - United States/English - Mapi. C-SSRS-BaselineScreening\_AU5.1\_eng-USorl.doc

| | Lifetime: Time<br>He/She Felt<br>Most Suicidal | | Past 24<br>Months | |
|---|---|---|---|---|
| ih to fall asleep and not wake up.<br>s up? | Yes | No | Yes | No |
| | _ | _ | | |
| ., "I've thought about killing myself") without thoughts of period. | Yes | No | Yes | No |
| out Intent to Act ring the assessment period. This is different than a specific kill self but not a specific plan). Includes person who would owhen, where or how I would actually do it and I would | Yes | No. | Yes | No |
| pecific Plan ent to act on such thoughts, as opposed to "I have the thoughts | Yes | No | Yes | No |
| d subject has some intent to carry it out.<br>? Do you intend to carry out this plan? | Yes | No | Yes | No |
| • . ( ) | _ | _ | _ | _ |
| as feeling the most suicidal. Description of Ideation Description of Ideation | Most | : Severe | Mo:<br>Seve | |
| k (4) Daily or almost daily (5) Many times each day | _ | | _ | |
| (4) 4-8 hours/most of day<br>(5) More than 8 hours/persistent or continuous | - | _ | _ | - |
| die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts | - | _ | | - |
| a of death) - that stopped you from wanting to die or (4) Deterrents most likely did not stop you (5) Deterrents definitely did not stop you (0) Does not apply | - | _ | _ | - |
| die or killing yourself? Was it to end the pain or living with this pain or how you were feeling) or h? (4) Mostly to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (5) Completely to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (0) Does not apply | - | _ | _ | - |
| | pecific Plan int to act on such thoughts, as opposed to "I have the thoughts in to act on such thoughts, as opposed to "I have the thoughts in the act on such thoughts, as opposed to "I have the thoughts in to act on such thoughts, as opposed to "I have the thoughts in to act on such thoughts, as opposed to "I have the thoughts in to act on such thoughts, as opposed to "I have the thoughts in to act on such thoughts, as opposed to "I have the thoughts in to act on such thoughts, as opposed to "I have the thoughts in the act on such thoughts, as opposed to "I have the thoughts in the subject has some intent to carry it out. I be subject has some intent to act out. I be sub | without thought about killing myself") without thoughts of seriod. Complete the seriod of the ser | "Twe thought about killing myself") without thoughts of period. Dut Intent to Act ring the assessment period. This is different than a specific kill self but not a specific plan). Includes person who would when, where or how I would actually do II and I would when I would actually as period of I would be seen to act on such thoughts, as opposed to "I have the thoughts." Type of ideation (i.e., I-5 from above, with I being act feeling the most suicidal. Description of Ideation Description of Ideation Whost Severe (4) Daily or almost daily (5) Many times each day (4) 4-8 hours most of day (5) More than 8 hours persistent or continuous die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (6) Does not attempt to control thoughts (7) Deservents definitely did not stop you (8) Deterrents most likely did not stop you (9) Dees not apply die or killing yourself? Was it to end the pain or living with this pain or how you were feeling) or he? (4) Mostly to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (5) Completely to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (6) Completely to end or stop the pain (you couldn't go on living with the pain or how you were feeling) | The thought about killing myself") without thoughts of Yes No Yes Period. |

| SUICIDAL BEHAVIOR<br>(Check all that apply, so long as these are separate events; must ask about all types) | | Life | time | Past<br>Mon | |
|---|---|---|---|---|---|
| Actual Attempt: | | Yes | No | Yes | No |
| A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as noneself. Intent does not have to be 100%. If there is any intenvidesire to die associated with the act, then it can be considered an attempt. There does not have to be any injury or harm, just the potential for injury or harm. If person pulls trigger who mouth but sun is broken so no injury results, this is considered an attempt. | actual suicide | | | | |
| inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumstances highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping five a high floor/story). Also, if someone denies intent to die, but they thought that what they did could be lethal, intent may be infer thave you made a suicide attempt? | m window of | | | | |
| Have you done anything to harm yourself?<br>Have you done anything dangerous where you could have died? | | | l#of | Total | |
| What did you do?<br>Did youas a way to end your life?<br>Did you want to die (even a little) when you? | A | Atte | mpts | Atten | npts |
| Were you trying to end your life when you ? Or did you think it was possible you could have died from ? Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress | faal hattar | | | | |
| of the you do I printy for other reasons? Million AN I intention of kining yourself (the to relieve stress get sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) if yes, describe: | , jeet better, | Yes | No | Yes | No |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | | ГΠ | П | | П |
| Interrupted Attempt: | | Yes | No | Yes | No |
| When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual aculd have occurred; and in the contract of the contract | an interrupted | | | | |
| attempt. Shooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pulli<br>Once they pull the trigger, even if the gun fails of fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken<br>edge. Hanging: Person has noose around neck but has not yet started to hang - is stopped from doing so.<br>Has there been a time when you started to do something to end your life but someone or something stopp | down from | Total | l#of | Total | # 05 |
| before you actually did anything?<br>If yes, describe: | eu you | | upted | intern | |
| Aborted Attempt: | | Yes | No | Yes | No |
| When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in a<br>destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being<br>something else | stopped by | | | | |
| Has there been a time when you started to do something to try to end your life but you stopped yourself b<br>actually did anything?<br>if yes, describe: | efore you | | l#of<br>rted | Total<br>abor | |
| Preparatory Acts or Behavior: | | | | | |
| Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, assembling a specific method (e.g., buying pills, purchasing a gur) or preparing for one's death by suicide (e.g., giving things a suicide note). | | Yes | No<br>□ | Yes | No |
| Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecti<br>getting a gun, giving valuables away or writing a suicide note)?<br>f yes, describe: | ng pills, | | | | |
| Suicidal Behavior: Suicidal behavior was present during the assessment period? | | Yes | No<br>□ | Yes | No |
| Answer for Actual Attempts Only | Most Recent<br>Attempt<br>Date: | Most Le<br>Attempt<br>Date: | thal | Initial/Fi<br>Attempt<br>Date: | |
| Actual Lethality Medical Damage: No physical damage or very minor physical damage (e.g., surface scratches). Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). | Enter Code | Enter | Code | Enter ( | Code |
| <ol> <li>Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact, third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures).</li> <li>Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third- degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area).</li> <li>Death</li> </ol> | | _ | _ | | _ |
| Potential Lethality: Only Answer if Actual Lethality=0<br>Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had<br>potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying<br>on train tracks with oncoming train but pulled away before run over). | Enter Code | Enter | Code | Enter ( | Code |
| ) = Behavior not likely to result in injury<br> = Behavior likely to result in injury but not likely to cause death<br>2 = Behavior likely to result in death despite available medical care | | _ | _ | | _ |
| 2008 Research Foundation for Mental Hysiene, Inc. C-SSRS—Baseline Screening (Version 1/14/09) | | | | | |

## RATING SCALE

(C-SSRS)

Since Last Visit

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <u>The Columbia Suicide</u> <u>History Form</u>, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103 -130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

C-SSRS Since Last Visit - United States/English - Mapi. C-SSRS-SinceLastMait\_AU5.1\_eng-USorl.doc



| k questions I and 2. If both are negative, proceed to "Sui- | | | |
|---|---|---|---|
| | cidal Behavior" section. If the answer to question 2 is "yes",<br>2 is "yes", complete "Intensity of Ideation" section below. | Since<br>Vi | |
| Wish to be Dead | | Yes | No |
| bject endorses thoughts about a wish to be dead or not alive anymore, or<br>we you wished you were dead or wished you could go to sleep and not t | | | |
| res, describe: | | | |
| Non-Specific Active Suicidal Thoughts | | Ī., | |
| neral non-specific thoughts of wanting to end one's life/commit suicide<br>eself/associated methods, intent, or plan during the assessment period. | (e.g., "I've thought about killing myself") without thoughts of ways to kill | Yes | No |
| ve you actually had any thoughts of killing yourself? | | | |
| res, describe: | A 4 | 7 | |
| | d during the assessment period. This is different than a specific plan with time, not a specific plan). Includes person who would say, "I thought about taking an | Yes | No |
| res, describe: | | | |
| Active Suicidal Ideation with Some Intent to Act, withou<br>tive suicidal thoughts of killing oneself and subject reports having some<br>I not do anything about them?<br>we you had these thoughts and had some intention of acting on them? | intent to act on such thoughts, as opposed to "I have the thoughts but I definitely | Yes | No |
| res, describe: | . 1 | | |
| Active Suicidal Ideation with Specific Plan and Intent | | | |
| oughts of killing oneself with details of plan fully or partially worked ou<br>we you started to work out or worked out the details of how to kill your | | Yes | No |
| res, describe: | • (7) | | |
| NTENSITY OF IDEATION | | | |
| | ere type of ideation (i.e.,1-5 from above, with 1 being the least severe | | |
| d 5 being the most severe). | \ \ | Mo | ost |
| ost Severe Ideation: | | Sev | ere |
| Type # (1-5) | Description of Ideation | | |
| equency ow many times have you had these thoughts? | | | |
| (1) Less than once a week (2) Once a week (3) 2-5 times in week | (4) Daily or almost daily (5) Many times each day | _ | _ |
| uration | | | |
| hen you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes | (4) 4-8 hours/most of day | | |
| (2) Less than 1 hour/some of the time | (5) More than 8 hours/persistent or continuous | - | _ |
| (3) 1-4 hours/a lot of time<br>ontrollability | | | |
| ould/can you stop thinking about killing yourself or wanting | | | |
| (1) Easily able to control thoughts | (4) Can control thoughts with a lot of difficulty | _ | _ |
| (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty | (5) Unable to control thoughts (0) Does not attempt to control thoughts | | |
| terrents | (-) | | |
| | pain of death) - that stopped you from wanting to die or acting on | | |
| oughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide | (4) Deterrents most likely did not stop you | | |
| (2) Deterrents probably stopped you | (5) Deterrents definitely did not stop you | _ | _ |
| (3) Uncertain that deterrents stopped you | (0) Does not apply | | |
| asons for Ideation<br>hat sort of reasons did you have for thinking about wanting | to die or killing yourself? Was it to end the pain or stop the way | | |
| | th this pain or how you were feeling) or was it to get attention, | | |
| venge or a reaction from others? Or both? | | | |
| Completely to get attention, revenge or a reaction from others Mostly to get attention, revenge or a reaction from others | (4) Mostly to end or stop the pain (you couldn't go on living with the pain or<br>how you were feeling) | _ | _ |
| (3) Equally to get attention, revenge or a reaction from others and to | (5) Completely to end or stop the pain (you couldn't go on living with the | | |
| end/stop the pain | pain or how you were feeling) | | |
| | (0) Does not apply | | |

| SUICIDAL BEHAVIOR | Since |
|---|---|
| Check all that apply, so long as these are separate events; must ask about all types) | Last Visit |
| Actual Attempt: A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as method to kill oneself. Intent lose not have to be 100%. If there is any intentidesire to die associated with the act, then it can be considered an actual suicide attempt. There does not tave to be any injury or harm, just the potential for injury or harm. If person pulls trigger while gun is in mouth but gun is broken so no injury | Yes No |
| results, this is considered an attempt. inferring Intent: Even if an individual demies intent/wish to die, it may be inferred clinically from the behavior or circumstances. For example, a highly ethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping from window of a high floor/story). | |
| Also, if someone denies intent to die, but they thought that what they did could be lethal, intent may be inferred.<br>Have you made a suicide attempt?<br>Have you done anything to harm yourself? | |
| Have you done anything dangerous where you could have died?<br>What did you do? | Total # of<br>Attempts |
| Did you as a way to end your life? Did you want to die (even a little) when you? Were you trying to end your life when you? | 4 |
| Or Did you think it was possible you could have died from? Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress, feel better, get sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) | ) |
| f yes, describe: | Yes No |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior?<br>Interrupted Attempt: | 0 0 |
| When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have occurred). Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. | Yes No |
| Shooting: Person has gum pointed toward self, gum is taken away by someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has noose around teck but has not yet started to hang - is stopped from doing so. | Total # of |
| Has there been a time when you started to do something to end your life but someone or something stopped you before you<br>actually did anything?<br>if yes, describe: | interrupted |
| News J Manuel | |
| Aborted Attempt: When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him herself, instead of being stopped by something else. Has there been a time when you started to do something to try to end your life but you stopped yourself before you actually did | Yes No Total # of |
| anything?<br>If yes, describe: | aborted |
| Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Heave you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? If yes, describe: | Yes No |
| Suicidal Behavior:<br>Suicidal behavior was present during the assessment period? | Yes No |
| Suicide: | Yes No |
| Answer for Actual Attempts Only | Most Lethal<br>Attempt<br>Date: |
| Actual Lethality/Medical Damage: Description of the property | Enter Code |
| <ol> <li>Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures).</li> <li>Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area).</li> <li>Death</li> </ol> | |
| Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: pur gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). | Enter Code |
| oe-Behavior not likely to result in injury<br>1 = Behavior likely to result in injury but not likely to cause death<br>2 = Behavior likely to result in death despite available medical care | |
| 2008 Research Foundation for Mental Hygiene, Inc. C-SSRS—Since Last Visit (Version 1/14/09) | |

#### APPENDIX 8. STANFORD SLEEPINESS SCALE (SSS)

#### Stanford Sleepiness Scale

This is a quick way to assess how alert you are feeling. If it is during the day when you go about your business, ideally you would want a rating of a one. Take into account that most people have two peak times of alertness daily, at about 9 a.m. and 9 p.m. Alertness wanes to its lowest point at around 3 p.m.; after that it begins to build again. Rate your alertness at different times during the day. If you go below a three when you should be feeling alert, this is an indication that you have a serious sleep debt and you need more sleep.

#### An Introspective Measure of Sleepiness The Stanford Sleepiness Scale (SSS)

| Degree of Sleepiness | Scale Rating |
|---|---|
| Feeling active, vital, alert, or wide awake | 1 |
| Functioning at high levels, but not at peak; able to concentrate | 2 |
| Awake, but relaxed; responsive but not fully alert | 3 |
| Somewhat foggy, let down | 4 |
| Foggy; losing interest in remaining awake; slowed down | 5 |
| Sleepy, woozy, fighting sleep; prefer to lie down | 6 |
| No longer fighting sleep, sleep onset soon; having dream-like thoughts | 7 |
| Asleep | Х |

#### 1. TITLE PAGE



#### PROTOCOL NUMBER: 217-MDD-201

# A PHASE 2, TWO-PART (OPEN-LABEL FOLLOWED BY DOUBLE-BLIND) STUDY EVALUATING THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND EFFICACY OF SAGE-217 IN THE TREATMENT OF ADULT SUBJECTS WITH MODERATE TO SEVERE MAJOR DEPRESSIVE DISORDER

**IND NUMBER: 132,131** 

Investigational Product SAGE-217

Clinical Phase 2a

Sponsor Sage Therapeutics, Inc.

Sponsor Contact , M.D., Ph.D.

Sage Therapeutics 215 First Street

Cambridge, MA 02142

Phone:

Sponsor Medical Monitor , M.D., M.B.A.

Sage Therapeutics 215 First Street

Cambridge, MA 02142

Phone:

Date of Original Protocol 24 October 2016

**Confidentiality Statement** 

The confidential information in this document is provided to you as an Investigator or consultant for review by you, your staff, and the applicable Institutional Review Board/Independent Ethics Committee. Your acceptance of this document constitutes agreement that you will not disclose the information contained herein to others without written authorization from the Sponsor.

#### PROTOCOL SIGNATURE PAGE

| Protocol Number: | 217-MDD-201 | |
|----------------------------|----------------------------|--------------------|
| Product: | SAGE-217 Oral Solution | |
| IND No.: | 132,131 | |
| Study Phase: | 2a | |
| Sponsor: | Sage Therapeutics | |
| Date of Original Protocol: | Version 1.0 24 October 201 | 6 |
| Sponsor Approval | | |
| , M.D., Ph.I | Э. | Date (DD/MMM/YYYY) |
| Sage Therapeutics | | |
| , Pharm.D, M | <u>I.</u> S., R.Ph. | Date (DD/MMM/YYYY) |
| Sage Therapeutics | | |
| , M.S.H.S. | | Date (DD/MMM/YYYY) |
| Sage Therapeutics | | |
| , Ph.D. | | Date (DD/MMM/YYYY) |
| Sage Therapeutics | | |

#### **INVESTIGATOR'S AGREEMENT**

I have received and read the Investigator's Brochure for SAGE-217. I have read the Clinical Protocol 217-MDD-201 and agree to conduct the study as outlined. I agree to maintain the confidentiality of all information received or developed in connection with this protocol.

| Printed Name of Investigator |
|------------------------------|
| Signature of Investigator |
| Date |

#### **CONTACTS IN CASE OF EMERGENCY**

**Table 1:** Emergency Contact Information

| Name | Address and Telephone Number |
|------|------------------------------|
| | Name |
## 2. SYNOPSIS

## Name of Sponsor/Company:

Sage Therapeutics

215 First Street

Cambridge, MA 02142

## **Name of Investigational Product:**

SAGE-217 Oral Solution

## Name of Active Ingredient:

**SAGE-217** 

**Title of Study:** A Phase 2, Two-Part (Open-Label Followed by Double-Blind) Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of SAGE-217 in the Treatment of Adult Subjects With Moderate to Severe Major Depressive Disorder

**Study centers:** Approximately 3 sites in Part A and approximately 15 sites in Part B

Phase of development: 2a

## Methodology:

This study will assess the safety, tolerability, pharmacokinetics (PK), and efficacy of SAGE-217 Oral Solution in adult subjects diagnosed with moderate to severe major depressive disorder (MDD).

There are two parts to the study:

Part A: Open-label dosing with SAGE-217 Oral Solution (14 days)

All subjects will receive a 30 mg SAGE-217 Oral Solution dose administered at 8:00 PM ( $\pm 15$  minutes) with food on Day 1 to Day 14 as tolerated.

**Part B**: Randomized, double-blind, parallel-group, placebo-controlled (14 days)

Based on the results of Part A, eligible subjects will be stratified based on use of antidepressant treatment (current/stable or not treated/withdrawn ≥30 days) and randomized within each stratum in a 1:1 fashion to receive SAGE-217 Oral Solution 30 mg or matching placebo for 14 days beginning on Day 1 as tolerated. All doses of study drug will be administered at 8:00 PM (±15 minutes) with food. Dose adjustments based on tolerability are detailed in Section 9.3.

Separate cohorts of subjects will be enrolled in Part A and Part B; subjects participating in Part A cannot enroll in Part B. Part B may be initiated after termination or completion of Part A if there is a clear signal of activity based on the 17-item Hamilton Rating Scale for Depression (HAM-D) scores and/or other scales being assessed.

Both parts of the study will consist of an up to 7-day Screening Period (Days -7 to -1), a 14-day Treatment Period, and a 2-week Follow-up Period. During the study Treatment Period, subjects must remain inpatient for the first 7 days at minimum and per Investigator's judgement thereafter.

Screening Period: The Screening Period begins with the signing of the informed consent form (ICF) at the Screening Visit, which can occur on any one calendar day of the 7-day window (from Day -7 through Day -1). The diagnosis of MDD must be made according to Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Axis I Disorders (SCID-I) performed by a qualified healthcare professional. Subjects will undergo preliminary screening procedures at the Screening Visit to determine eligibility, including completion of the HAM-D, Hamilton Anxiety Rating Scale (HAM-A), Clinical Global Impression - Severity (CGI-S), and Montgomery-Åsberg Depression Rating Scale (MADRS). The Screening Period assessments will be conducted on an outpatient basis. Most eligibility criteria are the same for both parts of the study.

## **Treatment Period:**

Part A – Once subjects are confirmed as eligible, they will receive a 30 mg dose of study drug at 8:00 PM ( $\pm15$  minutes) with food for 14 days (Day 1 to Day 14) as tolerated. Subjects who cannot tolerate 30 mg will receive 20 mg for the rest of the Treatment Period. Subjects who cannot tolerate 20 mg will be terminated from the study. The following assessments will be performed: HAM-D, HAM-A, and MADRS total scores and Clinical Global Impression – Improvement (CGI-I).

Part A may be terminated and Part B initiated if there is a clear signal of activity based on the HAM-D scores and/or other scales being assessed. Alternatively, upon completion of Part A, Part B may begin. The study may be terminated if there is clear lack of activity based on HAM-D scores during Part A. Separate cohorts of subjects will be enrolled in Part A and Part B; subjects participating in Part A cannot enroll in Part B.

Part B - Based on the results of Part A, eligible subjects will be stratified based on use of antidepressant treatment (current/stable or not treated/withdrawn  $\geq 30$  days) and randomized within each stratum to one of two treatment groups (SAGE-217 Oral Solution 30 mg or matching placebo) in a 1:1 ratio. Subjects will be administered study drug at 8:00 PM ( $\pm 15$  minutes) with food for 14 days. Subjects who cannot tolerate 30 mg will receive 20 mg for the rest of the Treatment Period. Subjects who cannot tolerate 20 mg will be terminated from the study.

In both parts of the study, subjects may be discharged after a minimum 7-day inpatient stay, following completion of the Day 7 assessments. If their clinical condition does not allow discharge, the Investigator may keep the subjects as inpatients for a longer period of time.

In both parts of the study, subjects discharged from the inpatient unit may receive treatment with study drug for the remainder of the 14-day Treatment Periods as outpatients. The outpatient phase treatment may be provided at the clinical site or, if suitable arrangements can be made, via home administration. Home administration of study drug will be performed according to a site-specific plan by a healthcare professional trained on the protocol and delivery of the study drug.

With the exception of subjects permitted to use current stable antidepressant treatment, initiation of psychotropic medications and other medications that may potentially have an impact on efficacy or safety endpoints will not be allowed between screening and completion of the Day 15 assessments (Parts A and B). Psychotropic medications, which must have been initiated at least 14 days prior to screening, must remain at a stable dose until completion of the Day 15 assessments (Parts A and B).

Efficacy and safety assessments will be performed periodically during the study, and blood samples will be collected for analysis of SAGE-217 as outlined in the Schedule of Events (Table 2 and Table 3).

**Follow-up Period:** Follow-up visits will be conducted on an outpatient basis. Follow-up visits for Parts A and B will be conducted at 1 week (21±1 day) and 2 weeks (28±3 days) after the last dose of study drug.

## **Objectives:**

#### Part A:

## **Primary:**

The primary objective of the study is to evaluate the safety and tolerability of SAGE-217 Oral Solution 30 mg.

## **Secondary:**

The secondary objective of Part A is to determine if treatment with SAGE-217 Oral Solution 30 mg for 14 days reduces depressive symptoms.

#### Part B:

## **Primary:**

The primary objective of the study is to evaluate the safety and tolerability of SAGE-217 Oral Solution 30 mg.

## Secondary:

The secondary efficacy objective for Part B of the study is to determine if treatment with SAGE-217 Oral Solution 30 mg reduces depressive symptoms in subjects with moderate to severe MDD compared to matching placebo.

#### **Endpoints:**

## Part A:

## **Primary:**

The primary endpoint is the safety and tolerability of SAGE-217 as assessed by the frequency and severity of adverse events; changes from baseline in clinical laboratory measures, vital signs, and electrocardiograms (ECGs); Stanford Sleepiness Scale (SSS) score; physical examination; and suicidal ideation using the Columbia-Suicide Severity Rating Scale (C-SSRS).

## **Secondary:**

Reduction in depressive symptoms as assessed by the following:

- Change from baseline in HAM-D total score at all time points;
- HAM-D response;
- HAM-D remission;
- Change from baseline in the MADRS total score at all time points;
- Change from baseline in HAM-D subscale and individual item scores at all time points; and
- CGI-I response.

## Part B:

## **Primary:**

The primary endpoint is the safety and tolerability of SAGE-217 as assessed by the frequency and severity of adverse events; changes from baseline in clinical laboratory measures, vital signs, and ECGs; SSS score; physical examination; and suicidal ideation using the C-SSRS.

#### **Secondary:**

Reduction in depressive symptoms, compared to placebo, as assessed by the following:

- Change from baseline in the 17-item HAM-D total score at all time points;
- HAM-D response;
- HAM-D remission;
- Change from baseline in the MADRS total score at all time points;
- Change from baseline in HAM-D subscale and individual item scores at all time points;
- CGI-I response; and
- 36-item short form survey (SF-36) and fatigue associated with depression (FAs-D) patient-reported outcome.

#### Pharmacokinetic:

The PK objective of Part A and Part B is:

• To assess the PK profile of SAGE-217 Oral Solution in plasma samples.

## Number of subjects (planned):

Approximately ten subjects will be enrolled in Part A. Up to 52 subjects may be randomized in Part B.

## Diagnosis and main criteria for inclusion:

## **Inclusion criteria:**

- 1. Subject has signed an ICF prior to any study-specific procedures being performed.
- 2. Subject is an ambulatory male or female between 18 and 65 years of age, inclusive.
- 3. Subject is in good physical health and has no clinically significant findings, as determined by the Investigator, on physical examination, 12-lead ECG, or clinical laboratory tests.
- 4. Subject agrees to adhere to the study requirements.
- 5. Subject has a diagnosis of MDD that has been present for at least a 4-week period as diagnosed by SCID-I.
- 6. Subject has a HAM-D total score of  $\geq$ 22 at screening and Day 1 (prior to dosing).
- 7. Subject has a HAM-A total score of ≥20 at screening and Day 1 (prior to dosing) (Part B only).
- 8. Subject is willing to delay start of other antidepressant or antianxiety medications and any new pharmacotherapy regimens, including as-needed benzodiazepine anxiolytics, during the screening and treatment periods.
- 9. Subject agrees to practice an acceptable method of highly effective birth control at screening and throughout study participation. Highly effective methods of birth control include sexual abstinence (for males and females); vasectomy; or a condom with spermicide in combination with a highly effective female partner's method (for males); and hormonal methods of contraception (ie, established use of oral, implantable, injectable, or transdermal hormones); placement of an intrauterine device; placement of an intrauterine system; and mechanical/barrier method of contraception (ie, condom or occlusive cap [diaphragm or cervical/vault cap] in conjunction with spermicide [foam, gel, film, cream, or suppository]) (for females).

#### **Exclusion criteria:**

- 1. Subject has a history of suicide attempt.
- 2. Subject has a recent history or active clinically significant manifestations of metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, musculoskeletal, dermatological, urogenital, neurological, or eyes, ears, nose, and throat disorders, or any other acute or chronic condition that, in the Investigator's opinion, would limit the subject's ability to complete or participate in this clinical study.
- 3. Subject has a history of treatment-resistant depression, defined as persistent depressive symptoms despite treatment with adequate doses of antidepressants from two different classes for an adequate amount of time (ie, at least 4 weeks of treatment).
- 4. Subject has a known allergy to SAGE-217, allopregnanolone, or related compounds.
- 5. Subject has a positive pregnancy test at screening or on Day 1 prior to the start of study drug administration.
- 6. Subject has detectable hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV), or human immunodeficiency virus (HIV) antibody at screening.
- 7. Subject has active psychosis per Investigator assessment.
- 8. Subject has a medical history of seizures.
- 9. Subject has a medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder.

- 10. Subject has a history of alcohol or drug dependence (including benzodiazepines) in the 12 months prior to screening.
- 11. Subject has had exposure to another investigational medication or device within 30 days prior to screening.
- 12. Subject has been treated or randomized in this study (eg, Part A) or any other study employing SAGE-217 previously (ie, subject may not have received study drug and then re-enroll).
- 13. Subject has had administration of psychotropics that have been initiated within 14 days prior to screening and/or are not being taken at a stable dose.
- 14. Use of any known strong inhibitors and/or inducers of cytochrome P450 (CYP)3A4 within the 14 days or five half-lives (whichever is longer) or consumed grapefruit juice, grapefruit, Seville oranges, or St. John's Wort or products containing these within 30 days prior to receiving the first dose of study drug.

## Investigational product, dosage and mode of administration:

SAGE-217 Oral Solution is available as a 6 mg/mL stock aqueous solution of SAGE-217 Drug Substance containing 40% hydroxypropyl- $\beta$ -cyclodextrin (HP $\beta$ CD) and 0.0025% sucralose, which is further diluted with Sterile Water for Injection to achieve the selected dose.

## **Duration of participation:**

<u>Part A</u>: Up to 38 days (14 days of treatment) <u>Part B</u>: Up to 38 days (14 days of treatment)

## Reference therapy, dosage and mode of administration:

Reference therapy is taste-matched placebo.

#### **Randomization:**

Subjects participating in Part A of the study will be administered study drug (SAGE-217 Oral Solution) in an open-label manner. Subjects in Part B will be randomized within each antidepressant treatment stratum to receive SAGE-217 Oral Solution or matching placebo oral solution in a 1:1 ratio. Subjects, clinicians, and the study team will be blinded to treatment allocation. The pharmacist and/or designated pharmacy staff, who will prepare the oral solutions according to the randomization schedule, will be unblinded.

## Dose Adjustment for Safety/Tolerability Reasons:

During the Treatment Period, subjects will be able to receive study drug as long as there are no dose-limiting safety/tolerability concerns. Subjects who experience moderate or severe adverse events that according to the clinical judgement of the Investigator are related to study drug while receiving the 30 mg dose of study drug will receive 20 mg for the remaining of the Treatment Period. Subjects who experience moderate or severe related adverse events while receiving the 20 mg dose of study drug may not be able to continue receiving study drug based on the evaluation and clinical judgment of the Investigator, and may be terminated from the study. Dosing may also be modified based on tolerability as assessed with SSS scores.

Part A may be terminated and Part B initiated if there is a clear signal of activity based on the HAM-D scores and/or other scales being assessed. The study may be terminated if there is clear lack of activity based on HAM-D scores during Part A. A Data Review Team will assess the HAM-D and other data on an ongoing basis during Part A.

## Inpatient Length of Stay and Discharge Instructions

The minimum length of inpatient stay in both parts of this study is 7 days. It is the Investigator's responsibility to assess whether the subject can safely be discharged home and continue taking study drug administered by a healthcare professional trained on the protocol and delivery of the study drug for the rest of the treatment days (Days 8 to 14 for Parts A and B) or by returning to the clinic daily. The Investigator may decide to extend the subject's inpatient stay to maximize safety oversight. In making this assessment, the Investigator may consider not only the drug tolerability but also clinical factors including, but not limited to, availability of social support, transportation, severity of symptoms, and suicidality.

Discharge instructions must include warnings about avoiding activities for which sedative effects of the study drug may impair performance, such as driving a motor vehicle and operating machinery.

## **Criteria for evaluation:**

#### **Efficacy:**

Reduction of depressive symptoms will be assessed by the change from baseline at various time points in HAM-D total score; HAM-D response; HAM-D remission; change from baseline in the MADRS total score; CGI-I response; change from baseline in HAM-D subscale and individual item scores; change from baseline in HAM-A total score; change from baseline in SF-36; and change from baseline in FAs-D.

## **Pharmacokinetics:**

Plasma samples will be collected to assay for concentrations of SAGE-217. The following PK parameters will be derived from the plasma concentrations (where evaluable): area under the concentration-time curve (AUC), AUC from time zero to infinity (AUC $_{\infty}$ ), maximum (peak) plasma concentration ( $C_{max}$ ), time at maximum (peak) plasma concentration ( $t_{max}$ ), steady-state drug concentration in the plasma during oral intake ( $C_{ss}$ ), and in the plasma at steady state during a dosing interval.

## Safety:

The safety and tolerability of SAGE-217 Oral Solution will be evaluated by frequency, type, and severity of adverse events; mean changes from baseline in clinical laboratory measures, vital signs, and ECGs; SSS score; physical examination; and suicidal ideation using the C-SSRS during both Part A and Part B.

## **Statistical methods:**

#### General

For the purpose of all safety and efficacy analyses where applicable, baseline is defined as the last measurement prior to the start of blinded study drug administration.

Continuous endpoints will be summarized with n, mean, standard deviation, median, minimum, and maximum. In addition, change from baseline values will be calculated at each time point and summarized descriptively. For categorical endpoints, descriptive summaries will include counts and percentages.

## **Analysis Populations and Methods:**

The Safety Population (for both Part A and Part B), defined as all subjects administered study drug, will be used to provide descriptive summaries of safety data. Adverse events will be classified by type, incidence, severity, and causality. The overall incidence of adverse events will be summarized by Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Data for vital signs, clinical laboratory measurements, ECG, physical examinations, and concomitant medication usage will also be summarized. Safety data will be summarized and examined for possible relationships between subject characteristics and plasma SAGE-217 concentrations, as appropriate. Suicidality data collected using the C-SSRS at baseline and at each visit during the active Treatment Period will be listed for all subjects. The C-SSRS listings will include behavior type and/or category for suicidal ideation and suicidal behavior of the C-SSRS. Out-of-range safety endpoints may be categorized as low or high, where applicable. Subjects will be summarized according to treatment received.

The Efficacy Population (for both Part A and Part B), defined as all subjects in the Safety Population who complete at least 1 day of dosing of study drug and have at least one post-baseline efficacy evaluation, will be used to analyze efficacy data. Efficacy data will be analyzed using appropriate descriptive statistics and pre-specified statistical methods, as well as other data presentation methods where applicable; subject listings will be provided for all efficacy data. For (the open-label) Part A, efficacy data will be summarized descriptively. For Part B, subjects will be analyzed according to randomized treatment.

For Part B, the change from baseline in HAM-D total score will be analyzed using a mixed effects model for repeated measures (MMRM); the model will include treatment, baseline HAM-D total score, antidepressant use strata, assessment time point, and time point-by-treatment as explanatory variables. All post-baseline time points will be included in the model. The primary comparison will be between SAGE-217 Oral Solution and matching placebo at the 15-day time point. Model-based point estimates (ie, least squares [LS] means), 95% confidence intervals, and p-values will be reported. An unstructured covariance structure will be used to model the within-subject errors. Continuous variables will be analyzed using similar methods.

Binary efficacy endpoints, including responder and remission endpoints, will be analyzed using logistic regression model.

The PK Population will consist of all subjects in the Safety Population with sufficient plasma concentrations for PK evaluations, and will be used to summarize PK data. PK parameters will be summarized using appropriate descriptive statistics and listed by subject. The PK parameters to be summarized where possible will include  $AUC_{\infty}$ ,  $C_{max}$ ,  $t_{max}$ ,  $t_{yz}$ , and  $C_{ss}$ .

## Sample Size Calculation

The sample size of ten subjects for Part A was selected based on clinical and not statistical considerations.

For Part B, assuming a two-sided t-test at an alpha level of 0.10, a sample size of 23 subjects per group would provide 80% power to detect an effect size of 0.75 between the SAGE-217 Oral Solution and matching placebo groups with regard to the secondary efficacy outcome variable of change from baseline in HAM-D total score. An effect size of 0.75 corresponds to a matching placebo-adjusted difference of 7.5 points in the change from baseline in HAM-D total score at 15 days with an assumed SD of 10 points. By including two treatment groups and using a 1:1 randomization, a total of 46 subjects are required. Assuming a non-evaluability rate of 10%, up to 52 subjects will be randomized.

**Table 2:** Schedule of Events (Part A)

| | <b>Screening Period</b> | | | | | ( | Open-L | abel Tr | eatmen | t Perio | d | | | | | Follo | ow-up Pe | eriod |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visits | OUTPATIENT | INPATIENT | | | | | | | INPATIENT or OUTPATIENT <sup>a</sup> | | | | | | | OUTPATIENT | | |
| Visit Days | D-7 to D-1 | D1* | D2 | D3 | D4 | D5 | D6 | <b>D7</b> | D8 | D9 | D10 | D11 | D12 | D13 | D14 | D15/<br>ET | D21<br>(+1d) | D28<br>(±3d) |
| Study Procedure | | | | | | | | | | | | | | | | | | |
| Informed Consent | X | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion | X | X | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | |
| Medical/Family History | X | | | | | | | | | | | | | | | | | |
| SCID-I | X | | | | | | | | | | | | | | | | | |
| Confinement | | | | | X | | | | | | | (X) | | | | | | |
| Physical Examination | X | | | | | | | | X | | | | | | | X | X | X |
| Body Weight/Height | X | | | | | | | | | | | | | | | X (wt<br>only) | X (wt<br>only) | X (wt only) |
| Clinical Laboratory<br>Assessments | X | | | | | | | | X | | | | | | | X | X | X |
| Drug & Alcohol Screen | X | X | | | | | | | | | | | | | | | | |
| Pregnancy Test | X | X | | | | | | | | | | | | | | X | | X |
| Hepatitis & HIV Screen | X | | | | | | | | | | | | | | | | | |
| Blood Sample | О | | | | | | | | | | | | | | | | | |
| Genetic Sample | 0 | | | | | | | | | | | | | | | | | |
| Vital Signs | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pulse Oximetry | | X | X | X | X | X | X | X | X | | | | | | | | | |
| 12-Lead ECG | X | X | X | | | | | X | | | | | | | X | | X | |
| C-SSRS | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| CGI-S | X | X | X | X | | | | | X | | | | | | | X | X | X |

| | <b>Screening Period</b> | | | | | ( | Open-L | abel Tr | eatmen | nt Perio | d | | | | | Foll | ow-up P | eriod |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visits | OUTPATIENT | INPATIENT | | | | | | INPATIENT or OUTPATIENT | | | | | | | OUTPATIENT | | | |
| Visit Days | D-7 to D-1 | D1* | D2 | D3 | D4 | D5 | D6 | <b>D7</b> | D8 | D9 | D10 | D11 | D12 | D13 | D14 | D15/<br>ET | D21<br>(+1d) | D28<br>(±3d) |
| Study Procedure | | | | | | | | | | | | | | | | | | |
| CGI-I <sup>k</sup> | | | X | X | | | | | X | | | | | | | X | X | X |
| HAM-A <sup>k</sup> | X | X | X | X | | | | | X | | | | | | | X | X | X |
| HAM-D <sup>k</sup> | X | X | X | X | X | X | X | X | X | | | | | | | X | X | X |
| MADRS <sup>k</sup> | X | X | X | X | X | X | X | X | X | | | | | | | X | X | X |
| SSS | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Plasma PK | | | | | | | | X | X | | | | | | X | X | | |
| Study Drug<br>Administration | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | |
| Adverse Events | | | | | | | | | X | | | | | | • | | | |
| Prior/Concomitant Medications | | | | | | | | | X | | | | | | | | | |

CGI-I = Clinical Global Impression - Improvement; CGI-S - Clinical Global Impression - Severity; C-SSRS = Columbia Suicide Severity Rating Scale; D = day; ET = early termination; ECG = electrocardiogram; HAM-A = Hamilton Anxiety Rating Scale; HAM-D = Hamilton Rating Scale for Depression, 17-item; HIV = human immunodeficiency virus; MADRS = Montgomery-Åsberg Depression Rating Scale; PK = pharmacokinetic; SCID-I = Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Axis I Disorders; SSS = Stanford Sleepiness Scale

- \*D1 procedures are to be completed prior to dosing
- <sup>a</sup> Outpatient visits may take place at the subject's residence or in the clinic.
- <sup>b</sup> Safety laboratory tests will include hematology, serum chemistry, coagulation, and urinalysis. Laboratory assessments are to be completed in the morning on Days 8 and 15 and during the follow-up visits on Day 21 and Day 28.
- <sup>c</sup> Urine toxicology for selected drugs of abuse and serum or breath test for alcohol.
- <sup>d</sup> Serum pregnancy test at screening and urine pregnancy test at Day 1 and Day 28.
- <sup>e</sup> Female subjects who prematurely discontinue will have a pregnancy test performed at the ET visit.
- f An optional blood sample for hormone and exploratory biochemistry testing, where consent is given.
- <sup>g</sup> An optional genetic sample for biomarker testing, where consent is given.
- h Vital signs include oral temperature (°C), respiratory rate, heart rate, and blood pressure (supine and standing). Vital signs will be obtained within ±5 minutes of the scheduled time point through 0.5 hours after dosing and ±30 minutes of the scheduled time point from 1 hour after dosing and greater, unless the subject is asleep between the hours of 23:00 h and 06:00 h. From Day 1 through Day 7, vital signs will be completed at the following time points: predose, 0.25, 0.5, 1, 2, and 12 hours after dosing. During the outpatient treatment period, vital signs will be completed prior to dosing and 1 hour after dosing. Vital signs may be repeated at the discretion of the Investigator or Visiting Home Healthcare Provider as clinically indicated.
- Will be performed 1 hour ±15 minutes after dosing on Days 1, 2, 7, and 14, and during the follow-up visit on Day 21.

- <sup>j</sup> The "Baseline/Screening" C-SSRS form will be completed at screening. The "Since Last Visit" C-SSRS form will be completed at any time of day at all subsequent time points.
- k To be completed to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28.
- To be completed within ±5 minutes of the scheduled time point through 0.5 hours after dosing and ±15 minutes of the scheduled time point from 1 hour after dosing and greater, unless the subject is asleep between 23:00 h and 06:00 h during the inpatient treatment period. From Day 1 through Day 7, SSS will be completed at the following time points: predose, 0.25, 0.5, 1, and 2 hours after dosing. During the outpatient treatment period, SSS will be completed prior to dosing and 1 hour after dosing.
- m Plasma samples for PK analysis in Part A and Part B will be collected predose and 0.25, 0.5, 1, 2, 10, and 12 hours postdose on Day 7 (within ±5 minutes of the scheduled time point through 0.5 hours after dosing and ±15 minutes of the scheduled time point from 1 hour after dosing and greater), prior to discharge on Day 8 for subjects being discharged or 16 hours postdose for subjects remaining as inpatients, predose on Day 14, and in the morning on Day 15. The time of study drug administration is time zero and all postdosing sampling times are relative to this time. In the event of a dose adjustment, an unscheduled PK sample should be collected just prior to the dose change. Plasma samples for PK analysis will be collected per protocol and subjects may need to be awoken for sample collection.
- <sup>n</sup> To include those taken within 30 days prior to informed consent and throughout the study.

 Table 3:
 Schedule of Events (Part B)

| | Screening Period | | | | Doul | ole-Blir | ıd, Plac | ebo-Co | ntrolle | d Treat | ment P | eriod | | | | Foll | ow-up Po | eriod |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visits | OUTPATIENT | INPATIENT | | | | | | | INPATIENT or OUTPATIENT <sup>a</sup> | | | | | | | OU | OUTPATIENT | |
| Visit Days | D-7 to D-1 | D1* | D2 | D3 | D4 | D5 | D6 | <b>D7</b> | D8 | D9 | D10 | D11 | D12 | D13 | D14 | D15/<br>ET | D21 (+1d) | D28<br>(±3d) |
| Study Procedure | | | | | | | | | | | | | | | | | | |
| Informed Consent | X | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion | X | X | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | |
| Medical/Family History | X | | | | | | | | | | | | | | | | | |
| SCID-I | X | | | | | | | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | | | | | | | |
| Confinement | | | | | X | | | | | | | (X) | | | | | | |
| Physical Examination | X | | | | | | | | X | | | | | | | X | X | X |
| Body Weight/Height | X | | | | | | | | | | | | | | | X (wt<br>only) | X (wt only) | X (wt<br>only) |
| Clinical Laboratory<br>Assessments | X | | | | | | | | X | | | | | | | X | X | X |
| Drug & Alcohol Screen | X | X | | | | | | | | | | | | | | | | |
| Pregnancy Test | X | X | | | | | | | | | | | | | | X | | X |
| Hepatitis & HIV Screen | X | | | | | | | | | | | | | | | | | |
| Blood Sample | О | | | | | | | | | | | | | | | | | |
| Genetic Sample | О | | | | | | | | | | | | | | | | | |
| Vital Signs | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pulse Oximetry | | X | X | X | X | X | X | X | X | | | | | | | | | |
| 12-Lead ECG | X | X | X | _ | | | _ | X | | | | | | | X | | X | |
| C-SSRS | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

| | <b>Screening Period</b> | | | | Doul | ole-Blir | d, Plac | ebo-Co | ntrolle | d Treat | ment P | eriod | | | | Foll | ow-up P | eriod |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visits | OUTPATIENT | INPATIENT | | | | | | INPATIENT or OUTPATIENT <sup>a</sup> | | | | | | | OUTPATIENT | | | |
| Visit Days | D-7 to D-1 | D1* | D2 | D3 | D4 | D5 | D6 | <b>D7</b> | D8 | D9 | D10 | D11 | D12 | D13 | D14 | D15/<br>ET | D21<br>(+1d) | D28<br>(±3d) |
| Study Procedure | | | | | | | | | | | | | | | | | | |
| CGI-S | X | X | X | X | | | | | X | | | | | | | X | X | X |
| CGI-I <sup>k</sup> | | | X | X | | | | | X | | | | | | | X | X | X |
| HAM-A <sup>k</sup> | X | X | X | X | | | | | X | | | | | | | X | X | X |
| HAM-D <sup>k</sup> | X | X | X | X | X | X | X | X | X | | | | | | | X | X | X |
| MADRS <sup>k</sup> | X | X | X | X | X | X | X | X | X | | | | | | | X | X | X |
| SF-36 <sup>k</sup> | X | X | | | | | | | X | | | | | | | X | X | X |
| FAs-D <sup>k</sup> | X | X | | | | | | | X | | | | | | | X | X | X |
| SSS | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Plasma PK | | | | | | | | X | X | | | | | | X | X | | |
| Study Drug<br>Administration | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | |
| Adverse Events | | | | | | | | | X | | | | | | | | • | |
| Prior/Concomitant<br>Medications | | | | | | | | | X | | | | | | | | | |

CGI-I = Clinical Global Impression - Improvement; CGI-S - Clinical Global Impression - Severity; C-SSRS = Columbia Suicide Severity Rating Scale; D = day; ET = early termination; ECG = electrocardiogram; FAs-D = fatigue associated with depression; HAM-A = Hamilton Anxiety Rating Scale; HAM-D = Hamilton Rating Scale for Depression, 17-item; HIV = human immunodeficiency virus; MADRS = Montgomery-Åsberg Depression Rating Scale; PK = pharmacokinetic; SCID-I = Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Axis I Disorders; SF-36 = 36-item short form survey; SSS = Stanford Sleepiness Scale \*D1 procedures are to be completed prior to dosing

<sup>&</sup>lt;sup>a</sup> Outpatient visits may take place at the subject's residence or in the clinic.

<sup>&</sup>lt;sup>b</sup> Safety laboratory tests will include hematology, serum chemistry, coagulation, and urinalysis. Laboratory assessments are to be completed in the morning on Days 8 and 15 and during the follow-up visits on Day 21 and Day 28.

<sup>&</sup>lt;sup>c</sup> Urine toxicology for selected drugs of abuse and serum or breath test for alcohol.

<sup>&</sup>lt;sup>d</sup> Serum pregnancy test at screening and urine pregnancy test at Day 1 and Day 28.

<sup>&</sup>lt;sup>e</sup> Female subjects who prematurely discontinue will have a pregnancy test performed at the ET visit.

f An optional blood sample for hormone and exploratory biochemistry testing, where consent is given.

g An optional genetic sample for biomarker testing, where consent is given.

- h Vital signs include oral temperature (°C), respiratory rate, heart rate, and blood pressure (supine and standing). Vital signs will be obtained within ±5 minutes of the scheduled time point through 0.5 hours after dosing and ±30 minutes of the scheduled time point from 1 hour after dosing and greater, unless the subject is asleep between the hours of 23:00 h and 06:00 h. From Day 1 through Day 7, vital signs will be completed at the following time points: predose, 0.25, 0.5, 1, 2, and 12 hours after dosing. During the outpatient treatment period, vital signs will be completed prior to dosing and 1 hour after dosing. Vital signs may be repeated at the discretion of the Investigator or Visiting Home Healthcare Provider as clinically indicated.
- Will be performed 1 hour ±15 minutes after dosing on Days 1, 2, 7, and 14, and during the follow-up visit on Day 21.
- The "Baseline/Screening" C-SSRS form will be completed at screening. The "Since Last Visit" C-SSRS form will be completed at any time of day at all subsequent time points.
- k To be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28.
- <sup>1</sup> To be completed within ±5 minutes of the scheduled time point through 0.5 hours after dosing and ±15 minutes of the scheduled time point from 1 hour after dosing and greater, unless the subject is asleep between 23:00 h and 06:00 h during the inpatient treatment period. From Day 1 through Day 7, SSS will be completed at the following time points: predose, 0.25, 0.5, 1, and 2 hours after dosing. During the outpatient treatment period, SSS will be completed prior to dosing and 1 hour after dosing.
- m Plasma samples for PK analysis in Part A and Part B will be collected predose and 0.25, 0.5, 1, 2, 10, and 12 hours postdose on Day 7 (within ±5 minutes of the scheduled time point through 0.5 hours after dosing and ±15 minutes of the scheduled time point from 1 hour after dosing and greater), prior to discharge on Day 8 for subjects being discharged or 16 hours postdose for subjects remaining as inpatients, predose on Day 14, and in the morning on Day 15. The time of study drug administration is time zero and all postdosing sampling times are relative to this time. In the event of a dose adjustment, an unscheduled PK sample should be collected just prior to the dose change. Plasma samples for PK analysis will be collected per protocol and subjects may need to be awoken for sample collection.
- <sup>n</sup> To include those taken within 30 days prior to informed consent and throughout the study.

# 3. TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES

## **TABLE OF CONTENTS**

| 1. | TITLE PAGE | 1 |
|---|---|---|
| 2. | SYNOPSIS | 5 |
| 3. | TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES | 18 |
| 4. | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 23 |
| 5. | INTRODUCTION | 25 |
| 5.1. | Background of Major Depressive Disorders and Unmet Medical Need | 25 |
| 5.2. | SAGE-217 Oral Solution | 26 |
| 5.3. | Summary of Nonclinical and Clinical Experience with SAGE-217 | 26 |
| 5.3.1. | Nonclinical Studies with SAGE-217 | 26 |
| | | 26 |
| | | 28 |
| 5.5. | Dose Justification. | 28 |
| 6. | STUDY OBJECTIVES AND PURPOSE | 29 |
| 6.1. | Part A | 29 |
| 6.1.1. | Primary Objective | 29 |
| 6.1.2. | Secondary Objective | 29 |
| 6.2. | Part B | 29 |
| 6.2.1. | Primary Objective | 29 |
| 6.2.2. | Secondary Objective | 29 |
| 6.3. | Pharmacokinetic Objective | 29 |
| 6.4. | Endpoints | 29 |
| 6.4.1. | Part A | 29 |
| 6.4.1.1. | Primary | 29 |
| 6.4.1.2. | Secondary | 29 |
| 6.4.2. | Part B | 30 |
| 6.4.2.1. | Primary | 30 |
| 6.4.2.2. | Secondary | 30 |
| 7. | INVESTIGATIONAL PLAN | 31 |
| 7.1. | Overall Study Design | 31 |

| 7.2. | Blinding and Randomization | 32 |
|---------|--------------------------------------------------------|----|
| 8. | SELECTION AND WITHDRAWAL OF SUBJECTS | 34 |
| 8.1. | Subject Inclusion Criteria | 34 |
| 8.2. | Subject Exclusion Criteria | 34 |
| 8.3. | Subject Withdrawal Criteria | 35 |
| 8.3.1. | Study Drug Withdrawal | 35 |
| 8.3.2. | Criteria for Study Termination | 36 |
| 9. | TREATMENT OF SUBJECTS | 37 |
| 9.1. | Number of Subjects | 37 |
| 9.2. | Treatment Assignment | 37 |
| 9.2.1. | Part A | 37 |
| 9.2.2. | Part B | 37 |
| 9.3. | Dose Adjustment Criteria | 37 |
| 9.4. | Prior/Concomitant Medications | 38 |
| 9.4.1. | Prior/Concomitant Medications | 38 |
| 9.4.2. | Restricted Medications | 38 |
| 9.5. | Treatment Compliance | 39 |
| 10. | STUDY DRUG MATERIALS AND MANAGEMENT | 40 |
| 10.1. | Study Drug | 40 |
| 10.2. | Batch Formula for Stock SAGE-217 Oral Solution 6 mg/mL | |
| 10.3. | Study Drug Packaging and Labeling | 40 |
| 10.4. | Study Drug Storage | 41 |
| 10.5. | Administration and Study Drug Accountability | 41 |
| 10.5.1. | Study Drug Administration | 42 |
| 10.5.2. | Study Drug Accountability | 42 |
| 10.6. | Study Drug Handling and Disposal | 42 |
| 11. | ASSESSMENT OF EFFICACY | 43 |
| 11.1. | Hamilton Rating Scale for Depression (HAM-D) | 43 |
| 11.2. | Montgomery-Åsberg Depression Rating Scale (MADRS) | 43 |
| 11.3. | Hamilton Anxiety Rating Scale (HAM-A) | 44 |
| 11.4. | Clinical Global Impression (CGI) | 44 |
| 11.5. | Short Form-36 (SF-36) | 45 |

| 11.6. | The Fatigue Associated With Depression (FAs-D) Patient-Reported Outcome (PRO) | 45 |
|---|---|---|
| 12. | PHARMACOKINETICS | 46 |
| 12.1. | Blood Sample Collection | 46 |
| 12.2. | Storage and Shipment of Pharmacokinetic Samples | 46 |
| 12.3. | Sample Analysis | 46 |
| 13. | ASSESSMENT OF SAFETY | 47 |
| 13.1. | Safety Parameters | 47 |
| 13.1.1. | Demographic/Medical History | 47 |
| 13.1.2. | Vital Signs | 47 |
| 13.1.3. | Weight and Height | 47 |
| 13.1.4. | Physical Examination | 47 |
| 13.1.5. | Electrocardiogram (ECG) | 47 |
| 13.1.6. | Laboratory Assessments | 47 |
| 13.1.6.1. | Hematology | 48 |
| 13.1.6.2. | Blood Chemistry | 48 |
| 13.1.6.3. | Urinalysis | 48 |
| 13.1.6.4. | Hormones and Exploratory Biochemistry | 48 |
| 13.1.6.5. | Virus Serology | 48 |
| 13.1.6.6. | Pregnancy Test | 48 |
| 13.1.6.7. | Genetic Testing | 49 |
| 13.1.6.8. | Drugs of Abuse and Alcohol | 49 |
| 13.1.7. | Columbia-Suicide Severity Rating Scale (C-SSRS) | 49 |
| 13.1.8. | Stanford Sleepiness Scale (SSS) | 50 |
| 13.2. | Adverse and Serious Adverse Events | 50 |
| 13.2.1. | Definition of Adverse Events | 50 |
| 13.2.1.1. | Adverse Event | 50 |
| 13.2.1.2. | Suspected Adverse Reaction | 50 |
| 13.2.1.3. | Serious Adverse Event | 50 |
| 13.3. | Relationship to Study Drug | 51 |
| 13.4. | Recording Adverse Events | 51 |
| 13.5. | Reporting Adverse Events | 52 |
| 13.6. | Emergency Identification of Study Drug | 52 |

| 14. | STATISTICS | 54 |
|---------|-------------------------------------------|----|
| 14.1. | Data Analysis Sets | 54 |
| 14.1.1. | Analysis Populations and Methods | 54 |
| 14.2. | Handling of Missing Data | 54 |
| 14.3. | General Considerations | 54 |
| 14.4. | Demographics and Baseline Characteristics | 54 |
| 14.5. | Efficacy Analyses | 54 |
| 14.6. | Safety Analyses | 55 |
| 14.6.1. | Adverse Events | 56 |
| 14.6.2. | Clinical Laboratory Evaluations | 56 |
| 14.6.3. | Physical Examinations | 56 |
| 14.6.4. | Vital Signs | 56 |
| 14.6.5. | 12-Lead Electrocardiogram | 56 |
| 14.6.6. | Prior and Concomitant Medications | 56 |
| 14.6.7. | Columbia Suicide Severity Rating Scale | 57 |
| 14.6.8. | Stanford Sleepiness Scale | 57 |
| 14.7. | Pharmacokinetic Analyses | 57 |
| 14.8. | Determination of Sample Size | 57 |
| 14.9. | Changes From Protocol Specified Analyses | 57 |
| 15. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 58 |
| 15.1. | Study Monitoring | 58 |
| 15.2. | Audits and Inspections | 58 |
| 15.3. | Institutional Review Board (IRB) | 59 |
| 16. | QUALITY CONTROL AND QUALITY ASSURANCE | 60 |
| 17. | ETHICS | 61 |
| 17.1. | Ethics Review | 61 |
| 17.2. | Ethical Conduct of the Study | 61 |
| 17.3. | Written Informed Consent | 61 |
| 18. | DATA HANDLING AND RECORDKEEPING | 62 |
| 18.1. | Inspection of Records | 62 |
| 18.2. | Retention of Records | 62 |
| 18.3. | Confidentiality | 62 |
| 19 | PUBLICATION POLICY | 64 |

| | 7-MDD-201 S<br>24 October 2016 | age Therapeutics |
|---|---|---|
| 20. | LIST OF REFERENCES | 65 |
| 21. | APPENDICES | 67 |
| APPENDIX | X 1. HAMILTON RATING SCALE FOR DEPRESSION, 17-ITEM (HAM-D) | |
| APPENDIX | X 2. MONTGOMERY-ÅSBERG DEPRESSION RATING SCALE (MADRS) | |
| APPENDIX | X 3. HAMILTON ANXIETY RATING SCALE (HAM-A) | 71 |
| APPENDIX | X 4. CLINICAL GLOBAL IMPRESSION—IMPROVEMENT SCA (CGI-I) AND SEVERITY SCALE (CGI-S) | <del></del> _ |
| APPENDIX | X 5. SHORT-FORM 36 (SF-36) | 73 |
| APPENDIX | X 6. THE FATIGUE ASSOCIATED WITH DEPRESSION (FAS-I<br>PATIENT-REPORTED OUTCOME (PRO) | |
| APPENDIX | X 7. COLUMBIA - SUICIDE SEVERITY RATING SCALE (C-SS | RS)80 |
| APPENDIX | X 8. STANFORD SLEEPINESS SCALE (SSS) | 86 |
| | LIST OF TABLES | |
| Table 1: | Emergency Contact Information. | 4 |
| Table 2: | Schedule of Events (Part A) | 12 |
| Table 3: | Schedule of Events (Part B) | 15 |
| Table 4: | Abbreviations and Specialist Terms | 23 |
| Table 5: | Batch Formula for 125 mL of Stock SAGE-217 Oral Solution 6 mg/ | mL40 |

## 4. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

The following abbreviations and specialist terms are used in this study protocol.

**Table 4:** Abbreviations and Specialist Terms

| Abbreviation or Specialist Term | Explanation |
|---|---|
| AUC | area under the concentration-time curve |
| $\mathrm{AUC}_{\infty}$ | area under the concentration-time curve from time zero to infinity |
| BMI | body mass index |
| CGI-I | Clinical Global Impression - Improvement |
| CGI-S | Clinical Global Impression - Severity |
| C <sub>max</sub> | maximum (peak) plasma concentration |
| CS | clinically significant |
| Css | steady-state drug concentration in the plasma during oral intake |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CYP450 | cytochrome P450 |
| DSM-5 | Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EP | European Pharmacopeia |
| FAs-D | fatigue associated with depression |
| GABA | γ-aminobutyric acid |
| GABA <sub>A</sub> | γ-aminobutyric acid-ligand gated chloride channel |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HAM-A | Hamilton Anxiety Rating Scale |
| HAM-D | 17-item Hamilton Rating Scale for Depression |
| HBsAg | hepatitis B surface antigen |
| HCV | hepatitis C virus |
| HIV | human immunodeficiency virus |
| НРВСО | hydroxypropyl-β-cyclodextrin |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |

| Abbreviation or Specialist Term | Explanation |
|---|---|
| IRB | Institutional Review Board |
| MAD | multiple-ascending dose |
| MADRS | Montgomery-Åsberg Depression Rating Scale |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MDD | major depressive disorders |
| MMRM | mixed effects model for reported measures |
| MTD | maximum tolerated dose |
| n | number |
| NCS | not clinically significant |
| NF | National Formulary |
| PK | pharmacokinetic(s) |
| PPD | postpartum depression |
| SAD | single-ascending dose |
| SCID-I | Structured Clinical Interview for DSM-5 Axis I Disorders |
| SD | standard deviation |
| SF-36 | 36-item short form survey |
| SOC | system organ class |
| SRC | Safety Review Committee |
| SSS | Stanford Sleepiness Scale |
| TEAE | treatment-emergent adverse event |
| t <sub>max</sub> | time at maximum (peak) plasma concentration |
| USP | United States Pharmacopeia |
| WHO | World Health Organization |
| WHO-DD | World Health Organization-Drug Dictionary |

## 5. INTRODUCTION

## 5.1. Background of Major Depressive Disorders and Unmet Medical Need

World Health Organization (WHO) has identified depression as the leading cause of disability worldwide, and a major contributor to the overall global burden of disease (<a href="http://www.who.int/mediacentre/factsheets/fs369/en/">http://www.who.int/mediacentre/factsheets/fs369/en/</a>). Globally, depression has been estimated to affect 350 million people.

In DSM-5, depression refers to an overarching set of diagnoses, including disruptive mood dysregulation disorder, major depressive disorder, persistent depressive disorder (dysthymia), premenstrual dysphoric disorder, substance/medication-induced depressive disorder, depressive disorder due to another medical condition, other specified depressive disorder, and unspecified depressive disorder.

In the US, the economic burden of depression, including workplace costs, direct costs and suicide-related costs, was estimated to be \$210.5 billion in 2010 (Greenberg 2015). As per WHO statistics, over 800,000 people die due to suicide every year, and suicide is the second leading cause of death in 15- to 29-year-olds. In the US, an estimated 10% to 15% of individuals with depression commit suicide (Angst 1999).

Antidepressants are mainstay of pharmacological treatment for depressive disorders. Selective serotonin reuptake inhibitors, serotonin and norepinephrine reuptake inhibitors, tricyclic antidepressants, monoamine oxidase inhibitors, and other compounds that affect monoaminergic neurotransmission, such as mirtrazapine and bupropion, represent the major classes of antidepressants. While antidepressants are widely used, large scale studies have demonstrated their limited efficacy. For example, in the STAR\*D trial where over 2800 patients were treated in "real world" settings, the HAM-D remission rate was 28% following 14 weeks of treatment with citalopram, a typical selective serotonin reuptake inhibitor (Trivedi 2006). Recent studies have shown a number of symptoms that remain untreated, such as cognitive impairment, sleep disturbances and anxiety, even in patients that are in remission over a long period of time after treatment (Conradi 2011; Romera 2013). A close examination of randomized placebo-controlled trials of antidepressants approved by the Food and Drug Administration in the treatment of both major or minor depressive disorders demonstrated Cohen's *d* effect sizes below 0.2 and high placebo response rates (Kirsch 2008; Fournier 2010), emphasizing the challenges in assessing antidepressant drug efficacy and the unmet need in the treatment of depression.

Converging preclinical and clinical evidence (Gerner 1981; Honig 1988; Drugan 1989; Luscher 2011; Mann 2014) implicates deficits in GABAergic neurotransmission in the pathophysiology of depressive disorders including MDD and PPD. Furthermore, several pieces of experimental data implicate deficiencies in the normal regulation of endogenous neuroactive steroids in depressive disorders (Maguire 2008; Maguire 2009). The neuroactive steroid class of compounds includes the endogenous neuroactive steroid, allopregnanolone. Allopregnanolone is a positive allosteric modulator of both synaptic and extrasynaptic GABA<sub>A</sub> receptors – the prominent inhibitory transmitter system in the brain. Depressed patients show low levels of GABA in the brain and of neurosteroids in the CSF and plasma, and antidepressant therapy

restores GABA levels in relevant animal models and neurosteroid concentrations in depressed patients (Luscher 2011; Schüle 2014).

## 5.2. SAGE-217 Oral Solution

The intended dosage form for oral administration is SAGE-217 Oral Solution to be compounded at the clinical pharmacy from components supplied by the Sponsor (SAGE-217 Drug Substance Powder in the Bottle, Excipients in the Bottle, and sucralose) and Sterile Water for Injection. SAGE-217 Oral Solution is a clear, colorless, aqueous hydroxypropyl-β-cyclodextrin (HPβCD) solution of SAGE-217 Drug Substance. One concentration, 6 mg/mL, is available for use in clinical studies. In addition to SAGE-217 Drug Substance, SAGE-217 Oral Solution contains HPβCD HPB Parenteral Grade, United States Pharmacopeia/European Pharmacopeia [USP/EP], to solubilize the drug substance, sucralose (USP/National Formulary [NF], to sweeten the solution, and water for injection to be provided by the clinical pharmacy. Refer to Table 5 for the composition of SAGE-217 Oral Solution 6 mg/mL.

The SAGE-217 Oral Solution 6 mg/mL stock solution is compounded at point of use. This stock solution is for oral administration after dilution to the intended dose by the clinical pharmacy.

## 5.3. Summary of Nonclinical and Clinical Experience with SAGE-217

## 5.3.1. Nonclinical Studies with SAGE-217

In nonclinical studies of SAGE-217, sedative-hypnotic effects were consistently observed at higher doses in both in vivo pharmacology studies and toxicology studies. The sedative-hypnotic impairments seen with SAGE-217 were typical for GABAA positive allosteric modulators, ranging from hyperexcitability and ataxia at the lower doses through deep sedation and ultimately anesthesia at higher doses. Depth and duration of sedation demonstrated a clear dose response over the range tested, with evidence of tolerance occurring with continued exposure. Tolerance to the effects of SAGE-217 on motor incoordination was not observed after 7 days of dosing.

The compound has been assessed in 14-day rat and dog toxicology studies with daily administration of SAGE-217 as a solution in HPβCD in dogs and Labrasol® in rats. The no-observed-adverse-effect-level was 3 mg/kg (females) and 22.5 mg/kg (males) in rats and 2.5 mg/kg in dogs. There were no adverse effects in dogs or rats in the main toxicology studies. A single observation of mortality occurred in one female rat at the high dose in a toxicokinetic study that was suspected to have been related to exaggerated pharmacology. Additional toxicology and pharmacology information is provided in the Investigator's Brochure.







## 5.5. Dose Justification

To date, the pharmacokinetics of SAGE-217 Oral Solution has been investigated in healthy volunteers within the context of the SAD and MAD studies (217-CLP-101 and 217-CLP-102, respectively). The MTD was determined to be 55 mg in the SAD study and 30 mg once daily (either AM or PM dosing) in the MAD study. Thus as a first step, while ensuring tolerability, a 30 mg dose has been chosen to maximize the potential therapeutic benefit in this first clinical study of MDD.

## 6. STUDY OBJECTIVES AND PURPOSE

## **6.1.** Part A

## 6.1.1. Primary Objective

The primary objective of the study is to evaluate the safety and tolerability of SAGE-217 Oral Solution 30 mg.

## 6.1.2. Secondary Objective

The secondary objective of Part A is to determine if treatment with SAGE-217 Oral Solution 30 mg for 14 days reduces depressive symptoms.

## **6.2.** Part B

## **6.2.1.** Primary Objective

The primary objective of the study is to evaluate the safety and tolerability of SAGE-217 Oral Solution 30 mg.

## **6.2.2.** Secondary Objective

The secondary efficacy objective for Part B of the study is to determine if treatment with SAGE-217 Oral Solution 30 mg reduces depressive symptoms in subjects with moderate to severe MDD compared to matching placebo.

## 6.3. Pharmacokinetic Objective

The PK objective of Part A and Part B is to assess the PK profile of SAGE-217 Oral Solution in plasma samples.

## 6.4. Endpoints

## 6.4.1. Part A

## **6.4.1.1.** Primary

The primary endpoint is the safety and tolerability of SAGE-217 as assessed by the frequency and severity of adverse events; changes from baseline in clinical laboratory measures, vital signs, and electrocardiograms (ECGs); Stanford Sleepiness Scale (SSS) score; physical examination; and suicidal ideation using the Columbia-Suicide Severity Rating Scale (C-SSRS).

## **6.4.1.2.** Secondary

Reduction in depressive symptoms as assessed by the following:

• Change from baseline in HAM-D total score at all time points;

- HAM-D response (defined as having a 50% or greater reduction from baseline in HAM-D total score);
- HAM-D remission (defined as having a HAM-D total score of  $\leq 7$ );
- Change from baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score at all time points;
- Change from baseline in HAM-D subscale and individual item scores at all time points;
- Change from baseline in Hamilton Anxiety Rating Scale (HAM-A) total score at all time points; and
- Clinical Global Impression Improvement (CGI-I) response (defined as a CGI-I score of "very much improved" or "much improved").

## 6.4.2. Part B

## **6.4.2.1.** Primary

The primary endpoint is the safety and tolerability of SAGE-217 as assessed by the frequency and severity of adverse events; changes from baseline in clinical laboratory measures, vital signs, and ECGs; SSS score; physical examination; and suicidal ideation using the C-SSRS.

## **6.4.2.2.** Secondary

Reduction in depressive symptoms, compared to placebo, as assessed by the following:

- Change from baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D) total score at all time points;
- HAM-D response;
- HAM-D remission:
- Change from baseline in the MADRS total score at all time points;
- Change from baseline in HAM-D subscale and individual item scores at all time points;
- Change from baseline in HAM-A total score at all time points;
- CGI-I response; and
- 36-item short form survey (SF-36) and fatigue associated with depression (FAs-D) patient-reported outcome.

## 7. INVESTIGATIONAL PLAN

## 7.1. Overall Study Design

This study is a two-part, multicenter, Phase 2a study to evaluate the safety, tolerability, PK, and efficacy of SAGE-217 Oral Solution in approximately 62 adult subjects with MDD. Part A of the study is an open-label design with SAGE-217 Oral Solution dosing for 14 days. Part B of the study is a randomized, double-blind, parallel-group, placebo-controlled design with SAGE-217 Oral Solution or matching placebo dosing for 14 days. Separate cohorts of subjects will be enrolled in Part A and Part B; subjects participating in Part A cannot enroll in Part B.

Parts A and B of the study will consist of an up to 7-day Screening Period (Days -7 to -1), a 14-day Treatment Period, and a 2-week Follow-up Period (through Day 28).

During the Screening Period (Day -7 to Day -1), after signing the informed consent form (ICF), subjects will be assessed for study eligibility, and the severity of each subject's MDD will be evaluated using HAM-D. The Screening Period assessments will be conducted on an outpatient basis.

If applicable, standard of care data collected prior to obtaining informed consent may also be included as screening data, if appropriate, such as laboratory tests, ECG, physical examination, and vital signs conducted within the preceding 48 hours, as long as the requirement for the screening assessment to be collected retrospectively is met in full. If applicable, to ensure protocol compliance, any standard of care data eligible for inclusion as screening data must include the precise nature and timing of data collection.

During the 14-day study Treatment Period of Parts A and B, subjects must remain inpatient for the first 7 days at minimum and per Investigator's judgement thereafter. The Follow-up Period assessments will be conducted on an outpatient basis.

The study will be conducted in two parts:

- Part A: Beginning on Day 1, subjects will receive open-label SAGE-217 Oral Solution at 8:00 PM (±15 minutes) with food (as outlined in Section 9.2.1). Subjects will receive SAGE-217 Oral Solution 30 mg from Day 1 to Day 14 as tolerated.
- Part B: Based on the results of Part A, eligible subjects will be stratified based on use of antidepressant treatment (current/stable or not treated/withdrawn ≥30 days) and randomized within each stratum in a 1:1 fashion to receive SAGE-217 Oral Solution or matching placebo for 14 days beginning on Day 1 as tolerated. All doses of study drug will be administered at 8:00 PM (±15 minutes) with food as outlined in Section 9.2.2.

Part A may be terminated and Part B initiated if there is a clear signal of activity based on the HAM-D scores and/or other scales being assessed. Alternatively, upon completion of Part A, Part B may begin. The study may be terminated if there is clear lack of activity based on HAM-D scores during Part A.

In Part A and Part B, study drug (SAGE-217 Oral Solution or matching placebo) will be administered at the study center for at least the first 7 days of the Treatment Period, which

includes Day 1 of study drug administration through completion of study drug administration on Day 14. Subjects may be discharged after a minimum 7-day inpatient stay, following completion of the Day 7 assessments. If their clinical condition does not allow discharge, the Investigator may keep the subjects as inpatients for a longer period of time. Subjects discharged from the inpatient unit may receive treatment with study drug for the remainder of the 14-day Treatment Period as outpatients. For the outpatient phase, dosing will be done at the clinical site or, if suitable arrangements can be made, via home administration where local regulations allow. Home administration of study drug will be performed according to a site-specific plan by a healthcare professional trained on the protocol and delivery of the study drug.

Subjects will be monitored for safety during the Treatment and Follow-up Periods including monitoring for adverse events/serious adverse events, routine clinical laboratory assessments, physical examination, vital signs, and ECG.

During the Treatment Period, subjects will be able to receive study drug as long as there are no dose-limiting safety/tolerability concerns. Subjects who experience moderate or severe adverse events that according to the clinical judgement of the Investigator are related to study drug while receiving the 30 mg dose of study drug will receive 20 mg for the remaining of the Treatment Period. Subjects who experience moderate or severe related adverse events while receiving the 20 mg dose of study drug may not be able to continue receiving study drug based on the evaluation and clinical judgment of the Investigator, and may be terminated from the study.

Dosing may also be modified based on tolerability as assessed with SSS scores. Any SSS score of  $\geq 6$  will be reassessed within 10 minutes. If a subject is receiving the 30 mg dose of study drug and has an SSS score of  $\geq 6$  that is confirmed on repeat assessment during normal waking hours, the dose will be decreased to 20 mg for the rest of the Treatment Period. If a subject is receiving the 20 mg dose of study drug and has an SSS score of  $\geq 6$  that is confirmed on repeat assessment during normal waking hours, then study drug will be discontinued and the subject will be terminated from the study.

## 7.2. Blinding and Randomization

Part A is open-label with no control group; therefore, there will be no randomization or blinding.

Part B is a double-blind, placebo-controlled study. Subjects who meet the entrance criteria will be stratified based on use of antidepressant treatment (current/stable or not treated/withdrawn ≥30 days) and randomly assigned within each stratum in a 1:1 ratio to receive SAGE-217 Oral Solution or taste-matched placebo according to a computer-generated randomization schedule. Once it has been determined that a subject meets eligibility criteria, the subject will be sequentially assigned a subject number from the randomization schedule provided to the unblinded pharmacist. Subject identification numbers will consist of the site number (eg, "01") followed by numbering starting with double zero (eg, 01-001, 01-002, 01-003 through 01-062).

The randomization schedule will be generated using SAS V9.2 or later. Only the clinic pharmacist or designated pharmacy staff, who is responsible for preparing the solutions, will be given a copy of the randomization schedule. In the event of a medical emergency, the pharmacist may reveal actual solution contents to the Investigator, who should also alert Sage of the emergency (see Section 13.6 for more details related to unblinding). In all cases where the study drug allocation for a subject is unblinded, pertinent information (including the reason for

Protocol 217-MDD-201 Version 1.0 24 October 2016 Sage Therapeutics

unblinding) must be documented in the subject's records and on the electronic case report form (eCRF). If the subject or study center personnel (other than pharmacist) have been unblinded, the subject will be terminated from the study. In addition, an unblinded Monitor will perform drug accountability during the study.

## 8. SELECTION AND WITHDRAWAL OF SUBJECTS

## 8.1. Subject Inclusion Criteria

The following inclusion criteria must be met for individuals to be eligible for the study.

- 1. Subject has signed an ICF prior to any study-specific procedures being performed.
- 2. Subject is an ambulatory male or female between 18 and 65 years of age, inclusive.
- 3. Subject is in good physical health and has no clinically significant findings, as determined by the Investigator, on physical examination, 12-lead ECG, or clinical laboratory tests.
- 4. Subject agrees to adhere to the study requirements.
- 5. Subject has a diagnosis of MDD that has been present for at least a 4-week period as diagnosed by Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Axis I Disorders (SCID-I).
- 6. Subject has a HAM-D total score of  $\geq 22$  at screening and Day 1 (prior to dosing).
- 7. Subject has a HAM-A total score of ≥20 at screening and Day 1 (prior to dosing) (Part B only).
- 8. Subject is willing to delay start of other antidepressant or antianxiety medications and any new pharmacotherapy regimens, including as-needed benzodiazepine anxiolytics, during the screening and treatment periods.
- 9. Subject agrees to practice an acceptable method of highly effective birth control at screening and throughout study participation. Highly effective methods of birth control include sexual abstinence (for males and females); vasectomy; or a condom with spermicide in combination with a highly effective female partner's method (for males); and hormonal methods of contraception (ie, established use of oral, implantable, injectable, or transdermal hormones); placement of an intrauterine device; placement of an intrauterine system; and mechanical/barrier method of contraception (ie, condom or occlusive cap [diaphragm or cervical/vault cap] in conjunction with spermicide [foam, gel, film, cream, or suppository]) (for females).

## 8.2. Subject Exclusion Criteria

Subjects will be excluded if they meet any of the following exclusion criteria.

- 1. Subject has a history of suicide attempt.
- 2. Subject has a recent history or active clinically significant manifestations of metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, musculoskeletal, dermatological, urogenital, neurological, or eyes, ears, nose, and throat disorders, or any other acute or chronic condition that, in the Investigator's opinion, would limit the subject's ability to complete or participate in this clinical study.

- 3. Subject has a history of treatment-resistant depression, defined as persistent depressive symptoms despite treatment with adequate doses of antidepressants from two different classes for an adequate amount of time (ie, at least 4 weeks of treatment).
- 4. Subject has a known allergy to SAGE-217, allopregnanolone, or related compounds.
- 5. Subject has a positive pregnancy test at screening or on Day 1 prior to the start of study drug administration.
- 6. Subject has detectable hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV), or human immunodeficiency virus (HIV) antibody at screening.
- 7. Subject has active psychosis per Investigator assessment.
- 8. Subject has a medical history of seizures.
- 9. Subject has a medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder.
- 10. Subject has a history of alcohol or drug dependence (including benzodiazepines) in the 12 months prior to screening.
- 11. Subject has had exposure to another investigational medication or device within 30 days prior to screening.
- 12. Subject has been treated or randomized in this study (eg, Part A) or any other study employing SAGE-217 previously (ie, subject may not have received study drug and then re-enroll).
- 13. Subject has had administration of psychotropics that have been initiated within 14 days prior to screening and/or are not being taken at a stable dose.
- 14. Use of any known strong inhibitors and/or inducers of CYP3A4 within the 14 days or five half-lives (whichever is longer) or consumed grapefruit juice, grapefruit, Seville oranges, or St. John's Wort or products containing these within 30 days prior to receiving the first dose of study drug.

## 8.3. Subject Withdrawal Criteria

If there is an adverse event or medical reason for the withdrawal, the subject should be followed medically until the condition has either resolved or is stable. Details of the reason for withdrawal should be recorded in the subject's eCRF.

Subjects who withdraw should, if possible, have a follow-up examination, including a physical examination, the appropriate investigations, vital signs, and clinical laboratory tests (including pregnancy tests), as outlined for the Day 15 visit (Table 2 and Table 3). All details of this follow-up examination should be recorded in the subject's medical source documents.

## 8.3.1. Study Drug Withdrawal

Participation in the study is strictly voluntary. Subjects are free to discontinue the study at any time without giving their reason(s).

A subject must be withdrawn from the study treatment in the event of any of the following:

- Withdrawal of the subject's consent;
- New onset of a condition that would have met exclusion criterion, is clinically relevant and affects the subject's safety, and discontinuation is considered necessary by the Investigators and/Sponsor;
- Occurrence of intolerable adverse events;
- Occurrence of pregnancy;
- Intake of nonpermitted concomitant medication;
- Subject noncompliance;
- Significant protocol deviation determined in consultation with the Medical Monitor.

If a subject failed to attend scheduled assessments during the course of the study, the Investigators must determine the reasons and the circumstances as completely and accurately as possible and document this in the subject's source documents.

Subjects may be withdrawn from the study if there is concern for the subject's safety or it is determined that the subject is no longer a qualified participant. Subjects who withdraw should, if possible, have a follow-up examination, including a physical examination, the appropriate investigations, vital signs, and clinical laboratory tests (including pregnancy tests), as outlined for the Day 15 visit (Table 2 and Table 3). All details of this follow-up examination should be recorded in the subject's medical source documents.

Subjects who withdraw or are withdrawn from the study will be replaced only if they withdraw prior to dosing. Subjects who are withdrawn from the study, fail to return or are no longer qualified will not be replaced.

## **8.3.2.** Criteria for Study Termination

Sage Therapeutics may terminate this study or any portion of the study at any time for safety reasons, including the occurrence of adverse events or other findings suggesting unacceptable risk to subjects, or for administrative reasons. In the event of study termination, Sage Therapeutics will provide written notification to the Investigator. Investigational sites must promptly notify their Institutional Review Board (IRB) and initiate withdrawal procedures for participating subjects.

## 9. TREATMENT OF SUBJECTS

## 9.1. Number of Subjects

Approximately ten subjects with MDD will be enrolled into Part A of the study. Up to 52 subjects may be randomized in Part B to ensure at least 46 evaluable subjects for Part B. Evaluable subjects are defined as those subjects receiving study drug with at least one post-baseline HAM-D assessment.

## 9.2. Treatment Assignment

Study drug will be administered with food in both the inpatient and outpatient treatment periods. Food intake will be standardized as specified by the Sponsor.

#### 9.2.1. Part A

Subjects participating in Part A of the study will take study drug (SAGE-217) in an open-label manner. Subjects will be administered a 30 mg dose of study drug at 8:00 PM ( $\pm 15$  minutes) with food for 14 days (Day 1 to Day 14) as tolerated.

## 9.2.2. Part B

Subjects participating in the randomized, double-blind, placebo-controlled portion of the study (Part B) will be randomly assigned to receive SAGE-217 Oral Solution 30 mg or matching placebo solution on a 1:1 basis according to a computer-generated randomization schedule; the randomization schedule will be stratified to allow for treatment balance within each use of antidepressant stratum.

Subjects, clinicians, and study team will be blinded to treatment allocation. The pharmacist, who will prepare the oral solutions according to the randomization schedule, and an unblinded Monitor, who will perform drug accountability during the study, will be unblinded.

## 9.3. Dose Adjustment Criteria

During the Treatment Period, subjects will be able to receive study drug as long as there are no dose-limiting safety/tolerability concerns.

In both Part A and Part B, subjects who experience moderate or severe adverse events that according to the clinical judgement of the Investigator are related to study drug while receiving the 30 mg dose of study drug will receive 20 mg for the remaining of the Treatment Period. Subjects who experience moderate or severe related adverse events while receiving the 20 mg dose of study drug may not be able to continue receiving study drug based on the evaluation and clinical judgment of the Investigator, and may be terminated from the study.

Dosing may also be modified based on tolerability as assessed with SSS scores. Any SSS score of  $\geq 6$  will be reassessed within 10 minutes. If a subject is receiving the 30 mg dose of study drug and has an SSS score of  $\geq 6$  that is confirmed on repeat assessment during normal waking hours, the dose will be decreased to 20 mg for the rest of the Treatment Period. If a subject is receiving the 20 mg dose of study drug and has an SSS score of  $\geq 6$  that is confirmed on repeat

assessment during normal waking hours, then study drug will be discontinued and the subject will be terminated from the study.

Part A may be terminated and Part B initiated if there is a clear signal of activity based on the HAM-D scores and/or other scales being assessed. The study may be terminated if there is clear lack of activity based on HAM-D scores during Part A. A Data Review Team will assess the HAM-D and other data on an ongoing basis during Part A.

## 9.4. Prior/Concomitant Medications

## 9.4.1. Prior/Concomitant Medications

Subjects will receive standard of care for adult patients diagnosed with moderate to severe MDD. Psychotropic medications, which must have been initiated at least 14 days prior to screening, must remain at a stable dose until completion of the Day 15 assessments (Parts A and B).

Eligible subjects will be stratified based on use of antidepressant treatment (current/stable or not treated/withdrawn ≥30 days) and randomly assigned within each stratum in a 1:1 ratio to receive SAGE-217 Oral Solution or taste-matched placebo.

In this study, psychotropic medications refer to central nervous system active medications taken to help depressive symptoms, and include antidepressants, benzodiazepines, and hypnotic agents. Subjects presenting to the study on antidepressants may be eligible to participate if they have been on a stable dose for at least 14 days. Those subjects on benzodiazepines and hypnotic agents may be considered for eligibility based on specific discussions between the Investigator and the Sponsor to ensure safety. Subjects on other psychotropic medications, including stimulants, antipsychotics, and mood stabilizers, are not eligible to participate in this study.

Any concomitant medication determined necessary for the welfare of the subject may be given at the discretion of the Investigator at any time during the study under the guidance outlined in Section 9.4.2. In both Part A and Part B, all medications should be documented throughout the study from 30 days prior to signing the ICF through Day 28 (±3 days) and recorded on the eCRF. Prior medications (ie, those taken prior to signing of ICF) that required washout for study entry will also be documented.

#### 9.4.2. Restricted Medications

Restrictions on specific classes of medications include the following:

- Initiation of new antidepressant therapy is prohibited upon admission to the study center for those eligible subjects who desire study participation. Those subjects already taking an antidepressant at the time of study entry (and meeting all study inclusion criteria) will be permitted to remain on the pre-existing antidepressant at their current dose if they were on this medication for at least 14 days prior to study enrollment.
- Benzodiazepines are to be avoided as much as possible. Eligible subjects taking a stable dose of benzodiazepine for at least 14 days prior to the study will be discussed on a case-by-case basis with the Sponsor to determine eligibility. Subjects may be permitted to continue to take their current dose of the benzodiazepine (to prevent

acute withdrawal), but no new benzodiazepine use will be permitted during the course of the study.

- The use of hypnotics for sleep/insomnia such as Ambien® and trazodone is to be avoided; use of hypnotics will be discussed on a case-by-case basis with the Sponsor.
- Anticonvulsants and atypical antipsychotics are prohibited.

## 9.5. Treatment Compliance

Investigational product will be prepared by the site pharmacist. The Investigator(s) or designee will record the time and dose of study drug administration in the source documents. Any reasons for noncompliance will also be documented, including:

- Missed visits;
- Interruptions in the schedule of administration; and
- Nonpermitted medications.

The time at which study procedures are conducted should follow the protocol timelines as closely as possible.

## 10. STUDY DRUG MATERIALS AND MANAGEMENT

## 10.1. Study Drug

SAGE-217 Oral Solution is available as a 6 mg/mL stock aqueous solution of SAGE-217 Drug Substance containing 40% HPβCD and 0.0025% sucralose, which is further diluted with Sterile Water for Injection to achieve the selected dose. The 6 mg/mL stock SAGE-217 Oral Solution will be compounded from SAGE-217 Drug Substance Powder in the Bottle and Excipient (s) in the Bottle (manufactured under current Good Manufacturing Practice [GMP] conditions and further admixed at the clinical site in preparation for dosing.

A matching placebo oral solution will be prepared for administration without the active ingredient, but including the HP $\beta$ CD and sucralose, as well as three taste-masking components to preserve the blinding. Detailed instructions for study drug (SAGE-217 Oral Solution 30 mg and matching placebo) preparation will be provided in the Pharmacy Manual.

## 10.2. Batch Formula for Stock SAGE-217 Oral Solution 6 mg/mL

Each bottle of SAGE-217 Oral Solution 6 mg/mL will be compounded at the clinical pharmacy from components manufactured and supplied by the Sponsor per the directions provided in the Pharmacy Manual. The batch formula for a 125 mL solution of the 6 mg/mL stock solution is shown in Table 5.

Table 5: Batch Formula for 125 mL of Stock SAGE-217 Oral Solution 6 mg/mL

| Ingredient | <b>Compendia Specification</b> | Concentration (mg/mL) | Amount (mg/Bottle) |
|---|---|---|---|
| SAGE-217 | not applicable | 6 | 750 |
| НРВСО | USP/EP | 457 | 57,100 |
| Sucralose | USP/NF | 0.025 | 3.124 |
| Water for Injection | USP | not applicable | 85,650 |

Abbreviations: EP = European Pharmacopeia; HPβCD = hydroxypropyl-β-cyclodextrin; NF = National Formulary; USP = United States Pharmacopeia

Additional excipients will be utilized in matching placebo to match the taste of SAGE-217 Oral Solution. They include sucrose octaacetate, tannic acid, and ammonium glycyrrhizate. The quantities of these excipients will vary depending on the dose of SAGE-217 to match the taste of each individual dose.

## 10.3. Study Drug Packaging and Labeling

The composition and pharmaceutical quality of the investigational product will be maintained according to the current GMP and Good Clinical Practice (GCP) guidelines and available for review in the study medication documentation. Study drug will be provided to the site as powder in the bottle and excipient(s) in the bottle units to be compounded in the pharmacy at a volume of 125 mL of a 6 mg/mL stock solution and then further diluted to approximately 40 mL at the identified doses. The taste-matching excipients will be provided to the clinical pharmacies via suitable suppliers or can be ordered directly by the clinical pharmacies. Study drug labels with
all required information and conforming to all applicable Code of Federal Regulations and GMP/GCP guidelines will be prepared by the clinical research organization.

#### 10.4. Study Drug Storage

Upon receipt of study drug, the Investigator or designee will inspect the materials and complete and return the acknowledgment of receipt form enclosed with the parcel. A copy of the signed receipt will be kept in the study files.

The study drug materials must be carefully stored at the temperature specified in the Pharmacy Manual (eg, clinical dosing solutions stored at approximately 2 to 8°C for 11 days with room temperature excursions allowed for up to 24 hours after preparation), safely and separately from other drugs. The study drug may not be used for any purpose other than the present study. After the study is completed, all unused study drug must be retained, returned as directed, or destroyed on site per the Sponsor's instructions.

The Investigator or designee will be responsible for ensuring appropriate storage, compounding, dispensing, inventory, and accountability of all clinical supplies. An accurate, timely record of the disposition of all clinical supplies must be maintained. The supplies and inventory must be available for inspection by the designated representatives of the Sponsor or the Sponsor's representatives on request, and must include the information below:

- The identification of the subject to whom the drug was dispensed;
- The date(s) and quantity of the drug dispensed to the subject; and
- The product lot/batch number.

The preparation of the study drugs must be documented on a 'Drug Preparation and Dispensing Log Form' or similar form.

The drug inventory and any clinical supplies that have been destroyed must be documented. This documentation must include at least the information below or as agreed with the Sponsor:

- The number of prepared units;
- The number of administered units;
- The number of unused units;
- The number of units destroyed at the end of the study;
- The date, method, and location of destruction.

# 10.5. Administration and Study Drug Accountability

Doses will be prepared as an approximate 40 mL oral solution to be swallowed all at once, followed by approximately 200 mL of water that has been used to rinse the dosing bottle. The start time of swallowing the approximately 40 mL oral solution is time zero for all assessments. Subjects may have assistance from the clinic staff when taking the study drug.

#### 10.5.1. Study Drug Administration

While confined in the clinical unit (at least Day 1 through Day 7 of Part A and Part B), subjects will receive study drug at 8:00 PM (±15 minutes) with food.

Food intake will be standardized as specified by the Sponsor. Subjects who experience moderate or severe related adverse events while receiving study drug may not be able to continue receiving study drug based on the evaluation and clinical judgment of the Investigator, and may be terminated from the study.

Subjects may be discharged after a minimum 7-day inpatient stay, following completion of the Day 7 assessments. If their clinical condition does not allow discharge, the Investigator may keep the subjects as inpatients for a longer period of time.

For non-confinement days (Days 8 through 14 of Parts A and B), dosing will be done at the clinical site or, if suitable arrangements can be made, via home administration where local regulations allow. Home administration of study drug will be performed according to a site-specific plan by a healthcare professional trained on the protocol and delivery of the study drug.

#### 10.5.2. Study Drug Accountability

The study drug provided is for use only as directed in this protocol.

The Investigator or designee must maintain a record of all study drug received, used, and discarded. It must be clear from the records which subject received which dose of active or matching placebo treatment.

The Sponsor will be permitted access to the study supplies at any time within usual business hours and with appropriate notice during or after completion of the study to perform drug accountability reconciliation. Only unblinded personnel will be able to access the study drug and accountability documentation from first dosing through database hard lock.

#### 10.6. Study Drug Handling and Disposal

The pharmacist or designee for drug accountability is to document the date and time of initial compounding, subsequent admixture of dosing solutions, administration of test article, and for which subject the study drug was intended (ie, record subject initials and birth date or other unique identifier).

At the end of the study, any unused study drug will be retained or returned to the Sponsor for destruction or destroyed locally per the Sponsor's directions. The disposition of study drug will be documented.

#### 11. ASSESSMENT OF EFFICACY

#### 11.1. Hamilton Rating Scale for Depression (HAM-D)

The primary outcome measure in Part B will be the change from baseline in 17-item HAM-D total score at the end of the Treatment Period (Day 15). The HAM-D will be administered before, during, and after the administration of open-label (Part A) and blinded (Part B) study drug.

The 17-item HAM-D will be used to rate the severity of depression in subjects who are already diagnosed as depressed (Hamilton 1960). The 17-item HAM-D comprises individual ratings related to the following symptoms: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. The HAM-D assessments are to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28. Every effort should be made for the same rater to perform all HAM-D assessments for an individual subject.

The HAM-D total score will be calculated as the sum of the 17 individual item scores. Item 16 can be rated according to history (item 16A) or actual weight change (item 16B). The item 16 score is calculated as the item 16 response that is not equal to 3 (ie, "Not assessed").

In addition to the primary efficacy endpoint of change from baseline in HAM-D total score (Part B), several secondary efficacy endpoints will be derived for the HAM-D. Hamilton Rating Scale for Depression subscale scores will be calculated as the sum of the items comprising each subscale. Hamilton Rating Scale for Depression response will be defined as having a 50% or greater reduction from baseline in HAM-D total score. Hamilton Rating Scale for Depression remission will be defined as having a HAM-D total score of ≤7. A copy of the HAM-D is provided in Appendix 1.

## 11.2. Montgomery-Åsberg Depression Rating Scale (MADRS)

The MADRS is a 10-item diagnostic questionnaire that psychiatrists use to measure the severity of depressive episodes in subjects with mood disorders. It was designed as an adjunct to the HAM-D that would be more sensitive to the changes brought on by antidepressants and other forms of treatment than the Hamilton Scale.

The MADRS assessments are to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28.

Higher MADRS scores indicate more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60 (McDowell 2006; Müller-Thomsen 2005).

The questionnaire includes questions on the following symptoms:

- 1. Apparent sadness
- 2. Reported sadness

- 3. Inner tension
- 4. Reduced sleep
- 5. Reduced appetite
- 6. Concentration difficulties
- 7. Lassitude
- 8. Inability to feel
- 9. Pessimistic thoughts
- 10. Suicidal thoughts

The MADRS total score will be calculated as the sum of the 10 individual item scores. A copy of the MADRS is provided in Appendix 2.

### 11.3. Hamilton Anxiety Rating Scale (HAM-A)

The 14-item HAM-A will be used to rate the severity of symptoms of anxiety (Hamilton 1959). Each of the 14 items is defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scoring for HAM-A is calculated by assigning scores of 0 (not present) to 4 (very severe), with a total score range of 0 to 56, where <17 indicates mild severity, 18 to 24 mild to moderate severity, and 25 to 30 moderate to severe severity.

The HAM-A assessments are to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28. Every effort should be made for the same rater to perform all HAM-A assessments for an individual subject.

The HAM-A total score will be calculated as the sum of the 14 individual item scores. A copy of the HAM-A is provided in Appendix 3.

## 11.4. Clinical Global Impression (CGI)

The CGI is a validated measure often utilized in clinical trials to allow clinicians to integrate several sources of information into a single rating of the subject's condition. The CGI scale consists of 3 items. Only the first 2 items are being used in this study.

The Clinical Global Impression - Severity (CGI-S) uses a 7-point Likert scale to rate the severity of the subject's illness at the time of assessment, relative to the clinician's past experience with subjects who have the same diagnosis. Considering total clinical experience, a subject is assessed on severity of mental illness at the time of rating as 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=extremely ill. The CGI-S assessments are to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28.

The CGI-I employs a 7-point Likert scale to measure the overall improvement in the subject's condition posttreatment. The Investigator will rate the subject's total improvement whether or not it is due entirely to drug treatment. Response choices include: 0=not assessed, 1=very much

improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse. The CGI-I is only rated at posttreatment assessments. By definition, all CGI-I assessments are evaluated against baseline conditions. CGI-I response will be defined as having a CGI-I score of "very much improved" or "much improved." The CGI-I assessments are to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28. A copy of the CGI is provided in Appendix 4.

## 11.5. Short Form-36 (SF-36)

The SF-36® Health Survey is a subject-reported 36-item instrument for measuring functional health and well-being in eight dimensions (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health) (Ware 2007). Scores are provided for each of the eight dimensions and are totaled into a Physical Component Summary and a Mental Component Summary. Higher SF-36 scores indicate a better state of health. The SF-36 requires approximately 10 minutes to complete, and can be self-administered or completed by interview in person or by telephone. In Part B, the SF-36 assessments are to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28.

A copy of the SF-36 is provided in Appendix 5.

# 11.6. The Fatigue Associated With Depression (FAs-D) Patient-Reported Outcome (PRO)

Fatigue is one of the most common symptoms of MDD. The Fatigue Associated with Depression Questionnaire (FAs-D) was developed to assess fatigue and its impact in patients with MDD. The 13-item patient-reported questionnaire was designed to assess fatigue associated with depression in the past week. Three scores are computed: a six-item fatigue experience subscale (fatigued, tired, exhausted, lack of energy, physically weak, and feeling like everything requires too much effort), a seven-item fatigue impact subscale (impact on household chores; family relationships; enjoyable activities; social activities with friends; self-care; intimate relationships; and productivity at work or school), and a total score (all 13 items). Items 12 (impact on intimate relationships) and 13 (impact on productivity at work or school) are not applicable to all subjects, so these items are not answered in some cases. The fatigue experience items are rated on a five-point scale with response options of "never," "rarely," "sometimes," "often," and "always." The impact items are rated on a five-point scale with response options of "not at all," "a little," "somewhat," "quite a bit," and "very much." The two subscales and the total score are computed as the mean of all answered items within each scale, and each scale score has a possible range of 1 to 5, with higher scores representing greater fatigue. In Part B, the FAs-D assessments are to be completed at 8:00 AM (±30 minutes) at each scheduled time point during the Treatment Period, and in the morning on Day 15, Day 21, and Day 28.

A copy of the FAs-D is provided in Appendix 6.

#### 12. PHARMACOKINETICS

#### **12.1.** Blood Sample Collection

Plasma samples for PK analysis in Part A and Part B will be collected predose and 0.25, 0.5, 1, 2, 10, and 12 hours postdose on Day 7 (within  $\pm 5$  minutes of the scheduled time point through 0.5 hours after dosing and  $\pm 15$  minutes of the scheduled time point from 1 hour after dosing and greater), prior to discharge on Day 8 for subjects being discharged or 16 hours postdose for subjects remaining as inpatients, predose on Day 14, and in the morning on Day 15. The time of study drug administration is time zero and all post-dosing sampling times are relative to this time. The Investigator or designee will arrange to have the plasma samples processed, stored, and transported as directed for bioanalysis.

In the event of a dose adjustment, an unscheduled PK sample should be collected just prior to the dose change. An additional PK sample may be collected at any time if clinically indicated and at the discretion of the Investigator (eg, for unusual or severe adverse events).

Each sample will be marked with unique identifiers such as the study number, subject number, and the nominal sample time. The date and actual time that the blood sample was taken will be recorded on the CRF or electronically with a bar code or other method.

#### 12.2. Storage and Shipment of Pharmacokinetic Samples

The plasma samples should be kept frozen at approximately -70 to -80°C until analyzed. They should be packed as directed to avoid breakage during transit and with sufficient dry ice to prevent thawing for at least 72 hours. A specimen-identification form must be completed and sent to the laboratory with each set of samples. The clinical site will arrange to have the plasma samples transported as directed for bioanalysis as detailed in the PK instructions.

# 12.3. Sample Analysis

Bioanalysis of plasma samples for the determination of SAGE-217 will be performed utilizing a validated liquid chromatography-tandem mass spectrometry method at a qualified laboratory.

#### 13. ASSESSMENT OF SAFETY

#### 13.1. Safety Parameters

Safety and tolerability of study drug will be evaluated in Parts A and B by vital signs measurements, clinical laboratory measures, physical examination, ECGs, concomitant medication usage, C-SSRS, SSS, and adverse event reporting.

#### 13.1.1. Demographic/Medical History

Age, race, and ethnic origin will be recorded at the Screening visit. The diagnosis of MDD will be determined using the SCID-I.

#### 13.1.2. Vital Signs

Vital signs include respiratory rate, oral temperature, and supine (for at least 5 minutes prior to the measurement) and standing systolic and diastolic blood pressure and heart rate. Vital signs will be obtained within  $\pm 5$  minutes of the scheduled time point through 0.5 hours after dosing and  $\pm 30$  minutes of the scheduled time point from 1 hour after dosing and greater, unless the subject is asleep between the hours of 23:00 h and 06:00 h.

From Day 1 through Day 7, vital signs and pulse oximetry will be performed at screening (vital signs only) and at the following time points: predose, 0.25, 0.5, 1, 2, and 12 hours after dosing. During the outpatient treatment period, vital signs will be completed prior to dosing and 1 hour after dosing. Vital signs may be repeated at the discretion of the Investigator or Visiting Home Healthcare Provider as clinically indicated.

#### 13.1.3. Weight and Height

Body weight and height will be measured at the Screening visit; weight will also be measured on in the morning on Day 15, and during the follow-up visits on Days 21 and 28.

#### 13.1.4. Physical Examination

A physical examination of all major body systems will be undertaken and recorded at the Screening visit, Day 8, Day 15, and Day 21, with a brief physical examination on Day 28.

#### 13.1.5. Electrocardiogram (ECG)

A 12-lead ECG will be assessed at the Screening visit and 1 hour  $\pm 15$  minutes after dosing on Days 1, 2, 7, and 14 and during the follow-up visit on Day 21. All time points are relative to the time of dosing. The standard intervals as well as any abnormalities will be recorded.

#### 13.1.6. Laboratory Assessments

Blood and urine samples will be collected for hematology, serum chemistry, coagulation, select hormone parameters, and urinalysis at the Screening visit, and in the morning on Days 8 and 15 and during the follow-up visits on Days 21 and 28. Where consent is given, an optional blood sample for hormone and exploratory biochemistry testing and optional genetic sample for biomarker testing will be collected at the Screening visit.

Serum and urine samples for pregnancy tests will also be collected. These assessments should be performed as outlined below.

All samples will be analyzed at the central laboratory. Subjects may be considered eligible for the study based on local laboratory results; however, screening samples must also be sent to the central laboratory.

All clinical laboratory test results outside the reference range will be interpreted by the Investigator as abnormal, not clinically significant (NCS) or abnormal, clinically significant (CS). Screening results considered abnormal, CS recorded at the Screening visit may make the subject ineligible for the study pending review by the Medical Monitor. Clinical laboratory results that are abnormal, CS during the study but within normal range at baseline and/or indicate a worsening from baseline will be considered adverse events, assessed according to Section 13.2.1, and recorded in the eCRF.

#### **13.1.6.1.** Hematology

Hematology tests will include complete blood count, including red blood cells, white blood cells with differentiation, hemoglobin, hematocrit, reticulocytes, and platelets. The coagulation panel will include activated partial thromboplastin time, prothrombin time, and international normalized ratio.

#### 13.1.6.2. Blood Chemistry

Serum chemistry tests will include serum electrolytes; renal function tests, including creatinine, blood urea nitrogen, bicarbonate or total carbon dioxide; liver function tests, including total bilirubin, aspartate aminotransferase, and alanine aminotransferase; total protein; and albumin.

#### **13.1.6.3.** Urinalysis

Urinalysis will include assessment of protein, blood, glucose, ketones, bile, urobilinogen, hemoglobin, leukocyte esterase, nitrites, color, turbidity, pH, and specific gravity.

#### 13.1.6.4. Hormones and Exploratory Biochemistry

Optional blood samples will be collected and may be analyzed for stress hormone levels, kynurenine biochemistry, and markers of inflammation. Future research may suggest other biochemical pathways as candidates for influencing not only response to SAGE-217 but also susceptibility to disorders for which SAGE-217 may be evaluated. Thus, the exploratory biochemistry may involve study of additional unnamed molecular pathways, but only as related to disease susceptibility and drug action.

#### **13.1.6.5. Virus Serology**

Subjects will be screened for hepatitis (HBsAg and anti-HCV) and HIV prior to being enrolled in the study.

#### 13.1.6.6. Pregnancy Test

Females of childbearing potential will be tested for pregnancy by serum pregnancy test at the Screening visit and by urine pregnancy test on Day 1 (predose) and at the follow-up visit on

Day 28. In addition, female subjects who prematurely discontinue before Day 28 will have a pregnancy test performed at the early termination visit.

#### 13.1.6.7. Genetic Testing

Where consent is given, an optional genetic sample for biomarker testing will be collected at the Screening visit.

The objective of this research is to collect and store blood samples for possible DNA extraction and exploratory research into how genes or specific genetic variation may influence response (ie, distribution, safety, tolerability, and efficacy) to SAGE-217. Specific genetic variations of interest include but are not limited to: classes of metabolizing enzymes (eg, cytochrome P450 supra-family genes), genes encoding enzymes involved in the production and metabolism of SAGE-217 (eg, AKR1C4 [ $3\alpha$ -hydroxysteroid dehydrogenase]), genes associated with the  $\gamma$ -aminobutyric acid (GABA) receptor (eg, GABRA1-A6, GABRB1-B3, GABRD, GABRE, GABRG1-3), and genes associated with the production and degradation of GABA.

Future research may suggest other genes or gene categories as candidates for influencing not only response to SAGE-217 but also susceptibility to disorders for which SAGE-217 may be evaluated. Thus, the genetic research may involve study of additional unnamed genes or gene categories, but only as related to disease susceptibility and drug action.

#### 13.1.6.8. Drugs of Abuse and Alcohol

A urine sample for assessment of selected drugs of abuse (including amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates, phencyclidine, and propoxyphene) and a serum or breath sample for alcohol screen will be collected at screening and predose on Day 1. Use of benzodiazepines at screening is not necessarily exclusionary, as subjects will be allowed to take psychotropics that have been initiated at least 14 days prior to admission to the study center at a stable dose following discussion with the Sponsor (see Section 9.3).

#### 13.1.7. Columbia-Suicide Severity Rating Scale (C-SSRS)

Suicidality will be monitored during the study using the C-SSRS (Posner 2011). This scale consists of a baseline evaluation that assesses the lifetime experience of the subject with suicidal ideation and behavior, and a post-baseline evaluation that focuses on suicidality since the last study visit. The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe).

If, in the opinion of the Investigator, the subject is showing clinically meaningful changes in suicidality, no further study drug will be administered and the subject will be referred to a psychologist or psychiatrist for further evaluation. This information will be tracked.

The "Baseline/Screening" C-SSRS form will be completed at screening (lifetime history and past 24 months). The "Since Last Visit" C-SSRS form will be completed at any time of day at all subsequent time points, as outlined in Table 2 and Table 3. The C-SSRS is provided in Appendix 5.

#### 13.1.8. Stanford Sleepiness Scale (SSS)

The SSS is subject-rated scale designed to quickly assess how alert a subject is feeling. Degrees of sleepiness and alertness are rated on a scale of 1 to 7, where the lowest score of '1' indicates the subject is 'feeling active, vital, alert, or wide awake' and the highest score of '7' indicates the subject is 'no longer fighting sleep, sleep onset soon; having dream-like thoughts'.

In both Part A and Part B, from Day 1 through Day 7, SSS will be completed at the following time points: predose, 0.25, 0.5, 1, and 2 after dosing. The scale is to be completed within  $\pm 5$  minutes of the scheduled time point through 0.5 hours after dosing and  $\pm 15$  minutes of the scheduled time point from 1 hour after dosing and greater, unless the subject is asleep between 23:00 h and 06:00 h during the inpatient treatment period. During the outpatient treatment period, SSS will be completed prior to dosing and 1 hour after dosing. All time points are relative to the time of dosing. The SSS is provided in Appendix 8.

#### 13.2. Adverse and Serious Adverse Events

#### **13.2.1.** Definition of Adverse Events

#### **13.2.1.1.** Adverse Event

An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. In clinical studies, an adverse event can include an undesirable medical condition occurring at any time, including baseline or washout periods, even if no study treatment has been administered.

#### 13.2.1.2. Suspected Adverse Reaction

A suspected adverse reaction is any adverse event for which there is a reasonable possibility that the drug caused the adverse event. For the purposes of Investigational New Drug safety reporting, "reasonable possibility" means there is evidence to suggest a causal relationship between the drug and the adverse event. Suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any adverse event caused by a drug.

#### 13.2.1.3. Serious Adverse Event

A serious adverse event is an adverse event occurring during any study phase and at any dose of the investigational product, comparator or placebo, that fulfils one or more of the following:

- It results in death
- It is immediately life-threatening
- It requires inpatient hospitalization or prolongation of existing hospitalization
- It results in persistent or significant disability or incapacity
- It results in a congenital abnormality or birth defect
- It is an important medical event that may jeopardize the subject or may require medical intervention to prevent one of the outcomes listed above.

All serious adverse events that occur after any subject has been enrolled, whether or not they are related to the study, must be recorded for the duration of the study on forms provided by Sage Therapeutics or designee.

# 13.3. Relationship to Study Drug

An Investigator who is qualified in medicine must make the determination of relationship to the investigational product for each adverse event (unrelated, possibly related or probably related). The Investigator should decide whether, in his or her medical judgment, there is a reasonable possibility that the event may have been caused by the investigational product. If no valid reason exists for suggesting a relationship, then the adverse event should be classified as "unrelated." If there is any valid reason, even if undetermined, for suspecting a possible cause-and-effect relationship between the investigational product and the occurrence of the adverse event, then the adverse event should be considered "related."

| Not Related: | No relationship between the experience and the administration of study drug; related to other |
|---|---|
| | etiologies such as concomitant medications or subject's clinical state. |
| Possibly | A reaction that follows a plausible temporal sequence from administration of the study drug and |
| Related: | follows a known response pattern to the suspected study drug. |
| | The reaction might have been produced by the subject's clinical state or other modes of therapy |
| | administered to the subject, but this is not known for sure. |
| Probably | A reaction that follows a plausible temporal sequence from administration of the study drug and |
| Related: | follows a known response pattern to the suspected study drug. |
| | The reaction cannot be reasonably explained by the known characteristics of the subject's clinical |
| | state or other modes of therapy administered to the subject. |

If the relationship between the adverse event/serious adverse event and the investigational product is determined to be "possible" or "probable", the event will be considered to be related to the investigational product for the purposes of expedited regulatory reporting.

## 13.4. Recording Adverse Events

Adverse events spontaneously reported by the subject and/or in response to an open question from the study personnel or revealed by observation will be recorded during the study at the investigational site. Clinically significant changes in laboratory values, blood pressure, and pulse need not be reported as adverse events unless they prompt corrective medical action by the Investigator, constitute a serious adverse event, or lead to discontinuation of administration of study drug.

Information about adverse events will be collected from the signing of the ICF until the final visit of the study for that subject. Adverse events that occur after the first administration of study drug will be denoted TEAEs.

All adverse events will be followed until they are resolved or have reached a clinical plateau with no expectation of future change.

The adverse event term should be reported in standard medical terminology when possible. For each adverse event, the Investigator will evaluate and report the onset (date and time), resolution or clinical plateau (date and time), severity, causality, action taken, outcome, and whether or not it caused the subject to discontinue the study.

Severity will be assessed according to the following scale:

- Mild (awareness of sign or symptom, but easily tolerated)
- Moderate (discomfort sufficient to cause interference with normal activities)
- Severe (incapacitating, with inability to perform normal activities)

#### 13.5. Reporting Adverse Events

All serious adverse events (regardless of causality) will be recorded from the signing of the ICF until the Day 28 follow-up visit. Any serious adverse events considered possibly or probably related to the investigational product and discovered by the Investigator at any time after the study should be reported. All serious adverse events must be reported to the Sponsor or Sponsor's designee immediately by phone and in writing within 24 hours of the first awareness of the event. The Investigator must complete, sign and date the serious adverse event pages, verify the accuracy of the information recorded on the serious adverse event pages with the corresponding source documents, and send a copy to Sage Therapeutics or designee.

Additional follow-up information, if required or available, should be sent to Sage Therapeutics or designee within 24 hours of receipt; a follow-up serious adverse event form should be completed and placed with the original serious adverse event information and kept with the appropriate section of the study file.

Sage Therapeutics or designee is responsible for notifying the relevant regulatory authorities of certain events. It is the Principal Investigator's responsibility to notify the IRB of all serious adverse events that occur at his or her site if applicable per the IRB's requirements. Investigators will also be notified of all unexpected, serious, drug-related events (7-/15-Day Safety Reports) that occur during the clinical study. Each site is responsible for notifying its IRB of these additional serious adverse events.

# 13.6. Emergency Identification of Study Drug

Part B of the study is double-blind. The pharmacist responsible for preparing the solutions will be unblinded and will retain an official paper copy of the randomization schedule. In addition, an unblinded Monitor will perform drug accountability during the study.

During the study, the blind is to be broken only when the safety of a subject is at risk and the treatment plan is dependent on the study treatment received. Unless a subject is at immediate risk, the Investigator must make diligent attempts to contact the Sponsor prior to unblinding the study treatment administered to a subject. Any request from the Investigator about the treatment administered to study subjects must be discussed with the Sponsor. If the unblinding occurs without the Sponsor's knowledge, the Investigator must notify the Sponsor as soon as possible and no later than the next business morning. All circumstances surrounding a premature unblinding must be clearly documented in the source records. Unless a subject is at immediate risk, any request for the unblinding of individual subjects must be made in writing to the Sponsor and approved by the appropriate Sponsor personnel, according to standard operating procedures. The blinding of the study will be broken after the database has been locked. Electronic copies of the randomization code will be made available to the laboratory performing the bioanalytical analyses in order to allow for limited analysis of samples from subjects receiving matching placebo.

Protocol 217-MDD-201 Version 1.0 24 October 2016 Sage Therapeutics

In all cases where the study drug allocation for a subject is unblinded, pertinent information must be documented in the subject's records and on the eCRF. If the subject or study center personnel (other than pharmacist) have been unblinded, the subject will be terminated from the study.

#### 14. STATISTICS

#### 14.1. Data Analysis Sets

#### 14.1.1. Analysis Populations and Methods

The Safety Population (for both Part A and Part B), defined as all subjects administered study drug, will be used to provide descriptive summaries of safety data.

The Efficacy Population (for both Part A and Part B), defined as all subjects in the Safety Population who complete at least 1 day of dosing of study drug and have at least one post-baseline efficacy evaluation, will be used to analyze efficacy data.

The PK Population will consist of all subjects in the Safety Population with sufficient plasma concentrations for PK evaluations, and will be used to summarize PK data.

#### 14.2. Handling of Missing Data

Every attempt will be made to avoid missing data. All subjects will be used in the analyses, as per the analysis populations, using all non-missing data available. No imputation process will be used to estimate missing data. A sensitivity analysis will be used to investigate the impact of missing data if  $\geq$ 5% of subjects have missing data.

#### 14.3. General Considerations

For the purpose of all safety and efficacy analyses where applicable, baseline is defined as the last measurement prior to the start of study drug administration.

Continuous endpoints will be summarized with n, mean, standard deviation (SD), median, minimum and maximum. In addition, change from baseline values will be calculated at each time point and summarized descriptively. For categorical endpoints, descriptive summaries will include counts and percentages.

# 14.4. Demographics and Baseline Characteristics

Demographic data, such as age, race, and ethnicity, and baseline characteristics, such as height, weight, and body mass index (BMI), will be summarized using the Safety Population.

Hepatitis, HIV, drug and alcohol, and pregnancy screening results will be listed, but not summarized as they are considered part of the inclusion/exclusion criteria.

Medical/family history will be listed by subject.

# 14.5. Efficacy Analyses

Efficacy data will be summarized using appropriate descriptive statistics and other data presentation methods where applicable; subject listings will be provided for all efficacy data. For (the open-label) Part A, efficacy data will be summarized descriptively. For Part B, subjects will be analyzed according to randomized treatment.

An analysis of ten subjects completing Part A is planned to inform Part B study conduct.

For Part B of the study, change from baseline to each assessment in HAM-D total score will be analyzed using a mixed effects model for repeated measures (MMRM); the model will include center, treatment, baseline HAM-D total score, antidepressant use strata, assessment time point, and time point-by-treatment as explanatory variables. Center will be treated as a random effect while all other explanatory variables will be treated as fixed effects. All post-baseline time points will be included in the model. The main comparison will be between SAGE-217 Oral Solution and matching placebo at the 15-day time point. Model-based point estimates (ie, least squares [LS] means), 95% confidence intervals, and p-values) will be reported where applicable. An unstructured covariance structure will be used to model the within-subject errors. Compound symmetry covariance structure will be used if there is a convergence issue with the unstructured covariance model.

Descriptive statistics for HAM-D total score and change from baseline values will be presented by assessment time point for Part A. Summaries will include n, mean, SD, median, minimum, and maximum.

Similar to those methods described above for Part B, an MMRM will be used for the analysis of the following variables: changes from baseline in MADRS total score and HAM-A total score, and select individual item and subscale scores. For each model, the comparison of interest will be between SAGE-217 Oral Solution and matching placebo at the 15-day time point. Model-based point estimates (ie, LS means), 95% confidence intervals, and p-values will be reported.

Logistic regression methods will be used for the analysis of the following binary variables: HAM-D response (defined as ≥50% reduction from baseline in HAM-D total score), HAM-D remission (defined as HAM-D total score of ≤7.0), and CGI-I response. Logistic regression models will include terms for center, treatment, antidepressant use strata, and baseline score. The comparison of interest will be the difference between SAGE-217 Oral Solution and matching placebo at the 15-day time point in Part B. Model-based point estimates (ie, odds ratios), 95% confidence intervals, and p-values will be reported. For the CGI-I response analysis, baseline CGI-S score will be included in the model.

For all scores, descriptive statistics, change from baseline values, and response variables will be presented by treatment and assessment time point. Summaries will include n, mean, SD, median, minimum, and maximum.

Similar to the main comparison of HAM-D total score in Part B, descriptive summary statistics will be provided and an MMRM model will be used to analyze the change from baseline in SF-36 and FAs-D.

# 14.6. Safety Analyses

Safety and tolerability of study drug will be evaluated by adverse events, concomitant medication usage, changes from baseline in physical examination, vital signs, clinical laboratory evaluations, and 12-lead ECG. Suicidality will be monitored by the C-SSRS. Sedation will be assessed using the SSS. Safety data will be listed by subject and summarized by treatment group. All safety summaries will be performed on the Safety Population.

#### 14.6.1. Adverse Events

The analysis of adverse events will be based on the concept of TEAEs. A TEAE is defined as an adverse event with onset after the start of study drug, or any worsening of a pre-existing medical condition/adverse event with onset after the start of study drug and until 7 days after the last dose. The incidence of TEAEs will be summarized overall and by Medical Dictionary for Regulatory Activities (MedDRA) Version 18.1 or higher System Organ Class (SOC) and preferred term. Incidences will be presented in order of decreasing frequency for the SAGE-217 Oral Solution treatment group. In addition, summaries will be provided by severity (mild, moderate, severe) and by causality (related, not related) to study drug (see Section 13.3).

Treatment-emergent adverse events leading to discontinuation and serious adverse events (see Section 13.2.1.3 for definition) with onset after the start of randomized study drug will also be summarized.

All adverse events and serious adverse events (including those with onset or worsening before the start of study drug) through the Day 28 follow-up visit will be listed.

#### 14.6.2. Clinical Laboratory Evaluations

Clinical laboratory results will be listed by subject and timing of collection. Mean changes from baseline in clinical laboratory measures will be summarized.

#### 14.6.3. Physical Examinations

Physical examinations in Parts A and B will be summarized at the Screening visit, Day 8, Day 15, Day 21, and Day 28 visits. Any clinically significant change in physical examination compared to those observed at screening should be noted as an adverse event.

#### **14.6.4.** Vital Signs

Vital sign results will be listed by subject and timing of collection. Mean changes from randomization in vital signs will be summarized by time point.

#### 14.6.5. 12-Lead Electrocardiogram

The following ECG parameters will be listed for each subject: heart rate, PR, QRS, QT, QTc, and QT interval calculated using the Fridericia method (QTcF). Any clinically significant abnormalities or changes in ECGs should be listed as an adverse event. Electrocardiogram findings will be listed by subject and visit.

#### 14.6.6. Prior and Concomitant Medications

Medications will be recorded at each study visit during the study and will be coded using World Health Organization-Drug dictionary (WHO-DD) September 2015, or later.

Medications will be presented according to whether they are being taken prior to and/or during the study (concomitant). Prior medications are defined as those taken during the 30 days prior to informed consent. Concomitant medications are defined as those with a start date on or after the first dose of study drug, or those with a start date before the first dose of study drug that are ongoing or with a stop date on or after the first dose of study drug. If medication dates are

incomplete and it is not clear whether the medication was concomitant, it will be assumed to be concomitant.

Details of prior and concomitant medications will be listed by subject, start date, and verbatim term.

#### 14.6.7. Columbia Suicide Severity Rating Scale

Suicidality data collected on the C-SSRS at baseline and by visit during the Treatment Period will be listed for all subjects. Listings will include behavior type and/or category for Suicidal Ideation and Suicidal Behavior of the C-SSRS.

#### 14.6.8. Stanford Sleepiness Scale

Sedation data collected on the SSS will be listed for all subjects. Changes in score over time will be represented graphically, and change from Day 1 will be measured.

#### 14.7. Pharmacokinetic Analyses

Pharmacokinetic parameters will be summarized using appropriate descriptive statistics. Time at maximum (peak) plasma concentration ( $t_{max}$ ) will be summarized using n, mean, SD, median, minimum, and maximum. All other PK parameters will be summarized using n, geometric mean, coefficient of variation, median, minimum, and maximum and listed by subject.

Plasma concentrations and PK parameters will be listed by subject.

In addition to typical descriptive statistics, summaries should include geometric mean, coefficient of variation, and geometric coefficient of variation.

# **14.8.** Determination of Sample Size

The sample size of ten subjects for Part A was selected based on clinical and not statistical considerations.

For Part B, assuming a two-sided t-test at an alpha level of 0.10, a sample size of 23 subjects per group would provide 80% power to detect an effect size of 0.75 between the SAGE-217 Oral Solution and matching placebo groups with regard to the secondary efficacy outcome variable of change from baseline in HAM-D total score. An effect size of 0.75 corresponds to a matching placebo-adjusted difference of 7.5 points in the change from baseline in HAM-D total score at 15 days with an assumed SD of 10 points. By including two treatment groups and using a 1:1 randomization, a total of 46 subjects are required. Assuming a non-evaluability rate of 10%, up to 52 subjects will be randomized.

# 14.9. Changes From Protocol Specified Analyses

Any changes from the analytical methods outlined in the protocol will be documented in the final statistical analysis plan.

#### 15. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

#### 15.1. Study Monitoring

Before an investigational site can enter a subject into the study, a representative of Sage Therapeutics or designee will visit the investigational study site to:

- Determine the adequacy of the facilities; and
- Discuss with the Investigator(s) and other personnel their responsibilities with regard to protocol adherence, and the responsibilities of Sage Therapeutics or designee or its representatives. This will be documented in a Clinical Study Agreement between Sage Therapeutics and the Investigator.

During the study, a monitor from Sage Therapeutics or designee will have regular contacts with the investigational site for the following:

- Provide information and support to the Investigator(s);
- Confirm that facilities remain acceptable;
- Confirm that the investigational team is adhering to the protocol, that data are being accurately recorded in the eCRFs, and that investigational product accountability checks are being performed;
- Perform source data verification. This includes a comparison of the data in the eCRFs with the subject's medical records at the hospital or practice, and other records relevant to the study. This will require direct access to all original records for each subject (eg, clinic charts);
- Record and report any protocol deviations not previously sent to Sage Therapeutics or designee; and
- Confirm adverse events and serious adverse events have been properly documented on eCRFs and confirm any serious adverse events have been forwarded to Sage Therapeutics or designee and those serious adverse events that met criteria for reporting have been forwarded to the IRB.

The monitor will be available between visits if the Investigator(s) or other staff needs information or advice.

# 15.2. Audits and Inspections

Authorized representatives of Sage Therapeutics, a regulatory authority, an Independent Ethics Committee (IEC) or an IRB may visit the site to perform audits or inspections, including source data verification. The purpose of a Sage Therapeutics or designee audit or inspection is to systematically and independently examine all study-related activities and documents to determine whether these activities were conducted, and data were recorded, analyzed, and accurately reported according to the protocol, GCP guidelines of the International Council for Harmonisation (ICH), and any applicable regulatory requirements. The Investigator should contact Sage Therapeutics immediately if contacted by a regulatory agency about an inspection.

# 15.3. Institutional Review Board (IRB)

The Principal Investigator must obtain IRB approval for the investigation. Initial IRB approval and all materials approved by the IRB for this study, including the subject consent form and recruitment materials, must be maintained by the Investigator and made available for inspection.

#### 16. QUALITY CONTROL AND QUALITY ASSURANCE

The Investigator and institution will permit study-related monitoring, audits, IRB review, and regulatory inspections as requested by the Food and Drug Administration, the Sponsor, or the Sponsor's designee, including direct access to source data/documents (ie, original medical records, laboratory reports, hospital documents, progress reports, signed ICFs) in addition to eCRFs.

Quality assurance and quality-control systems with written standard operating procedures will be followed to ensure this study will be conducted and data will be generated, documented (recorded), and reported in compliance with the protocol, GCP, and the applicable regulatory requirements.

The site's dedicated study monitor will arrange to visit the Investigator at regular intervals during the study. The monitoring visits must be conducted according to the applicable ICH and GCP guidelines to ensure protocol adherence, quality of data, drug accountability, compliance with regulatory requirements, and continued adequacy of the investigational site and its facilities.

During these visits, eCRFs and other data related to the study will be reviewed and any discrepancies or omissions will be identified and resolved. The study monitor will be given access to study-relevant source documents (including medical records) for purposes of source data verification.

During and/or after completion of the study, quality-assurance officers named by Sage Therapeutics or the regulatory authorities may wish to perform on-site audits. The Investigator is expected to cooperate with any audit and provide assistance and documentation (including source data) as requested.

Quality control will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly.

Agreements made by the Sponsor with the Investigator/institution and any other parties involved with the clinical study will be in writing in a separate agreement.

#### 17. ETHICS

#### 17.1. Ethics Review

The final study protocol, including the final version of the ICF, must be approved or given a favorable opinion in writing by an IRB or IEC as appropriate. The Investigator must submit written approval to Sage Therapeutics or designee before he or she can enroll any subject into the study.

The Principal Investigator is responsible for informing the IRB or IEC of any amendment to the protocol in accordance with local requirements. In addition, the IRB or IEC must approve all advertising used to recruit subjects for the study. The protocol must be re-approved by the IRB or IEC upon receipt of amendments and annually, as local regulations require.

The Principal Investigator is also responsible for providing the IRB with reports of any reportable serious adverse drug reactions from any other study conducted with the investigational product. Sage Therapeutics or designee will provide this information to the Principal Investigator.

Progress reports and notifications of serious adverse drug reactions will be provided to the IRB or IEC according to local regulations and guidelines.

#### 17.2. Ethical Conduct of the Study

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and its most recent amendment (2008) and are consistent with ICH/GCP and other applicable regulatory requirements.

#### 17.3. Written Informed Consent

The Principal Investigator will ensure that the subject is given full and adequate oral and written information about the nature, purpose, possible risk, and benefit of the study. Subjects must also be notified that they are free to discontinue from the study at any time. The subject should be given the opportunity to ask questions and allowed time to consider the information provided before signing the ICF.

As additional assessments, the ICF will contain provisions for optional consent for the collection of blood samples for hormone and biomarker testing during screening and the collection of breast milk for biobanking and PK analysis purposes. The ICF, as specified by the clinical site's IRB, must follow the Protection of Human Subjects regulations listed in the Code of Federal Regulations, Title 21, Part 50.

The subject's signed and dated informed consent must be obtained before conducting any study procedures.

The Principal Investigator(s) must maintain the original, signed ICF. A copy of the signed ICF must be given to the subject.

#### 18. DATA HANDLING AND RECORDKEEPING

Procedures for data handling (including electronic data) used in this protocol will be documented in a Data Management Plan.

Electronic CRFs will be completed for each study subject. It is the Investigator's responsibility to ensure the accuracy, completeness, and timeliness of the data reported in the subject's eCRF. Source documentation supporting the eCRF data should indicate the subject's participation in the study and should document the dates and details of study procedures, adverse events, and subject status.

The Investigator will have access to the electronic data capture system and will receive a copy of the subject eCRF data at the end of the study. For subjects who discontinue or terminate from the study, the eCRFs will be completed as much as possible, and the reason for the discontinuation or termination clearly and concisely specified on the appropriate eCRF.

#### 18.1. Inspection of Records

Sage Therapeutics or designee will be allowed to conduct site visits to the investigational facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the monitor to inspect the drug storage area, study drug stocks, drug accountability records, subject charts and study source documents, and other records related to study conduct.

#### 18.2. Retention of Records

The Principal Investigator must maintain all documentation relating to the study for a period of 2 years after the last marketing application approval or, if not approved, 2 years following the discontinuation of the test article for investigation. If it becomes necessary for Sage Therapeutics or the Regulatory Authority to review any documentation relating to the study, the Investigator must permit access to such records.

# **18.3.** Confidentiality

To maintain subject privacy, all eCRFs, study reports, and communications will identify the subject by the assigned subject number. The Investigator will grant monitor(s) and auditor(s) from the Sponsor or its designee and regulatory authority(ies) access to the subject's original medical records for verification of data gathered on the eCRFs and to audit the data collection process. The subject's confidentiality will be maintained and will not be made publicly available to the extent permitted by the applicable laws and regulations.

Subjects will be notified that registration information, results, and other information about this study will be submitted to ClinicalTrials.gov, a publicly available trial registry database; however, protected health information of individual subjects will not be used.

All information regarding the investigational product supplied by Sage Therapeutics to the Investigator is privileged and confidential information. The Investigator agrees to use this information to accomplish the study and will not use it for other purposes without consent from the Sponsor. It is understood that there is an obligation to provide the Sponsor with complete data obtained during the study. The information obtained from the clinical study will be used towards the development of the investigational product and may be disclosed to regulatory authorities, other Investigators, corporate partners, or consultants, as required.

#### 19. PUBLICATION POLICY

All information concerning SAGE-217 is considered confidential and shall remain the sole property of Sage Therapeutics. The Investigator agrees to use this information only in conducting the study and shall not use it for any other purposes without written approval from Sage Therapeutics. No publication or disclosure of study results will be permitted except as specified in a separate, written, agreement between Sage Therapeutics and the Investigator.

#### **20.** LIST OF REFERENCES

Angst J, Angst F, Stassen HH. Suicide risk in patients with major depressive disorder. J Clin Psychiatry. 1999;60 Suppl 2:57-62; discussion 75-6, 113-6.

Conradi HJ, Ormel J, de Jonge P. Presence of individual (residual) symptoms during depressive episodes and periods of remission: a 3-year prospective study. Psychol Med. 2011 Jun;41(6):1165-74.

Drugan RC, Morrow AL, Weizman R, et al. Stress-induced behavioral depression in the rat is associated with a decrease in GABA receptor-mediated chloride ion flux and brain benzodiazepine receptor occupancy. Brain Res. 1989;487: 45–51.

DSM-5. Diagnostic and statistical manual of mental disorders (5th ed.). American Psychiatric Association 2013. Arlington, VA: American Psychiatric Publishing.

Fournier JC, DeRubeis RJ, Hollon SD, et al. Antidepressant drug effects and depression severity—a patient-level meta-analysis. JAMA. 2010;303:47-53.

Gerner RH, Hare TA. GABA in normal subjects and patients with depression, schizophrenia, mania, and anorexia nervosa. Am J Psychiatry. 1981;138:1098–101.

Greenberg PE, Fournier AA, Sisitsky T, Pike CT, Kessler RC. The economic burden of adults with major depressive disorder in the United States (2005 and 2010). J Clin Psychiatry. 2015 Feb;76(2):155-62.

Hamilton M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32:50-5.

Hamilton M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960;23:56-62.

Honig A, Bartlett JR, Bouras N, Bridges PK. Amino acid levels in depression: a preliminary investigation. J Psychiatr Res. 1988; 22:159–64.

Kirsch I, Deacon BJ, Huedo-Medina TB, et al. Initial severity and antidepressant benefits: A meta-analysis of data submitted to the Food and Drug Administration. PLoS Med. 2008;5(2):e45.

Luscher B, Shen Q, Sahir N. The GABAergic deficit hypothesis of major depressive disorder. Mol Psychiatry. 2011;16(4):383-406.

Maguire J, Mody I. GABA(A)R plasticity during pregnancy: Relevance to postpartum depression. Neuron. 2008;59(2);207-13.

Maguire J, Ferando I, Simonsen C, Mody I. Excitability changes related to GABAA receptor plasticity during pregnancy. J Neurosci. 2009;29(30):9592-601.

Mann JJ, Oguendo MA, Watson KT, et al. Anxiety in major depression and cerebrospinal fluid free gamma-aminobutyric acid. Depress Anxiety. 2014;31(10):814-21.

McDowell, I. Measuring Health: A guide to rating scales and questionnaires. 2006: 3rd Ed. New York: Oxford University Press.

Müller-Thomsen T, Arlt S, Mann U, Mass R, Ganzer S. Detecting depression in Alzheimer's disease: evaluation of four different scales. Arch Clin Neuropsychol. 2005;20:271-6.

Posner K, Brown GK, Stanley B, et al. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011;168(12):1266-77.

Romera I, Pérez V, Ciudad A, et al. Residual symptoms and functioning in depression, does the type of residual symptom matter? A post-hoc analysis. BMC Psychiatry. 2013 Feb 11;13:51.

Schüle C, Nothdurfter C, Rupprecht R. The role of allopregnanolone in depression and anxiety. Prog Neurobiol. 2014 Feb;113:79-87.

Trivedi MH, Rush AJ, Wisniewski SR, et al. (STAR\*D Study Team). Evaluation of outcomes with citalopram for depression using measurement-based care in STAR\*D: implications for clinical practice. Am J Psychiatry. 2006 Jan;163(1):28-40.

Ware JE Jr, Kosinski M, Bjorner JB, et al. User's Manual for the SF-36v2 Health Survey. 2nd ed. Lincoln, RI: QualityMetric Incorporated; 2007.

# 21. APPENDICES

# APPENDIX 1. HAMILTON RATING SCALE FOR DEPRESSION, **17-ITEM (HAM-D)**

| | Patient Name: | Date: |
|---|---|---|
| | Hamilton Rating Scale fo | or Depression (17-items) |
| | Instructions: For each item select the "cue" which best characterizes th | the patient during the past week. |
| 1. | Depressed Mood (sadness, hopeless, helpless, worthless) Absent These feeling states indicated only on questioning These feeling states spontaneously reported verbally Communicates feeling states nonverbally, i.e., through facial expression, posture, voice and tendency to weep A Patient reports VIRTUALLY ONLY these feeling states in his spontaneous verbal and nonverbal communication | 9. Agitation 0 None 1 "Playing with" hand, hair, etc. 2 Hand-wringing, nail-biting, biting of lips 10. Anxiety - Psychic 0 No difficulty 1 Subjective tension and irritability 2 Worrying about minor matters |
| 2. | Absent Self-reproach, feels he has let people down Ideas of guilt or rumination over past errors or sinful deeds Present illness is a punishment. Delusions of guilt Hears accusatory or denunciatory voices and/or experiences | 3 Apprehensive attitude apparent in face or speech 4 Fears expressed without questioning 11. Anxiety - Somatic 0 Absent Physiological concomitants of anxiety such 1 Mild Gastrointestinal - dry mouth, wind, indigesti 2 Moderate diarrhea, cramps, belching |
| 3. | threatening visual hallucinations Suicide Absent Feels life is not worth living Wishes he were dead or any thoughts of possible death to self Suicide ideas or gesture Attempts at suicide (any serious attempt rates 4) | 3 Severe Cardiovascular – palpitations, headaches 4 Incapacitating Respiratory - hyperventilation, sighing Urinary frequency Sweating |
| 4. | Insomnia - Early No difficulty falling asleep Complains of occasional difficulty falling asleep i.e., more than hour Complains of nightly difficulty falling asleep | Heavy feelings in abdomen. Difficulty eating without staff urging. Requests or requires laxatives or medications for bowels or medication for G.I. symptoms. |
| 5. | | <ul> <li>13. Somatic Symptoms - General <ul> <li>None</li> <li>Heaviness in limbs, back or head, backaches, headache, muscle aches, loss of energy and fatigability</li> <li>Any clear-cut symptom rates 2</li> </ul> </li> <li>14. Genital Symptoms <ul> <li>Absent</li> <li>Not ascertained</li> </ul> </li> </ul> |
| 6. | Insomnia - Late No difficulty Waking in early hours of the morning but goes back to sleep Unable to fall asleep again if gets out of bed | Mild Symptoms such as: loss of libido,<br>2 Severe menstrual disturbances Hypochondriasis Not present |
| 7. | Work and Activities No difficulty Thoughts and feelings of incapacity, fatigue or weakness related to activities; work or hobbies Loss of interest in activity; hobbies or work – either directly reported by patient, or indirect in listlessness, indecision and vacillation (feels he has to push self to work or activities) Decrease in actual time spent in activities or decrease in | Not present Self-absorption (bodily) Preoccupation with health Frequent complaints, requests for help, etc. Hypochondriacal delusions 16. Loss of Weight A. When Rating by History: No weight loss |
| 8. | productivity. In hospital, rate 3 if patient does not spend at least three hours a day in activities (hospital job or hobbies) exclusive of ward chores. 4 Stopped working because of present illness. In hospital, rate 4 if patient engages in no activities except ward chores, or if patient fails to perform ward chores unassisted. | Probable weight loss associated with present illness Definite (according to patient) weight loss B. On Weekly Ratings by Ward Revolution. When Actual |
| J. | (slowness of thought and speech; impaired ability to concentrate; decreased motor activity) Normal speech and thought Slight retardation at interview Obvious retardation at interview Interview difficult Complete stupor | Insight Acknowledges being depressed and ill Acknowledges illness but attributes cause to bad food, climate, overwork, virus, need for rest, etc. Denies being ill at all Intel Score: |

68

Total Score:

# APPENDIX 2. MONTGOMERY-ÅSBERG DEPRESSION RATING **SCALE (MADRS)**

#### Montgomery-Asberg Depression Rating Scale (MADRS)

The rating should be based on a clinical interview moving from broadly phrased questions about symptoms to more detailed ones which allow a precise rating of severity. The rater must decide whether the rating lies on the defined scale steps (0, 2, 4, 6) or between them (1, 3, 5) and then report the appropriate number. The items should be rated with regards to how the patient has done over the past week.

#### 1. Apparent sadness

Representing despondency, gloom and despair (more than just ordinary transient low spirits), reflected in speech, facial expression, and posture. Rate by depth and inability to brighten up.

- 0 = No sadness.
- 2 = Looks dispirited but does brighten up without difficulty.
- 4 = Appears sad and unhappy most of the time.
- 6 = Looks miserable all the time. Extremely despondent

#### 2. Reported sadness

Representing reports of depressed mood, regardless of whether it is reflected in appearance or not. Includes low spirits, despondency or the feeling of being beyond help and without hope.

- 0 = Occasional sadness in keeping with the circumstances.
- 2 = Sad or low but brightens up without difficulty.
  4 = Pervasive feelings of sadness or gloominess. The mood is still influenced by external circumstances.
- 6 = Continuous or unvarying sadness, misery or despondency.

#### 3. Inner tension

Representing feelings of ill-defined discomfort, edginess, inner turmoil, mental tension mounting to either panic, dread or anguish. Rate according to intensity, frequency, duration and the extent of reassurance called for.

- 0 = Placid. Only fleeting inner tension.
- 2 = Occasional feelings of edginess and ill-defined discomfort.
- 4 = Continuous feelings of inner tension or intermittent panic which the patient can only master with some
- 6 = Unrelenting dread or anguish. Overwhelming panic.

#### 4. Reduced sleep

Representing the experience of reduced duration or depth of sleep compared to the subject's own normal pattern when well.

- 0 = Sleeps as normal.
- 2 = Slight difficulty dropping off to sleep or slightly reduced, light or fitful sleep.
- 4 = Moderate stiffness and resistance
- 6 = Sleep reduced or broken by at least 2 hours.

#### 5. Reduced appetite

Representing the feeling of a loss of appetite compared with when-well. Rate by loss of desire for food or the need to force oneself to eat.

- 0 = Normal or increased appetite.
- 2 = Slightly reduced appetite.
- 4 = No appetite. Food is tasteless.
- 6 = Needs persuasion to eat at all.

#### 6. Concentration difficulties

Representing difficulties in collecting one's thoughts mounting to an incapacitating lack of concentration. Rate according to intensity, frequency, and degree of incapacity produced.

- 0 = No difficulties in concentrating.
- 2 = Occasional difficulties in collecting one's thoughts.
- 4 = Difficulties in concentrating and sustaining thought which reduced ability to read or hold a conversation.
- 6 = Unable to read or converse without great difficulty.

#### 7. Lassitude

Representing difficulty in getting started or slowness in initiating and performing everyday activities.

- 0 = Hardly any difficulty in getting started. No sluggishness.
- 2 = Difficulties in starting activities.
- 4 = Difficulties in starting simple routine activities which are carried out with effort.
   6 = Complete lassitude. Unable to do anything without help.

#### 8. Inability to feel

Representing the subjective experience of reduced interest in the surroundings, or activities that normally give pleasure. The ability to react with adequate emotion to circumstances or people is reduced.

- 0 = Normal interest in the surroundings and in other people.
- 2 = Reduced ability to enjoy usual interests.
- 4 = Loss of interest in the surroundings. Loss of feelings for friends and acquaintances.
- 6 = The experience of being emotionally paralysed, inability to feel anger, grief or pleasure and a complete or even painful failure to feel for close relatives and friends.

#### 9. Pessimistic thoughts

Representing thoughts of guilt, inferiority, self-reproach, sinfulness, remorse and ruin.

- 0 = No pessimistic thoughts.
- 2 = Fluctuating ideas of failure, self-reproach or self- depreciation.
- 4 = Persistent self-accusations, or definite but still rational ideas of guilt or sin. Increasingly pessimistic about the future.
- 6 = Delusions of ruin, remorse or irredeemable sin. Self- accusations which are absurd and unshakable.

#### 10. Suicidal thoughts

Representing the feeling that life is not worth living, that a natural death would be welcome, suicidal thoughts, and preparations for suicide. Suicide attempts should not in themselves influence the rating.

- 0 = Enjoys life or takes it as it comes.
- 2 = Weary of life. Only fleeting suicidal thoughts.
- 4 = Probably better off dead. Suicidal thoughts are common, and suicide is considered as a possible solution, but without specific plans or intenstion.
- 6 = Explicit plans for suicide when there is an opportunity. Active preparations for suicide.

© 1979 The Royal College of Psychiatrists. The Montgomery Åsberg Depression Rating Scale may be photocopied by individual researchers or clinicians for their own use without seeking permission from the publishers. The scale must be copied in full and all copies must acknowledge the following source: Montgomery, S.A. & Åsberg, M. (1979). A new depression scale designed to be sensitive to change. *British Journal of Psychiatry*, **134**, 382-389. Written permission must be obtained from the Royal College of Psychiatrists for copying and distribution to others or for republication (in print, online or by any other medium).

# APPENDIX 3. HAMILTON ANXIETY RATING SCALE (HAM-A)

| | low is a list of phrases that des<br>which he/she has these conditi | | | e patients by finding the answer w<br>of the fourteen questions. | which best describes the extent |
|---|---|---|---|---|---|
| 0 = | Not present, | I = Mild, | 2 = Moderate, | 3 = Severe, | 4 = Very severe |
| ı | Anxious mood | 0 1 2 3 4 | 8 | Somatic (sensory) | 0 1 2 3 4 |
| W | orries, antidipation of the wors | st, fearful anticipation, irritabil | | Tinnitus, blurring of vision, hot and cold flushes, feelings of weakness, pricking sensation. | |
| | Tension<br>elings of tension, fatigability, sta<br>sily, trembling, feelings of restle | | Tad | Cardiovascular symptoms<br>hycardia, palpitations, pain in ches<br>ngs, missing beat. | 0 1 2 3 4<br>t, throbbing of vessels, fainting |
| | Fears<br>dark, of strangers, of being lef<br>owds. | [0] [1] [2] [3] [4] it alone, of animals, of traffic, | of 10 | Respiratory symptoms | 0 1 2 3 4 |
| 4 | Insomnia | [0] [1] [2] [3] [4] | 11 | Gastrointestinal symptoms | 0 1 2 3 4 |
| | ficulty in falling asleep, broken<br>waking, dreams, nightmares, n | | abd | Difficulty in swallowing, wind abdominal pain, burning sensations,<br>abdominal fullness, nausea, vomiting, borborygmi, looseness of<br>bowels, loss of weight, constitution. | |
| S<br>Di | Intellectual<br>ficulty in concentration, poor | 0 [ 2 3 4 memory. | 12 | Genitourinary symptoms | 0 1 2 3 4 |
| 6<br>La | Depressed mood<br>ss of interest, lack of pleasure | 0 1 2 3 4<br>In hobbies, depression, early | mer | Frequency of micturition, urgency of micturition, amenorrhag,<br>menorrhagia, development of frigidity, premature ejaculation, loss of<br>libido, impotence. | |
| diu | irnal swing. | | 13 | Autonomic symptoms | 0 [ 2 3 4 |
| 7 Somatic (muscular) [0] [1] [2] [3] [4] Pains and aches, twitching, stiffness, myodonic jerks, grinding of teeth, unsteady voice, increased muscular tone. | | of hear | mouth, flushing, pallor, tendency<br>dache, raising of hair. | 1555 St | |
| | and an expensive and an | MATTER | Fidg | Behavior at interview<br>eting, restlessness or pacing, trem<br>ined face, sighing or rapid respirat | |

# APPENDIX 4. CLINICAL GLOBAL IMPRESSION–IMPROVEMENT SCALE (CGI-I) AND SEVERITY SCALE (CGI-S)

#### 1. Severity of illness

Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?

 $\begin{array}{ll} 0 = Not \ assessed & 4 = Moderately \ ill \\ I = Normal, \ not \ at \ all \ ill & 5 = Markedly \ ill \\ 2 = Borderline \ mentally \ ill & 6 = Severely \ ill \end{array}$ 

3 = Mildly ill 7 = Among the most extremely ill patients

2. Global improvement: Rate total improvement whether or not, in your judgement, it is due entirely to drug treatment.

Compared to his condition at admission to the project, how much has he changed?

#### 3. Efficacy index: Rate this item on the basis of drug effect only.

Select the terms which best describe the degrees of therapeutic effect and side effects and record the number in the box where the two items intersect.

EXAMPLE: Therapeutic effect is rated as 'Moderate' and side effects are judged 'Do not significantly interfere with patient's functioning'.

| Therapeutic effect | | Side effects | | | |
|---|---|---|---|---|---|
| | | None | Do not significantly<br>interfere with<br>patient's functioning | Significantly interferes<br>with patient's<br>functioning | Outweighs<br>therapeutic<br>effect |
| Marked | Vast improvement. Complete or nearly complete remission of all symptoms | 01 | 02 | 03 | 04 |
| Moderate | Decided improvement. Partial remission of symptoms | 05 | 06 | 07 | 08 |
| Minimal | Slight improvement which doesn't alter status of care of patient | 09 | 10 | П | 12 |
| Unchanged | d or worse | 13 | 14 | 15 | 16 |
| Not assessed = 00 | | | | | |

Reproduced from Guy W, editor. ECDEU Assessment Manual for Psychopharmacology. 1976. Rockville, MD, U.S. Department of Health, Education, and Welfare

# **APPENDIX 5. SHORT-FORM 36 (SF-36)**

#### SF-36 QUESTIONNAIRE

| Name: | Ref. Dr: | | | Date: |
|---|---|---|---|---|
| ID#: | Age: | | Gender: M / F | |
| Please answer the 36 questions of | the Health Survey comp | letely, honestly, | and without intern | uptions. |
| GENERAL HEALTH: | THE STATE OF THE S | | | |
| In general, would you say your h | ealth is:<br>erv Good | Good | OFair | Poor |
| Compared to one year ago, how | would you rate your hea | alth in general | now? | |
| Somewhat better now than one year | Charles and the second | | | |
| About the same | year ago | | | |
| Somewhat worse now than one | year ago | | | |
| Much worse than one year ago | * | | | |
| LIMITATIONS OF ACTIVITIES:<br>The following items are about activities? If so, how much? | ies you might do during a | typical day. Do | es your health now | limit you in the |
| Vigorous activities, such as runni | ing, lifting heavy objects | s, participating | in strenuous spo | rts. |
| CYes, Limited a lot | Yes, Limited a Little | | ONo, Not Limited | at all |
| Moderate activities, such as movi | ng a table, pushing a va | acuum cleaner, | bowling, or playi | ng golf |
| CYes, Limited a Lot | Yes, Limited a Little | | ONo, Not Limited | |
| Lifting or carrying groceries Over Limited a Lot | OYes, Limited a Little | | CNo, Not Limited | at all |
| Climbing several flights of stairs<br>Yes, Limited a Lot | OYes, Limited a Little | | ○No, Not Limited | at all |
| Climbing one flight of stairs Yes, Limited a Lot | OYes, Limited a Little | | ONo, Not Limited | at all |
| Bending, kneeling, or stooping<br>CYes, Limited a Lot | OYes, Limited a Little | | CNo, Not Limited | at all |
| Walking more than a mile<br>CYes, Limited a Lot | OYes, Limited a Little | | CNo, Not Limited | at all |
| Walking several blocks Yes, Limited a Lot | OYes, Limited a Little | | CNo, Not Limited | at all |
| Walking one block Yes, Limited a Lot | ○Yes, Limited a Little | | ○No, Not Limited | at all |

| Bathing or dressing yourself | | | |
|---|---|---|---|
| CYes, Limited a Lot | OYes, Limited a I | Little | No, Not Limited at all |
| PHYSICAL HEALTH PROBLEM<br>During the past 4 weeks, have y<br>a result of your physical health? | | ving problems with you | r work or other regular daily activities as |
| Cut down the amount of time y | ou spent on work or | other activities | |
| | CNo | other dedvices | |
| Accomplished less than you w | ould like | | |
| CYes | CNo | | |
| Were limited in the kind of wo | k or other activities | | |
| CYes | CNo | | |
| Had difficulty performing the v | | (for example, it took | extra effort) |
| CYes | CNo | | |
| EMOTIONAL HEALTH PROBLE<br>During the past 4 weeks, have y<br>a result of any emotional probler | ou had any of the follow | | r work or other regular daily activities as |
| Cut down the amount of time y | ou spent on work or | other activities | |
| Accomplished less than you w | ould like<br>ONo | | |
| Didn't do work or other activiti | es as carefully as usu<br>No | ial | |
| SOCIAL ACTIVITIES:<br>Emotional problems interfered | with your normal soc | cial activities with fam | illy, friends, neighbors, or groups? |
| CNot at all CSlight | y OModerate | ly OSeve | re CVery Severe |
| PAIN:<br>How much bodily pain have you had during the past 4 weeks? | | | |
| CNone Overy Mild | CMild CMd | oderate OSe | vere Overy Severe |
| During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? | | | |
| CNot at all OA little | oit OModera | tely Cquite | a bit Extremely |

None of the Time

| ENERGY AND EMOTIONS: |
|---|
| These questions are about how you feel and how things have been with you during the last 4 weeks. For each |
| question, please give the answer that comes closest to the way you have been feeling. |
| Did you feel full of pep? |
| CAll of the time |
| CMost of the time |
| CA good Bit of the Time |
| Some of the time |
| CA little bit of the time |
| CNone of the Time |
| Have you been a very nervous person? |
| CAll of the time |
| CMost of the time |
| CA good Bit of the Time |
| CSome of the time |
| CA little bit of the time |
| CNone of the Time |
| Have you felt so down in the dumps that nothing could cheer you up? |
| CAll of the time |
| CMost of the time |
| CA good Bit of the Time |
| CSome of the time |
| A little bit of the time |
| None of the Time |
| Have you felt calm and peaceful? |
| All of the time |
| Most of the time |
| A good Bit of the Time |
| Some of the time |
| A little bit of the time |
| CNone of the Time |
| Did you have a lot of energy? |
| CAll of the time |
| Most of the time |
| CA good Bit of the Time |
| Some of the time |
| CA little bit of the time |

| Have you felt downhearted and All of the time Most of the time A good Bit of the Time Some of the time A little bit of the time None of the Time | blue? |
|---|---|
| Did you feel worn out? All of the time Most of the time A good Bit of the Time Some of the time A little bit of the time None of the Time | |
| Have you been a happy person All of the time Most of the time A good Bit of the Time Some of the time A little bit of the time None of the Time | ? |
| Did you feel tired? All of the time Most of the time A good Bit of the Time Some of the time A little bit of the time None of the Time | |
| | nuch of the time has your physical health or emotional problems interfered with<br>ng with friends, relatives, etc.)? |
| All of the time Most of the time Some of the time A little bit of the time | |

# Sage Therapeutics

| GENERAL HEALTH: How true or false is each of the following statements for you? | | | | |
|---|---|---|---|---|
| I seem to get sick a little easier than other people Definitely true Mostly true Don't know Mostly false | | | | |
| I am as healthy as anyl | body I know | CDon't know | OMostly false | Opefinitely false |
| Lexpect my health to g | | CDOTT KNOW | Mostly laise | Definitely false |
| Definitely true | Mostly true | Opon't know | Mostly false | ODefinitely false |
| My health is excellent Definitely true | Mostly true | ODon't know | Mostly false | Opefinitely false |

# APPENDIX 6. THE FATIGUE ASSOCIATED WITH DEPRESSION (FAs-D) PATIENT-REPORTED OUTCOME (PRO)

Some people experience fatigue when they are depressed. The following items ask you to rate fatigue you have experienced that you think may be related to depression.

| In the PAST WEEK, how often have you felt | | Never | Rarely | Sometimes | Often | Always |
|---|---|---|---|---|---|---|
| 1. Fat | tigued | 1 | 2 | 3 | 4 | 5 |
| 2. Tir | red | 1 | 2 | 3 | 4 | 5 |
| 3. Ex | hausted | 1 | 2 | 3 | 4 | 5 |
| 4. Lik | ke you had no energy | 1 | 2 | 3 | 4 | 5 |
| 5. Ph | ysically weak | 1 | 2 | 3 | 4 | 5 |
| 6. Slo | owed down | 1 | 2 | 3 | 4 | 5 |
| 7. Lik | ke everything requires too much effort | 1 | 2 | 3 | 4 | 5 |

Now think about the impact of this fatigue that is related to depression. The following items ask about the impact of this fatigue on various aspects of your life.

| In the PAST WEEK, how much has your fatigue | Not at all | A little | Somewhat | Quite a bit | Very much |
|---|---|---|---|---|---|
| Limited your ability to complete daily household chores | 1 | 2 | 3 | 4 | 5 |
| <ol> <li>Interfered with family activities or relationships</li> </ol> | 1 | 2 | 3 | 4 | 5 |
| 10. Interfered with doing things you enjoy | 1 | 2 | 3 | 4 | 5 |
| 11. Interfered with social activities, like spending time with friends | 1 | 2 | 3 | 4 | 5 |
| 12. Interfered with taking care of yourself (e.g., bathing, dressing, brushing your teeth) | 1 | 2 | 3 | 4 | 5 |
| 13. Kept you from getting out of bed | 1 | 2 | 3 | 4 | 5 |

| Do v | vou have a si | pouse or significant other? | □ Yes | □ No |
|------|---------------|-----------------------------|-------|------|

If no, leave item 14 blank.

If yes, please answer item 14.

| In the PAST WEEK, how much has your fatigue | Not at all | A little | Somewhat | Quite a bit | Very much |
|---|---|---|---|---|---|
| 14. Interfered with your intimate relationship (i.e., with a spouse or significant other) | 1 | 2 | 3 | 4 | 5 |

**Do you have a job or go to school?**  $\Box$  Yes  $\Box$  No

If no, leave items 15 and 16 blank.

If yes, please answer items 15 and 16.

| In the past week, how much has your fatigue | Not at all | A little | Somewhat | Quite a bit | Very much |
|---|---|---|---|---|---|
| 15. Prevented you from going to work or school | 1 | 2 | 3 | 4 | 5 |
| <ol><li>Limited your productivity at work or<br/>school</li></ol> | 1 | 2 | 3 | 4 | 5 |

# APPENDIX 7. COLUMBIA - SUICIDE SEVERITY RATING SCALE (C-SSRS)

# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Baseline/Screening Version

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <u>The Columbia Suicide History Form</u>, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103-130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

© 2008 The Research Foundation for Mental Hygiene, Inc.

| SUICIDAL IDEATION | | | | |
|---|---|---|---|---|
| Ask questions 1 and 2. If both are negative, proceed to "Suicidal Behavior" section. If the answer to | Lifetim | e: Time | Past | |
| question 2 is "yes", ask questions 3, 4 and 5. If the answer to question 1 and/or 2 is "yes", complete | He/Sh | | Mor | |
| "Intensity of Ideation" section below. | Most S | meigai | | |
| <ol> <li>Wish to be Dead</li> <li>Subject endorses thoughts about a wish to be dead or not alive anymore, or wish to fall asleep and not wake up.</li> </ol> | Yes | No | Yes | No |
| Have you wished you were dead or wished you could go to sleep and not wake up? | | | | |
| If yes, describe: | " | | | |
| 2. Non-Specific Active Suicidal Thoughts | | | | |
| General non-specific thoughts of wanting to end one's life/commit suicide (e.g., "I've thought about killing myself") without thoughts | Yes | No | Yes | No |
| of ways to kill oneself/associated methods, intent, or plan during the assessment period. Have you actually had any thoughts of killing yourself? | | | | |
| If yes, describe: | | | | |
| 3. Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act Subject endorses thoughts of suicide and has thought of at least one method during the assessment period. This is different than a | Yes | No | Yes | No |
| specific plan with time, place or method details worked out (e.g. thought of method to kill self but not a specific plan). Includes person | | | | |
| who would say, "I thought about taking an overdose but I never made a specific plan as to when, where or how I would actually do | | ш | | _ |
| itand I would never go through with it." Have you been thinking about how you might do this? | | | | |
| If yes, describe: | | | | |
| 4. Active Suicidal Ideation with Some Intent to Act, without Specific Plan | | | | |
| Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "Thave the | Yes | No | Yes | No |
| thoughts but I definitely will not do anything about them." | | | | |
| Have you had these thoughts and had some intention of acting on them? | | | | |
| If yes, describe: | | | | |
| 5. Active Suicidal Ideation with Specific Plan and Intent | *** | 2. | *** | |
| Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out. Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan? | Yes | No | Yes | No |
| If yes, describe: | | | | |
| • | | | | |
| INTENSITY OF IDEATION The following features should be rated with respect to the most severe type of ideation (i.e., 1.5 from above, with I being | Г | | Г | |
| INTENSITY OF IDEATION The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. | | | | |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. | M | net | Me | net |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being | Me<br>Sev | ost | Mo<br>Sev | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (1-5) Description of Ideation | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (1-5) Description of Ideation Past X Months - Most Severe Ideation: Type # (1-5) Description of Ideation Frequency | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Past X Months - Most Severe Ideation: Type # (I-5) Description of Ideation Frequency How many times have you had these thoughts? | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Past X Months - Most Severe Ideation: Type # (I-5) Description of Ideation Frequency How many times have you had these thoughts? | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (1-5) Description of Ideation Past X Months - Most Severe Ideation: Type # (1-5) Description of Ideation Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (4) 4-8 hours/most of day | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (5) More than 8 hours/persistent or continuous | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (1-5) Description of Ideation Past X Months - Most Severe Ideation: Type # (1-5) Description of Ideation Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (4) 4-8 hours/most of day | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (5) More than 8 hours/persistent or continuous (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to die if you want to? | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Type # (I-5) Description of Ideation Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts with a lot of difficulty | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (5) More than 8 hours/persistent or continuous (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to die if you want to? | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Past X Months - Most Severe Ideation: Type # (I-5) Description of Ideation Perquency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Feeting - few seconds or minutes (2) Less than 1 hour/some of the time (5) More than 8 hours/persistent or continuous (3) 1-4 hours/a lot of time Controllability Control any ou stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts with little difficulty (5) Unable to control thoughts with a lot of difficulty (5) Unable to control thoughts (3) Can control thoughts with some difficulty (6) Does not attempt to control thoughts Deterrents | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Type # (I-5) Description of Ideation Type # (I-6) Description of Ideation Type # (I-7) Description of Ideation Type # (I-8) Description of Ideation When many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (5) More than 8 hours/persistent or continuous (3) 1-4 hours/a lot of time Controllability Condictan you stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts with a lot of difficulty (5) Unable to control thoughts with some difficulty (6) Does not attempt to control thoughts Are there things - anyone or anything (e.g., family, religion, pain of death) - that stopped you from wanting to | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Past X Months - Most Severe Ideation: Type # (I-5) Description of Ideation Percuency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (5) More than 8 hours/persistent or continuous (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts with some difficulty (5) Unable to control thoughts (3) Can control thoughts with some difficulty (5) Unable to control thoughts Are there things - anyone or anything (e.g., family, religion, pain of death) - that stopped you from wanting to die or acting on thoughts of committing suicide? | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Past X Months - Most Severe Ideation: Type # (I-5) Description of Ideation Perequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (5) More than 8 hours/persistent or continuous (3) 1-4 hours/a lot of time Controllability Condid-can you stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts with little difficulty (5) Unable to control thoughts with a lot of difficulty (5) Unable to control thoughts with a lot of difficulty (5) Unable to control thoughts Are there things - anyone or anything (e.g., family, religion, pain of death) - that stopped you from wanting to die or acting on thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents definitely stopped you from attempting suicide (2) Deterrents definitely did not stop you (5) Deterrents definitely did not stop you | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Past X Months - Most Severe Ideation: Type # (I-9) Description of Ideation Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (5) More than 8 hours/persistent or continuous (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts with little difficulty (5) Unable to control thoughts with a lot of difficulty (5) Unable to control thoughts with an old of difficulty (5) Unable to control thoughts Are there things - anyone or anything (e.g., family, religion, pain of death) - that stopped you from wanting to die or acting on thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents definitely stopped you (5) Deterrents most likely did not stop you (6) Dees not apply | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Past X Months - Most Severe Ideation: Type # (I-5) Description of Ideation Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts with some difficulty (5) Unable to control thoughts with some difficulty (5) Unable to control thoughts with some difficulty (5) Unable to control thoughts with some difficulty (6) Does not attempt to control thoughts Are there things - anyone or anything (e.g., family, religion, pain of death) - that stopped you from wanting to die or acting on thoughts of committing suicide? (1) Deterrents definitely stopped you (3) Uncertain that deterrents stopped you (3) Uncertain that deterrents stopped you (4) Deterrents definitely did not stop you (5) Deterrents definitely did not stop you (6) Deterrents definitely did not stop you (7) Deterrents definitely did not stop you (8) Deterrents definitely did not stop you (9) Does not apply | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Past X Months - Most Severe Ideation: Type # (I-9) Description of Ideation Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (5) More than 8 hours/persistent or continuous (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts with little difficulty (5) Unable to control thoughts with a lot of difficulty (5) Unable to control thoughts with an old of difficulty (5) Unable to control thoughts Are there things - anyone or anything (e.g., family, religion, pain of death) - that stopped you from wanting to die or acting on thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents definitely stopped you (5) Deterrents most likely did not stop you (6) Dees not apply | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Past X Months - Most Severe Ideation: Type # (I-5) Description of Ideation Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Pleeting - Iew seconds or minutes (5) More than 8 hours/persistent or continuous (3) 1-4 hours/a lot of time (5) More than 8 hours/persistent or continuous (2) Less than 1 hour/some of the time (5) More than 8 hours/persistent or continuous (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts with little difficulty (5) Unable to control thoughts with a lot of difficulty (3) Can control thoughts with some difficulty (5) Unable to control thoughts 3) Can control thoughts with some difficulty (6) Does not attempt to control thoughts Deterrents Are there things - anyone or anything (e.g., family, religion, pain of death) - that stopped you from wanting to die or acting on thoughts of committing suicide? (1) Deterrents definitely stopped you (5) Deterrents most likely did not stop you (5) Deterrents most likely did not stop you (6) Does not apply Reasons for Ideation What sort of reasons did you have for thinking about wanting to die or killing yourself? Was it to end the pain or stop the way you were feeling (in other words you couldn't go on living with this pain or how you were feeling or was it to get attention, revenge or a reaction from others? Or both? | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (i-5) Description of Ideation | | | 220000 | 1000 |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. Lifetime - Most Severe Ideation: Type # (I-5) Description of Ideation Past X Months - Most Severe Ideation: Type # (I-5) Description of Ideation Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day Duration When you have the thoughts how long do they last? (1) Pleeting - Iew seconds or minutes (5) More than 8 hours/persistent or continuous (3) 1-4 hours/a lot of time (5) More than 8 hours/persistent or continuous (2) Less than 1 hour/some of the time (5) More than 8 hours/persistent or continuous (3) 1-4 hours/a lot of time Controllability Could/can you stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts with little difficulty (5) Unable to control thoughts with a lot of difficulty (3) Can control thoughts with some difficulty (5) Unable to control thoughts 3) Can control thoughts with some difficulty (6) Does not attempt to control thoughts Deterrents Are there things - anyone or anything (e.g., family, religion, pain of death) - that stopped you from wanting to die or acting on thoughts of committing suicide? (1) Deterrents definitely stopped you (5) Deterrents most likely did not stop you (5) Deterrents most likely did not stop you (6) Does not apply Reasons for Ideation What sort of reasons did you have for thinking about wanting to die or killing yourself? Was it to end the pain or stop the way you were feeling (in other words you couldn't go on living with this pain or how you were feeling or was it to get attention, revenge or a reaction from others? Or both? | | | 220000 | 1000 |

© 2008 Research Foundation for Mental Hygiene, Inc.

C-SSRS—Baseline/Screening (Version 1/14/09)


| SUICIDAL BEHAVIOR (Check all that apply, so long as these are separate events; must ask about all types) | | Life | time | Past<br>Years | |
|---|---|---|---|---|---|
| Actual Attempt: | | Yes | No | Yes | No |
| A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as moneself. Intent does not have to be 100%. If there is any intent/desire to die associated with the act, then it can be considered at attempt. There does not have to be any injury or harm, just the potential for injury or harm. If person pulls trigger whi mouth but gun is broken so no injury results, this is considered an attempt. Inferring Intent: Even if an individual deries intent/wish to die, it may be inferred clinically from the behavior or circumstances | n actual suicide<br>ile gun is in<br>. For example, a | | | | |
| highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping from high floor/story). Also, if someone denies intent to die, but they thought that what they did could be lethal, intent may be inferre Have you made a suicide attempt? | | | | | |
| Have you done anything to harm yourself? | | | l#of | Total | |
| Have you done anything dangerous where you could have died? What did you do? | | Atte | mpts | Atte | mpts |
| Did you as a way to end your life? | | - | _ | _ | _ |
| Did you want to die (even a little) when you? Were you trying to end your life when you ? | | | | | |
| Or Did you think it was possible you could have died from ? | | | | | |
| Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress, | feel better, | | | | |
| get sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) If yes, describe: | | | 123 | | <b>N</b> T |
| n you deallow. | | 100000 | No | Yes | No |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | | | | | |
| Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual have occurred). | l attempt would | Yes | No | Yes | No |
| Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather tha attempt. Shooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pullin they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down Hanging: Person has noose around neck but has not yet started to hang - is stopped from doing so. | ng trigger. Once | | | | |
| Has there been a time when you started to do something to end your life but someone or something stopp | ed you before | | l#of<br>upted | Total<br>interr | |
| you actually did anything? If yes, describe: | | | _ | | _ |
| Aborted Attempt: | | Yes | No | Yes | No |
| When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in a destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being something else. | | | | | |
| Has there been a time when you started to do something to try to end your life but you stopped yourself be actually did anything? | efor e you | | l#of<br>orted | Total<br>abou | |
| If yes, describe: | | _ | | - | |
| Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things at suicide note). | | Yes | No | Yes | No |
| Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting | ng pills, | | | | |
| getting a gun, giving valuables away or writing a suicide note)? If yes, describe: | \$555. | | | | |
| Suicidal Behavior: | | Yes | No | Yes | No |
| Suicidal behavior was present during the assessment period? | | | | | |
| Answer for Actual Attempts Only | Most Recent<br>Attempt<br>Date: | Most Leth<br>Attempt<br>Date: | | Initial/Fi<br>Attempt<br>Date: | rst |
| Actual Lethality/Medical Damage: | Enter Code | Enter ( | - | Enter | Code |
| No physical damage or very minor physical damage (e.g., surface scratches). Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree | | | | | |
| burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes | | | | | |
| intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage, medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death | | | | | |
| Potential Lethality: Only Answer if Actual Lethality=0 | Enter Code | Enter C | ode: | Enter | Code |
| Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). | | | 0.000000 | | |
| 0 = Behavior not likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | | _ | - | - | _ |

 $\mathbb C$  2008 Research Foundation for Mental Hygiene, Inc.

C-SSRS—Baseline/Screening (Version 1/14/09)


# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Since Last Visit

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <u>The Columbia Suicide History Form</u>, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103-130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

© 2008 The Research Foundation for Mental Hygiene, Inc.

| CUICIDAL IDEATION | | | |
|---|---|---|---|
| | uicidal Behavior" section. If the answer to question 2 is "yes",<br>r 2 is "yes", complete "Intensity of Ideation" section below. | | e Last<br>'isit |
| Wish to be Dead Subject endorses thoughts about a wish to be dead or not alive anymore, of Have you wished you were dead or wished you could go to sleep and no. | | Yes | No |
| If yes, describe: | | - | _ |
| 2. Non-Specific Active Suicidal Thoughts General, non-specific thoughts of wanting to end one's life/commit suicic oneself/associated methods, intent, or plan during the assessment period. Have you actually had any thoughts of killing yourself? | le (e.g., "I've thought about killing myself") without thoughts of ways to kill | Yes | No |
| If yes, describe: | | | |
| | od during the assessment period. This is different than a specific plan with time, it not a specific plan). Includes person who would say, "I thought about taking an | Yes | No |
| If yes, describe: | | | |
| 4. Active Suicidal Ideation with Some Intent to Act, witho Active suicidal thoughts of killing oneself and subject reports having som definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them | e intent to act on such thoughts, as opposed to "I have the thoughts but I | Yes | No |
| If yes, describe: | | | |
| 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked of Have you started to work out or worked out the details of how to kill you | | Yes | No |
| If yes, describe: | | | |
| INTENSITY OF IDEATION | | | |
| | evere type of ideation (i.e., 1-5 from above, with 1 being the least severe | M | lost |
| Most Severe Ideation: | | Se | vere |
| Type# (1-5) | Description of Ideation | | |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in weel | k (4) Daily or almost daily (5) Many times each day | - | |
| Duration When you have the thoughts, how long do they last? | | | |
| (1) Fleeting - few seconds or minutes | (4) 4-8 hours/most of day<br>(5) More than 8 hours/persistent or continuous | - | |
| (2) Can control thoughts with little difficulty | tg to die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts | - | |
| Deterrents Are there things - anyone or anything (e.g., family, religion, thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents probably stopped you (3) Uncertain that deterrents stopped you | pain of death) - that stopped you from wanting to die or acting on (4) Deterrents most likely did not stop you (5) Deterrents definitely did not stop you (0) Does not apply | _ | _ |
| Reasons for Ideation What sort of reasons did you have for thinking about wantin | g to die or killing yourself? Was it to end the pain or stop the way ith this pain or how you were feeling) or was it to get attention, (4) Mostly to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (5) Completely to end or stop the pain (you couldn't go on living with the pain or how you were feeling) | _ | |

© 2008 Research Foundation for Mental Hygiene, Inc.

(0) Does not apply
C-SSRS—Since Last Visit (Version 1/14/09)

| SUICIDAL BEHAVIOR (Check all that apply, so long as these are separate events; must ask about all types) | Since Last<br>Visit |
|---|---|
| Actual Attempt: A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as method to kill oneself. Intent does not have to be 100%. If there is any intent/desire to die associated with the act, then it can be considered an actual suicide attempt. There does not have to be any injury or harm, just the potential for injury or harm. If person pulls trigger while gun is in mouth but gun is broken so no injury results, this is considered an attempt. | Yes No |
| Inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumstances. For example, a highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping from window of a high floor/story). Also, if someone denies intent to die, but they thought that what they did could be lethal, intent may be inferred. Have you made a suicide attempt? | |
| Have you done anything to harm yourself? | Total # of |
| Have you done anything dangerous where you could have died? What did you do? | Attempts |
| Did you as a way to end your life? | 1985 |
| Did you want to die (even a little) when you? | |
| Were you trying to end your life when you? | |
| Or did you think it was possible you could have died from? Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress, feel better, g et | |
| sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) If yes, describe: | |
| | Yes No |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | |
| Interrupted Attempt: | 10000111 51.01 |
| When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have occurred). | Yes No |
| Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. Shooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has noose around neck but has not yet started to hang - is stopped from doing so. | |
| Has there been a time when you started to do something to end your life but someone or something stopped you before you | Total # of |
| actually did anything? | interrupted |
| If yes, describe: | |
| Aborted Attempt: | Yes No |
| When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. | |
| Has there been a time when you started to do something to try to end your life but you stopped yourself before you | |
| actually did anything? | Total # of<br>aborted |
| If yes, describe: | aborted |
| Preparatory Acts or Behavior: | |
| Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a | Yes No |
| specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, | |
| giving valuables away or writing a suicide note)? | |
| If yes, describe: | |
| Suicidal Behavior: | Yes No |
| Suicidal behavior was present during the assessment period? | |
| Suicide: | Yes No |
| Answer for Actual Attempts Only | Most Lethal |
| | Attempt<br>Date: |
| Actual Lethality/Medical Damage: | Enter Code |
| No physical damage or very minor physical damage (e.g., surface scratches). Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). | |
| <ol><li>Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel).</li></ol> | |
| <ol> <li>Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns<br/>less than 20% of body; extensive blood loss but can recover; major fractures).</li> </ol> | |
| 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body, | - |
| extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death | |
| Potential Lethality: Only Answer if Actual Lethality=0 | Enter Co.4 |
| Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious | Enter Code |
| lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). | |
| 0 = Behavior not likely to result in injury | |
| 1 = Behavior likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | |

### APPENDIX 8. STANFORD SLEEPINESS SCALE (SSS)

#### Stanford Sleepiness Scale

This is a quick way to assess how alert you are feeling. If it is during the day when you go about your business, ideally you would want a rating of a one. Take into account that most people have two peak times of alertness daily, at about 9 a.m. and 9 p.m. Alertness wanes to its lowest point at around 3 p.m.; after that it begins to build again. Rate your alertness at different times during the day. If you go below a three when you should be feeling alert, this is an indication that you have a serious sleep debt and you need more sleep.

#### An Introspective Measure of Sleepiness The Stanford Sleepiness Scale (SSS)

| Degree of Sleepiness | Scale<br>Rating |
|---|---|
| Feeling active, vital, alert, or wide awake | 1 |
| Functioning at high levels, but not at peak; able to concentrate | 2 |
| Awake, but relaxed; responsive but not fully alert | 3 |
| Somewhat foggy, let down | 4 |
| Foggy; losing interest in remaining awake; slowed down | 5 |
| Sleepy, woozy, fighting sleep; prefer to lie down | 6 |
| No longer fighting sleep, sleep onset soon; having dream-like thoughts | 7 |
| Asleep | X |